**Official Title:** P3-T: Novel mHealth Technologies to Enhance PrEP Adherence among Thai YMSM, Collaborative Adaptation and Evaluation

NCT Number: NCT04413708

Document Date: March 16, 2021



This form effective August 28, 2017

## Part A. Study Information

## 1.1 Project Title

If the research is federally funded, the project title should match the grant title.

orative

| | ovel mHealth Technologies to Enhance PrEP Adherence among Thai MSM: Collabed aptation and Evaluation |
|---|---|
| 1.2 Pr | roject Information: |
| 1. | Source of Funding: |
| | □ Association □ NIH □ Foundation □ NSF □ Duke University □ DOD (Department, School, Institute, Program) □ USDA □ None □ Other Federal: □ Other: □ Enter grant number: 1 R21 TW010965-01 |
| 2. | Is this research part of a Bass Connections project? ☐Yes ☒ No If yes, include all the students in Part B: Researcher Information and Assurances. |
| 3. | Research Site, if research is taking place abroad: Bangkok, Thailand |
| 4. | Will the research take place in public elementary or secondary schools? $\square$ Yes $\boxtimes$ No If yes, identify the school district(s): $\underline{\hspace{1cm}}$ |
| 5. | Potentially Vulnerable Subject Populations: Please check all that apply. |
| | <ul> <li>☑ Children, as defined at research site (under 18 years old in NC)</li> <li>☐ Cognitively impaired persons, for example, people with dementia</li> <li>☐ Prisoners</li> <li>☐ Refugees</li> <li>☒ Stigmatized populations</li> <li>☐ Undocumented immigrants</li> <li>☐ Victims of abuse</li> <li>☐ Other:</li> </ul> |

## Part B: Researcher Information and Assurances

Researchers: (Faculty, Undergraduate or Graduate Student, Research Associate, Postdoctoral Fellow)

All signatories certify to the following:

- 1. I will not begin the research until written approval is secured from the IRB. Note: Approval will not be provided unless <u>certification to conduct research with human subjects</u> is current.
- 2. I will conduct this study as described in the approved protocol.
- 3. If any changes are anticipated, I will submit a <u>Request to Amend an Approved Protocol</u>, and I will not implement the changes until I receive approval from the IRB.
- 4. I will contact the IRB staff promptly if any of the following events occur: <u>unanticipated risks of harm to participants</u>, protocol deviations, and findings during the study that would affect the risks of participation.

| Name: Sara LeGrand | Department or School: <b>DGHI</b> |
|---|---|
| E-mail Address: sara.legrand@duke.edu | Phone Number: 919-438-0448 |
| ☐ Faculty ☐ Undergraduate ☐ Graduate student ☐ | Postdoc Research associate Other: |
| Signature: Sava Le Grand | Date: 9/16/19 |
| Name: Shashika Bandara | Department or School: DGHI |
| E-mail Address: shashika.bandara@duke.edu | Phone Number: 919-613-5449 |
| Faculty Undergraduate Graduate student | Postdoc Research associate Other: |
| Signature: | Date: 9/16/19 |
| Name: Caitlin Piccone Department or School: Duke Glob | |
| | Health Institute |
| E-mail Address & NetID: | Phone Number: <b>941-301-9494</b> |
| caitlin.piccone@gmail.com; CMM158 | |
| Research Associate | Postdoc Research associate Other: Voluntee |
| Signature: Dicconn | Date: 11/26/2019 |
| S USE ONLY section is to be completed by IRB staff or IRB members only | |
| PROVED as Exempt Expedited or | Full |

#### Part C: Research Protocol

## 2. Research Question

2.1 What is the research question?

Can an existing pre-exposure prophylaxis (PrEP) adherence app developed for young men who have sex with men (YMSM) in the US be successfully adapted, implemented and show trends toward efficacy (i.e., improved adherence) for YMSM in Bangkok, Thailand?

2.2 Provide background information about the research that will help the reviewer understand the research. Avoid discipline-specific jargon.

In Thailand, gay, bisexual, and other men who have sex with men (MSM) account for 41% of new HIV infections with an increasing trend in infections over time. 1,2 Young MSM (YMSM) are at a significantly greater risk of HIV infection than older MSM with YMSM, ages 15-21, experiencing a 12.1% rate of new HIV infections. 1,2 There is an urgent need to implement novel behavioral and biomedical interventions for YMSM in Thailand that are culturally and developmentally appropriate, engaging for youth, and scalable.

Pre-exposure prophylaxis (PrEP), a combination of tenofovir and emtricitabine, taken once daily is a safe, effective method of preventing HIV among YMSM.<sup>3-5</sup> However, efficacy is highly correlated with adherence and evidence suggests poorer adherence among younger populations.<sup>3,5,6</sup> It is imperative that we develop adherence interventions for YMSM initiating PrEP that take advantage of technologies that are already embedded in their lives. The *accessibility, affordability, anonymity* and *acceptability* of smartphones in Thailand make them the intervention medium of choice for engaging youth and a logical platform to deliver an adherence intervention targeting PrEP.<sup>7</sup> Further, smartphone interventions address and overcome issues that impede engagement with in-person interventions such as inconvenience, transportation, and stigma.<sup>8</sup>

This R21 study, titled "Novel mHealth Technologies to Enhance PrEP Adherence among Thai MSM: Collaborative Adaptation and Evaluation", adapts our theory-based smartphone app platform, **CHARGE** (Comprehensive health adherence using gaming and social engagement), to improve PrEP adherence among YMSM in Thailand and conducting a pilot study to assess study feasibility, acceptability, and potential impact. We propose a partnership between Duke University, Chulalongkorn University, Thai Red Cross AIDS Research Centre, and the University of North Carolina- Chapel Hill (UNC), and a robust plan to increase mHealth capacity at Thai Red Cross AIDS Research Centre (TRC-ARC).

**CHARGE** is a theory-based, comprehensive smartphone app platform for YMSM that utilizes social networking and game-based mechanics as well as evidenced-based features to improve medication adherence. **CHARGE** is a product born from the collaborative effort of researchers and health game developers working closely with members of the target population in the United States (US). Built on a successful, evidence-based platform designed by our collaborating technology partner, Ayogo, and tested by our study team, **CHARGE** is flexible, allowing for customization and adaptations for different cultural and linguistic contexts, and responsive to changes in technology.

The social networking features of **CHARGE** are designed to capitalize on social involvement as a means through which YMSM can receive information and social support, experience social norms and reflective appraisals, and feel a sense of connectedness to peers. <sup>9,10</sup> Peers have been recognized as a highly important source of sexual health and HIV prevention information and support among Thai YMSM. The gaming features of **CHARGE** are goal-oriented and immersive and provide a challenging and motivating environment for behavior change. <sup>11-14</sup> As a result, **CHARGE** is ideal for engaging YMSM in behavior change, by maintaining attention, avoiding boredom and attrition. <sup>15</sup>

The specific aims of this grant are to:

- 1. Conduct formative research to inform adaptions of the **CHARGE** platform for YMSM in Thailand. Using an iterative research design, we will work with members of the target population through focus groups, key informant interviews, a youth advisory board (YAB), and usability testing to tailor the platform for maximal relevance and usability for HIV-negative Thai YMSM (aged 16-24).
- Conduct a pilot randomized control trial (RCT) study of the app built using the CHARGE platform with 60 YMSM newly starting PrEP in Thailand to a) assess study feasibility and acceptability, and b) explore the potential impact on PrEP adherence.

We are submitting this protocol for IRB approval of Aim 2 of the study. We have chosen not to amend the Aim 1 protocol to be consistent with the procedures followed by our collaborating university in Thailand.

UNC will rely on the Duke Campus IRB for their role in this study. Co-investigators from UNC include Drs. Lisa Hightow-Weidman and Kathryn Muessig. They will assist the mPIs (Drs. LeGrand and Songtaweesin) with data interpretation, manuscript preparation and dissemination of study findings.

Please note that the app built on the **CHARGE** platform is called **P3-T** based on findings from Aim 1. It will henceforth be referred to as P3-T.

## 3. Participant Population

3.1 List and describe the proposed participant population(s). Include the expected number of participants in each population.

**Aim 2, Pilot RCT:** ~60 YMSM. Inclusion criteria: male sex at birth, self-identify as MSM, ages 16-24, plan to start PrEP in next 14 days, able to speak and read Thai, and own an Android or iOS smartphone. Exclusion criteria: Currently participating in another experimental PrEP adherence intervention, plan to move out of Bangkok in the next 6 months, unable to be consented due to an active substance use or psychological condition.

## 4. Description of Activities

4.1 Describe the study activities and how long each activity will take. If the study involves observation, describe the setting and events to observe.

**Aim 2:** Conduct a pilot study of P3-T with 60 YMSM newly starting PrEP in Bangkok, Thailand to a) assess study feasibility and acceptability, and b) explore the potential impact on PrEP adherence.

## **Study Activities:**

All study activities will be conducted at TRC-ARC in Bangkok, Thailand.

Baseline Study Visit: After participants are consented, they will complete a baseline web-based computer-assisted self-interviewing (CASI) survey that includes questions about sociodemographic characteristics, factors related to PrEP adherence, sexual risk, STIs and potential outcome mediators and moderators. Next, participants will be randomized in a 1:1 ratio into the P3-T arm or standard of care (SOC) study arm. P3-T arm: Study staff will help the participant download and install the P3-T app on the participant's phone and provide a guided tour of the app. Participants will be encouraged to explore all components of the app and use it routinely. Study staff will also inform P3-T arm participants about SOC services available to them at the clinic. SOC arm: Study staff will inform participants of SOC services available to them at the clinic. Services include individualized, youth-focused PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and at visits every 3 months after that. Study staff will also provide participants with written or online materials/resources that provide information about taking PrEP. The baseline study visit is expected to take approximately 2½ to 3 hours.

Follow-up Study Visits (3 and 6 months): All study participants will complete follow-up CASI surveys at 3 and 6 months. Individuals in the P3-T arm will answer additional survey questions about app usability and satisfaction at the 3-month follow-up. CASI data at all time points will be linked for each individual based on study ID number (SID). All participants will have their blood drawn via venipuncture at 3 and 6 months for collection of dried blood spots (DBS). All laboratory staff are certified to collect blood via venipuncture and will follow all guidelines outlined in the "WHO guidelines on drawing blood: Best practices in phlebotomy" to minimize risks associated with venipuncture blood draws. Participants will have 2mL of blood drawn from their arm or the top of their hand at each follow-up visit. The total amount of blood drawn during the 6-month study will not exceed 4ml. The amount of blood being drawn at each follow-up visit along with the cumulative amount of blood drawn throughout the study are considered to involve no more than minimal risk to participants. The DBS collection protocol is detailed under Attachment A. Follow-up study visits are expected to take approximately 2½ hours.

At the 3-month visit we will conduct in-depth interviews with 10 P3-T arm participants. We will purposefully sample 5 moderate/high app users (defined as usage of app at least 4x/week over the course of the trial) and 5 low/no app users (defined as usage of app <4x/week over the course of the trial). Interviews will be conducted by Thai study staff. We expect that the 3-month study visit will be 30-45 minutes longer for participants selected for in-depth interviews.

- 4.2 List here all surveys, questionnaires, structured and unstructured interview questions, focus group guides, and any other instruments. Provide a description of the type and range of questions for unstructured interviews. Compile these documents as Attachment A.
  - CASI survey: Baseline visit

The baseline survey will include questions about sociodemographic characteristics, PrEP adherence factors, sexual risk, STIs and potential outcome mediators and moderators.

CASI survey: Follow-up visits (3 and 6 months)

Follow-up surveys will include questions about sociodemographic characteristics, PrEP adherence factors, sexual risk, STIs and potential outcome mediators and moderators. Individuals in the P3-T arm will answer additional survey questions about app usability and satisfaction at the 3-month follow-up.

- In-depth interviews: 3-month follow-up visit
  - in-depth interviews will be conducted with 10 P3-T arm participants. We will purposefully sample 5 moderate/high app users (defined as usage of app at least 4x/week over the course of the trial) and 5 low/no app users (defined as usage of app <4x/week over the course of the trial or those participants who were initially high users but usage was not sustained over the full 3 months). The interview will ask participants about their experience and impressions of the app, how they used it, and how it may have impacted their behaviors during the 3-month intervention period. CASI survey data collected at baseline, 3 and 6 months will be linked with interview data for these participants.

| _ | $\mathbf{r}$ | | | | • | 4 | | | | 4 |
|-----------|--------------|---|------------|----|---|---|---|---|---|---|
| <b>7.</b> | R | • | <b>~</b> 1 | rı | | t | m | Δ | n | t |

Resource: Guide on Recruitment.

5.1 Describe the procedures for recruiting potential participants.

Study staff at TRC-ARC will discuss the study with YMSM who are initiating PrEP at their sites. Counselors will approach potential study participants to assess their interest in joining the study. Those interested in participating will be screened for eligibility. We will also use social media advertising to recruit participants.

5.2 Check all the recruitment methods that apply and provide text and or scripts for each method.

| | Introductory letter or e-mail messages |
|-------------|---------------------------------------------------------------|
| | Flyers/posters |
| | Newspaper ads |
| $\boxtimes$ | Text for social networking sites or other on-line recruitment |
| $\boxtimes$ | Script(s) for personal contact |
| | Other. Please describe: |

All scripts and text will be translated into Thai and back-translated into English by the Thai study team.

#### Script for personal contact

| Hello, | |
|---|---|
| My name is | . Thank you for your interest in the P3-T research study we are conducting at |
| TŘC-ARC. | |

P3-T is an app for young men who have sex with men (YMSM) who are starting PrEP for HIV prevention. The app helps YMSM create tailored strategies for taking your meds daily and tracks how often you take them, provides information about PrEP and sexual health, and you can anonymously connect with other YMSM on PrEP.

The P3-T research study is looking for YMSM to help test it! The purpose is to see if using an app helps people take their PrEP more regularly. Participation in the P3-T study is six months long and involves 3 study visits: an enrollment visit and follow up visits at 3 and 6 months. Participants complete a survey at every study visit and give a blood sample at the 3- and 6-month visits. The study will also involve daily use of the intervention materials (about 5-10 minutes) for the first three months of the study period. Since this is a randomized study, some people will get the app and some will not.

All participants will earn \$XX for each study visit they complete. Those who get the app may earn additional money. They can earn up to \$XX based on their app use. And some app users will be selected to complete an exit interview at the 3-month visit and can earn an addition \$XX for participating. Are you interested in participating in the P3-T study?

#### If no, not interested in participating:

Thank you for your time. One last thing - if you know of other YMSM who might be interested in this research study, please tell them to contact us. Thank you!

### If yes, interested in participating:

Great! In order to find out if you are eligible, you will need to take a brief study eligibility screener. After you take the screener, I will let you know if you are eligible for the study and schedule you for your enrollment visit. Would you like me to screen you for study eligibility now?

#### If yes, interested in screening now:

Okay, let's begin. [Script for consent to be screened will be read (see RCT Eligibility Screening Form)]. If individual consents to be screened, the screener will be administered. If they do not consent, they will be thanked for their time. If screened and ineligible, they will be told that they do not meet the study eligibility criteria and will be thanked for their time.

If eligible, study staff will explain the study procedures in detail. If they are still interested in participating, they will be scheduled for their enrollment/baseline visit. They will also be asked to tell other YMSM who might be interested in this research study to contact us.

#### If no, not interested in screening now:

Okay, can we schedule a more convenient time for you to complete the brief screener either in person or over the phone? [A time to complete screener will be scheduled].

#### Social media advertisement text

- Ready to start PrEP? Think you will need support for taking your pills? We are looking for young gay
  and bi men for a study that is testing an app to support PrEP adherence. Contact us at xxxx for more
  information!
- Ready to start PrEP? Worried you will forget to take your pill every day? We've got an app that may help. Take part in the P3-T Research Study and help us test the app! Contact us at xxxx for more information!
- We're looking for young gay and bi men between 16-24 years of age for a study that is testing a PrEP adherence app. Contact us at xxxx for more information! Contact us at xxxx for more information!
- We are looking for young HIV negative men who have sex with men (MSM) for a study that is testing an app to support PrEP adherence. Contact us at xxxx for more information!
- We're looking for young people to help us test out a new PrEP adherence app. You may be eligible if you are between the ages of 16-24 and a gay or bisexual man. Contact us at xxxx for more information!
- 5.3 Describe the process for screening participants prior to enrollment in the study. Include screening instruments in Attachment A. Explain what will happen to any information collected during screening for participants who are not chosen to join the study and for those who are chosen.

Aim 2: Individuals will be screened for eligibility in-person. An online RCT Eligibility Screening Form has been developed using Qualtrics software. For individuals interested in the study, the RCT Eligibility Screening Form can be administered by study staff or completed by the individual. The RCT Eligibility Screening Form will include questions that determine if an individual meets the RCT inclusion criteria. Individuals assessed as ineligible for the study will have the reason(s) for ineligibility recorded in an online Screening Log developed using Qualtrics. (Note to IRB: We do not provide this info to prevent them from knowing the criteria, thus potentially rescreening as eligible.) Individuals who are eligible but decline to participate will be asked if they are willing to provide their reason for declining participation; responses will be logged in the Screening Log. For individuals who are ineligible or decline to participate in the study, no personally identifying information will be recorded in the Screening Log. (Note to IRB: We will retain these data –without identifiers– so that we can create our CONSORT diagram for publication.) For those eligible and interested in participating in the study, we will collect the individual's name and contact information including phone number(s), email address(es), and social media contacts on the individual's Screening Form. These data will not be linked to other study data. When study accrual ends, study staff will obliterate the name and contact information for all individuals who were eligible and interested in study participation, but did not consent to participate in the study.

### 6. Risks of Harm

## Risks of Harm, Part 1: The Research Topic

6.1 If the research questions might upset or distress participants, please discuss.

It is possible that the study may precipitate emotional discomfort and/or an emotional response when participants answer questions about potentially sensitive topics such as sexual identity, sexual behavior, PrEP use and medication adherence. Further, participants may feel embarrassed about discussing sensitive issues.

6.2 Describe strategies to mitigate the risks.

All participants will be told during the informed consent process that their participation is voluntary and that they can choose to stop participating at any time without any penalty or loss of any benefit to which they might otherwise be entitled and that discontinuation of study participation is in no way related to being able to receive care or services at the study sites.

To minimize harm, participants are not required to answer any questions or provide any information that they do not wish to provide. They are also not required to use any features of the app that they do not wish to use (P3-T arm).

Based on our experiences using similar data collection methods with YMSM, the likelihood and seriousness of the risk of emotional discomfort and/or an emotional response is minimal and we will strive to create a safe and comfortable environment for all study participants.

To also minimize the risk of participants feeling uncomfortable about answering personal survey questions, we will use Computer-Assisted Self Interviewing (CASI) methods for all study surveys. Using CASI, participants read survey questions on a laptop, tablet or mobile phone and use a mouse click/keyboard/touchscreen to input the answers themselves. Study staff will be available to assist participants with questions or technical difficulties with the CASI. Participants will also be able to refuse to answer any question that makes them uncomfortable.

While participants will be informed that they may refuse to answer any questions at any time, responses or reactions to certain questions may indicate distress on the part of the participants. If at any time during the study, a participant divulges to study staff that he is at risk for harm, including but not limited to being abused or experiencing violence, if harm is suspected or likely, or if the participant states he is suicidal/homicidal, measures will be taken to ensure his safety locally. Reporting will be made as appropriate to the situation and the legal statutes, and referrals will be provided for appropriate support, counseling, or treatment resources.

#### Risks of Harm, Part 2: Physical Harm or Discomfort

6.3 If there are any risks of physical harm or discomfort, please describe.

The risks of drawing blood via venipuncture include discomfort at the site of puncture, a small risk of bruising and fainting, and a rare risk of infection.

6.4 What are the steps to mitigate the potential risks?

All laboratory staff are certified to collect blood via venipuncture and will follow all guidelines outlined in the "WHO guidelines on drawing blood: Best practices in phlebotomy" to minimize risks associated with venipuncture blood draws. Participants will have 2mL of blood drawn from their arm or the top of their hand at each follow-up visit. The total amount of blood drawn during the 6-month study will not exceed 4ml. The amount of blood being drawn at each follow-up visit along with the cumulative amount of blood drawn throughout the study are considered to involve no more than minimal risk to participants.

6.5 Are there people who should be excluded from the study because of the potential risks?

No

## Risks of Harm Part 3: Risks Associated with Information that Identifies Participants

This part addresses the collection of direct identifiers such as names and email addresses, and the collection of other information that could be used to deduce the names of research participants.

Images of participants' face are considered direct identifiers; currently audio-recordings are not.

There are four sections to this part: Recruitment, Data Collection and Storage, Data Protection Plan, and Reporting.

#### 1. Recruitment

6.6 If individually identifiable information is needed to contact and recruit participants, for example, email addresses, describe the identifiers, and explain how the information will be collected and what will happen to the identifiers after the recruitment process is complete.

We anticipate that most recruitment will occur in-person. Study staff will discuss the study with individuals who show up in person for services at the study sites and express interest in the study or may meet study eligibility criteria. Recruitment may also occur over the phone. Individuals who see a social media ad or hear about the study another way may call study staff; study staff will discuss the study with these individuals. Therefore, no identifiable information will be needed to contact and recruit participants.

| 2. Data Collection an | d Storage | | | | | | |
|---|---|---|---|---|---|---|---|
| 6.7 Do you plan to collect participants' responses? data are considered identification. | Note: If you | | ` | | | | he |
| □ No<br>⊠ Yes | | | | | | | |
| TC 1 '1 41 1' | 1 | *11 | <br> | TC 1 | , 1 | . 1 . | |

If yes, describe the direct identifiers you will associate with participants' responses. If relevant, describe data you will collect that could be used by someone with knowledge about the study population to deduce someone's identity. Explain why it is necessary to collect identifiers.

All study data will be stored on a centrally provisioned Duke Box folder with the name: \PROJECT\_CHPIR\_THAI-R21.

Aim 2: Direct identifiers will include full names (RCT Eligibility Screening Form for those eligible & Informed Consent for study participation); email address(es), phone number(s), and social media contacts (RCT Eligibility Screening Form for those eligible). Contact information for those eligible will be collected through the RCT Eligibility Screening Form created in Qualtrics. These direct identifiers are needed to ensure the study team's ability to contact eligible individuals about the enrollment visit or follow-up study visits. Full names are needed as part of informed consent for study participation and will be collected on paper forms. Individuals enrolled in the study will be assigned a study ID number (SID). A linking file will be created that includes SIDs and full participant names. The RCT Eligibility Screening Form files will be downloaded from Qualtrics and stored in a secure Duke Box folder separate from the secure Duke Box folder that contains the linking file. Informed Consent forms for study participation will be scanned to a password-protected and encrypted computer and subsequently transferred to a secure Duke Box folder separate from the secure Duke Box folder that contains the linking file. Consent forms will be destroyed after a scanned copy has been uploaded to Duke Box. Access to the RCT Eligibility Screening Form and Informed Consent files will be limited to study staff who need contact participants about enrollment or study visits and/or to verify completion of Informed Consent. Access to the linking file will be limited to the mPIs and study Project Coordinators. Only SIDs will be used to identify study participant data (e.g. survey data, lab results indicating intracellular levels of tenofovir-diphosphate (TFV-DP) and emtricitabine triphosphate (FTC-TP), in-depth interview transcripts, etc.)

| 6.8 Would the inadvertent disclosure of identifiable data place participants at risk of h | arm? |
|---|---|
| ☐ No<br>⊠ Yes | |

#### If no, skip Section 3. Data Protection Plan, and go to Section 4. Reporting.

If yes, describe the specific harms that could occur if individually identifiable data were disclosed in the box below. Also, complete Section 3. Data Protection Plan.

The identification of participants' sexual behaviors or sexual minority status could have negative social and economic consequences.

#### 3. Data Protection Plan

If your participants could be harmed by an inadvertent release of identifiable data, the data are classified as sensitive.

Responses to the questions in this section will assist IRB reviewers, and are needed by the Duke University Information Security Technology Office (ITSO) to assess your data protection plan. ITSO will review the data protection plan to ensure appropriate measures are in place to protect data. The IRB will send the entire protocol to ITSO.

Please review the <u>Developing Data Protection Plans</u> for a list of best practices and ITSO recommendations.

6.9 Who is your departmental or unit IT contact?

Patrick Daniels

6.10 Who is responsible for data security, including upgrades?

Patrick Daniels

6.11 Where will you store data? If data will not be stored on an ITSO-approved storage medium, where will they be stored?

Qualtrics (BAA), secure Duke Box folders, locked storage cabinet/locked office at study sites (paper copies of Informed Consent Forms only before they are scanned, uploaded to Duke Box, and destroyed).

6.12 How will transfers of data from the data collection site to the data storage medium described above be handled?

Informed Consent Forms for study participation:

The Thai study team will scan paper consent forms to a password-protected & encrypted computer and transfer the scans to the appropriate secure Duke Box folder. Once successfully transferred to Duke Box, the scanned files will be deleted from the computer and paper consent forms will be destroyed.

RCT eligibility screening and surveys (baseline, 3 months, 6 months):

These will be administered using Qualtrics. The Duke study team will download these documents from Qualtrics on a password-protected and encrypted computer and transfer the files to their appropriate secure Duke Box folder. Once successfully transferred to Duke Box, the files will be deleted from the computer.

#### Lab results:

Results from the analysis of DBS from the Program for HIV Prevention and Treatment (PHPT) Research Unit at Chiang Mai University will be sent via email in a password protected document. The results will only be identified by SID as the samples sent the lab will only be identified by SID. One received, the Thai mPI will download the document on a password-protected and encrypted computer and transfer the files to their appropriate secure Duke Box folder. The blood samples used to create DBS will be stored at Chulalongkorn University lab and destroyed 3 years after study completion. DBS stored at PHPT will be destroyed 3 years after study completion.

Note to IRB: Regarding HIV status- participants are tested for HIV prior to collection of blood for drug levels. The test performed as part of our study does not test for HIV. However, if we learn that anyone tests positive for HIV while participating in the study, they will be immediately offered care/treatment by TRC-ARC and will be discontinued from our study.

Linking File:

The linking file will be housed in a secure Duke Box folder separate from all study data. The Thai mPI or study coordinator will be responsible for updating the linking file when a new participant enrolls in the study (i.e., full name of participant assigned to SID). The updated version of the linking file will be saved in the secure Duke Box folder. 6.13 Do you plan to create a key linking unique identifiers participants' responses? If yes, describe the key, where it will be stored, how it will be protected, and who will have access to it (list by name). The linking file will contain SIDs and full participant names. The file will be stored in a secure Duke Box folder separate from all study data. Access will be limited to mPIs (Sara LeGrand, Wipaporn Songtaweesin) and study project coordinators (Duke- Shashika Bandara, TRC-ARC-Nuttawut Teachatanawat). 6.14 Who will have access to the identifiable data? (List by name.) Access will be limited to mPIs (Sara LeGrand, Wipaporn Songtaweesin) and study project coordinators (Duke- Shashika Bandara, TRC-ARC- Nuttawut Teachatanawat). 6.15 How will access to the identifiable data be controlled? Only the identified individuals will have access to the secure Duke Box folder. 6.16 Where will data be analyzed? Who will perform the analysis? The data will be analyzed at Duke and TRC-ARC on a password protected & encrypted computer. All analysis files will be saved on a secure folder in Duke Box. Analyses will be conducted by the Duke mPI (LeGrand), project coordinator (Bandara), statistician (TBD), and Thai mPI (Songtaweesin). 6.17 If the data need to be de-identified, what are the plans for de-identifying data? Describe when in the process the data will be de-identified and identify who will do the de-identification. In some cases, a third-party broker may be required to de-identify the data. N/A 6.18 Will you apply for a Certificate of Confidentiality to protect the data from subpoena, if for example, you have identifiable data about illegal drug use or unlawful behavior? Already issued by NIH 6.19 Is a non-Duke entity giving you Protected Health Information? If yes, please provide the data disclosure agreement as an attachment to this form. No Yes 6.20 If you have entered into a data use agreement that specifies a data destruction date, what is the data destruction date? N/A

4. Reporting

Yes

6.21 Will you use participants' names in your research reports?

13

| 6.22 If no, based on your research topic, setting, and reported characteristics of your participants, could their identities be readily deduced? |
|---|
| ☐ Yes<br>☑ No |
| 7. Benefits |
| 7.1 Describe any anticipated direct benefits of the research for individual participants. If the research provides no direct benefits to participants, state "None." |
| Individual participants may benefit through increased PrEP adherence and reduced risk for HIV acquisition. |
| 8. Compensation |
| Guide: The Guide to Compensating Research Participants provides more information on different methods of compensation, including drawings and lotteries, and compensation restrictions. |
| 8.1 Will participants receive gifts, payments, or tokens of appreciation? |
| No Yes |
| If yes, please describe: |
| All participants will earn \$20 for each study visit they complete (baseline, 3 months, 6 months). P3-T arm participants can earn up to \$15 based on their app use. This is a component of the behavioral economics feature of the app. Each user's "bank account" is seeded with \$1.50 and they can earn an additional \$13.50 for daily app use (total=\$15). Users are awarded \$0.15 for engaging with the app each day, but lose \$0.05 for each day they do not engage with the app. Accounts balances will never go below \$0. However, if they reach \$0 and begin using the app again, their balance can increase above \$0 (increase \$0.15 per each day of use, but can still lose \$0.05 for each day of non-use. P3-T arm participants selected for an in-depth interview at the 3-month visit will earn \$20 for participating. |
| 8.2 If participants will receive payment, under what conditions will they receive partial or no payment? |
| They will not receive a payment for any study visits missed or if they are not invited or otherwise do not complete an in-depth interview. App use payments will only be made at a follow-up study visit, so if they do not attend one, they will not receive their app use payment. |
| 9. Photographs, Videos, and Audio-recordings |
| 9.1 If participants will be photographed or video-recorded, explain why the images (photos or videos) are necessary to answer the research question. The IRB will consider approving the collection of photographs or videos only |

if they are necessary to answering the research question.

N/A

No No

| Il participants be audio-recorded either individually or in groups? Audio-recordings of groups is allowed y if all participants in the group have given their explicit permission to be recorded. |
|---|
| <ul><li>No</li><li>Yes</li></ul> |
| If yes, what happen to the recordings? |

• Clarify whether they will be destroyed after they have been transcribed.

• If they will be saved for further research and education, explain where the recordings will be stored and how they might be used.

Audio recordings of in-depth interviews will be permanently destroyed within 6 months of study completion. Until then, they will be stored in a secure folder in Duke Box. They will be kept in case there is a need to verify transcriptions or fill in missing data from transcriptions (e.g., transcriptionist could not understand participant).

**Guide**: For guidance about when photographic releases are needed and to see sample release language, go to the Guide for Releases for Images and Recordings.

#### 10. Informed Consent Process

The informed consent process involves two parts:

- 1) The process of sharing information about the research study and
- 2) The documentation (a signed consent form or an audio- or video-recorded statement by the research participant) that the process took place
- Please see information below about request for waiver of written consent to screen participants for study activities and waiver of parental permission/consent for minors.

There will always need to be a process for sharing information about the research study with prospective participants. In some circumstances it may be appropriate to request that the IRB waive the requirement to document consent.

If one or more of the following is true, the IRB may be able to waive the requirement to document consent. Please check any that apply to the study.

Participants do not read and write. (If there is a risk of harm, a third-party witness will be present.)

Data will be collected on-line. Participants will have the option to "click" to the survey if they would like to take part in the study.

The study data will be collected through a telephone interview. If appropriate, provide a copy of the consent process for participant's reference.

Participants will complete a mailed survey. Prepare a cover letter that includes all the elements of informed consent. People who wish to take part will return the survey; thereby, demonstrating their consent. They do not need to sign a consent form.

The research will take place in settings where written consent is considered disrespectful or in settings in which asking people to sign a document would cause distress.

The primary risk to participants is a breach of confidentiality and a signed consent form or audio-recorded statement would be the only documented link between individuals and their participation in the study. (Example: a study about people with HIV/AIDS.)

#### Waiver of written consent to screen participants for study activities:

An online consent process for eligibility screening for study activities is proposed. The introduction to the online screener includes all the required elements for consent (45 CFR 46.116). No identifying information on volunteers is recorded during the online screening until a participant is determined eligible (i.e., by marking "I do consent to be screened for eligibility in the online screener). Therefore, there will be no identifying link of who agreed to be screened or not screened for the study. In addition, the screening presents minimal risk to participants and involves no procedures that would require written consent outside of a research context. Under these conditions the IRB is authorized to modify the requirements to obtain a signed consent form for some or all subjects (45 CFR 46.117 [c]).

#### Waiver of parental permission/consent for minors (ages 16-17):

We request that the Campus IRB grant a waiver of parental consent to participate in this research study for youth participants who are 16 to 17 years of age.

- This study involves no more than minimal risk to the subjects.
- A waiver of parental permission/consent will not adversely affect the rights and welfare of the subjects. In fact, failure to waive parental permission/consent may have adverse effects as sexual minority youth often have not disclosed their sexual minority status to their parents and requiring consent would require unwanted disclosure that may have negative emotional, social, financial, and/or physical consequences.
- The research could not practicably be carried out without the waiver. A requirement for parental permission/consent in this type of study could not only affect a person's willingness to participate but could also potentially impact the ability of researchers to engage in this type of research with sexual minority youth. Without a waiver, we would be challenged by selection bias as we would only be able to recruit youth whose parents are both aware of and comfortable with their sexual orientation. Commonly these youth have explored their sexual orientation without their parents' knowledge as the youth struggle with issues of disclosure and its consequences within the social, religious, and economic context of their families. Additionally, contacting a parent/legal guardian could constitute a breach of confidentiality for these minor subjects and could potentially put some youth at risk for abuse or ousting from the home if parents/legal guardians are not aware of the subject's sexual minority status or sexual risk behaviors. If the purpose of requiring parental permission/consent as stated in CFR is to protect the minor subject, then requiring parental permission/consent for youth in these circumstances is not a reasonable requirement.

#### Waiver of written consent at 3 and 6 month study activities:

The project is requesting a waiver to document informed consent for the follow-up visits at 3 and 6 months after initial consent is signed. This request is from the local Thai team and IRB.

This is standard practice approved by the Thai IRB and is standard practice for all locally and internationally funded clinical trials at the research site. The Thai team has told the research team that Thailand is a much more verbal rather than written communication culture and they feel that for local settings it is probably more helpful for participants to be verbally reminded what they will be tested for that day (this is standard practice even outside research) and to confirm this has been done we can make a note that they have provided verbal consent in the electronic medical records and track in REDCap for research purposes.

#### **REFERENCES:**

- 1. van Griensven F, Thienkrua W, McNicholl J, et al. Evidence of an explosive epidemic of HIV infection in a cohort of men who have sex with men in Thailand. AIDS 2013;27:825-32.
- 2. UNICEF. Situational analysis of young people at high risk of HIV exposure in Thailand2014.
- 3. Grant RM, Anderson PL, McMahan V, et al. Uptake of pre-exposure prophylaxis, sexual practices, and HIV incidence in men and transgender women who have sex with men: a cohort study. The Lancet infectious diseases 2014;14:820-9.
- 4. Grant RM, Anderson PL, McMahan V, et al. Results of the iPrEx open-label extension (iPrEx OLE) in men and transgender women who have sex with men: PrEP uptake, sexual practices, and HIV incidence. Oral Abstract Session # TUAC0105LB presented at AIDS 2014 in Melbourne, Australia, July 20-25, 2014 Abstract available at: <a href="http://pagaids2014org/abstractsaspx?aid=11143">http://pagaids2014org/abstractsaspx?aid=11143</a> July 20-25, 2014.
- 5. Grant RM, Lama JR, Anderson PL, et al. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. The New England journal of medicine 2010;363:2587-99.
- 6. Amico KR, Stirratt MJ. Adherence to preexposure prophylaxis: current, emerging, and anticipated bases of evidence. Clin Infect Dis 2014;59 Suppl 1:S55-60.
- 7. Anand T, Nitpolprasert C, Trachunthong D, et al. A novel Online-to-Offline (O2O) model for pre-exposure prophylaxis and HIV testing scale up. J Int AIDS Soc 2017;20:1-11.
- 8. mHealth: New horizons for health through mobile technologies. 2011. at <a href="http://www.who.int/goe/publications/goe/mhealth-web.pdf">http://www.who.int/goe/publications/goe/mhealth-web.pdf</a>.)
- 9. Ramirez-Valles J. The protective effects of community involvement for HIV risk behavior: a conceptual framework. Health education research 2002;17:389-403.
- 10. Ramirez-Valles J, Kuhns LM, Campbell RT, Diaz RM. Social integration and health: community involvement, stigmatized identities, and sexual risk in Latino sexual minorities. Journal of health and social behavior 2010;51:30-47.
- 11. Baranowski T, Baranowski J, Cullen K, et al. Squire's Quest! Dietary outcome evaluation of a multimedia game. American journal of preventive medicine 2003;24:52-61.

- 12. Brown SJ, Lieberman DA, Germeny BA, Fan YC, Wilson DM, Pasta DJ. Educational video game for juvenile diabetes: results of a controlled trial. Medical informatics = Medecine et informatique 1997;22:77-89.
- 13. Lieberman D. Interactive video games for health promotion: Effects on knowledge, self-efficacy, social support, and health. In: Street R, ed. Health Promotion and interactive technology: Theoretical applications and future directions. Mahwah, NJ: Lawrence Erlbaum Associates; 1997:103-20.
- 14. Kato PM, Cole SW, Bradlyn AS, Pollock BH. A video game improves behavioral outcomes in adolescents and young adults with cancer: a randomized trial. Pediatrics 2008;122:e305-17.
- 15. McGonigal J. Reality is Broken: Why Games Make Us Better and How They Can Change the World. New York: The Penguin Press; 2012.

## Attachment A

All documents will be translated into Thai and back-translated into English by the Thai study team.

Contents include:

- 1. CASI Survey Baseline
- 2. CASI Survey 3-month- P3-T arm
- 3. CASI Survey 3-month- SOC arm
- 4. CASI Survey 6-month
- 5. DBS Collection Protocol
- 6. RCT Eligibility Screening Form

## **CASI Survey Baseline**

## **P3-T RCT Baseline**

Instructions for study staff member:

- Tell the participant:
  - At this time, we would like you to complete the baseline survey
  - Let me know if they have any trouble understanding any of the questions. I will help to clarify the question(s) for you.
  - Please leave the browser open once you have completed the survey and let me know that you are finished.
  - Don't worry I will not be able to access your survey answers with the browser left open.
- After these instructions have been given, enter and re-enter the participant's study ID and participant code below and hand the computer to the participant to complete the survey.

**Enter the participant's Study ID (3 digits)** 

Re-enter the participant's Study ID (3 digits)

Participant code is the first letter of the participant's first name and the two digit day of their birth.

ex: first name: Jane; Birthdate: February 05 = J05

Re-enter the Participant Code

#### ID: 93

Thank you for participating in the P3-T study! The purpose of the study is to test a PrEP adherence app for young gay and bi men who are starting PrEP. As part of the P3-T study, you will take three surveys: one today, one at your follow up appointment in 3 months, and one at your follow up appointment in 6 months.

Try to answer every question as best you can. If you need help, please ask the study staff.

| Your answers will be used only for research purposes. Let's get started! |
|---|
| Age |
| ID: 94 |
| First, tell us a little about yourself. |
| Shortname / Alias: age |
| ID: 95 |
| What is your age? |
| Location |
| Shortname / Alias: postal |
| ID: 100 |
| What is the postal code for the location where you primarily live?* |
| What is the postal code for the location where you primarily live?* |
| What is the postal code for the location where you primarily live?* |
| What is the postal code for the location where you primarily live?* ——————————————————————————————————— |
| Education |
| Education Shortname / Alias: schoollevel |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* ( ) None, no formal schooling |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* ( ) None, no formal schooling ( ) Primary school |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* ( ) None, no formal schooling ( ) Primary school ( ) Lower secondary school |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* ( ) None, no formal schooling ( ) Primary school ( ) Lower secondary school ( ) Upper secondary school |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* ( ) None, no formal schooling ( ) Primary school ( ) Lower secondary school ( ) Upper secondary school |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* () None, no formal schooling () Primary school () Lower secondary school () Upper secondary school () Higher education |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* () None, no formal schooling () Primary school () Lower secondary school () Upper secondary school () Higher education |
| Education Shortname / Alias: schoollevel ID: 108 What is the highest level of school that you have completed?* () None, no formal schooling () Primary school () Lower secondary school () Upper secondary school () Higher education Employment, Income |

Are you currently employed?\* ( ) Yes

20

| ( ) No |
|---|
| Logic: Hidden unless: #12 Question "Are you currently employed?" is one of the following answers ("Yes") |
| Shortname / Alias: employedhours |
| ID: 110 |
| Are you employed full-time or part-time? Part-time means that you work less than 35 hours per week during most weeks.* ( ) Full time |
| ( ) Part time |
| ( ) Decline to answer |
| Shortname / Alias: income_30d |
| ID: 564 |
| How much money did you make altogether during the past 30 days?* |
| ( ) Don't know |
| Shortname / Alias: incomelevel ID: 111 |
| How would you describe your income level?* ( ) Low income |

- () Middle income
- () High income

# Food, Shelter

Shortname / Alias: cutmeal

ID: 112

In the past 3 months, how often did you or your family have to cut meal size or skip a meal because there was not enough money for food?\*

- () Almost every week
- () Several weeks but not every week
- () Only a few weeks

| ( ) Did not have to skip or cut the size of meals |
|---|
| ( ) Decline to answer |
| Shortname / Alias: shelter |
| ID: 113 |
| In the past 3 months, have you spent at least one night (check all that apply):* [] In a shelter? |
| [] In a public place not intended for sleeping (e.g., bus station, car, abandoned building)? |
| [] On the street or anywhere outside (e.g., park, sidewalk)? |
| [] Temporarily doubled up with a friend or family member? |
| [] In a temporary housing program? |
| [] In a welfare or voucher hotel/motel? |
| [] In jail, prison, or a halfway house? |
| [] In drug treatment, a detox unit, or drug program housing? |
| [] In a hospital, nursing home, or hospice? |
| [] I have not spent a night in any of the above places. |
| [ ] Decline to answer |
| Arrest Incorporation |
| Arrest, Incarceration |
| Note to IRB: We included the arrest/incarceration questions because these situations are not uncommon among our target population, largely due to arrests due to substance use. Because arrests and/or incarceration can have impact on PrEP adherence, we think it is important to know if these events have occurred |

Logic: Show/hide trigger exists.

Shortname / Alias: arrested

ID: 114

Have you ever been arrested?\*

() Yes

( ) No

Logic: Hidden unless: #18 Question "Have you ever been arrested?" is one of the following answers ("Yes")

Shortname / Alias: arrested3mo

| ID: 115 |
|---|
| Have you been arrested in the past 3 months?* |
| () Yes |
| ( ) No |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: jail |
| ID: 116 |
| Have you ever been put in jail, prison or juvenile detention?* |
| () Yes |
| ( ) No |
| Logic: Hidden unless: #20 Question "Have you ever been put in jail, prison or juvenile |
| detention?" is one of the following answers ("Yes") |
| Shortname / Alias: jail3mo |
| ID: 117 |
| Have you been put in jail, prison or juvenile detention in the past 3 months?* ( ) Yes |
| ( ) No |
| Sexual Identity and Awareness |
| ID: 565 |
| The following questions ask about your sexual identity and relationship status. |
| The following questions ask about your sexual identity and relationship status. |
| Please answer to the best of your ability. |
| Shortname / Alias: sexualid |
| ID: 102 |
| What is your current sexual identity?* ( ) Gay, homosexual, same gender loving |
| () Bisexual |
| () Queer |
| ( ) Straight or heterosexual ( ) Other, specify::* |

| Shortname / Alias: familyawareness |
|---|
| ID: 103 |
| How many of your immediate family members know about your sexual identity? "Immediate family members" includes family members you live with or family members you interact with often. If you do not have regular contact with any family members, please select "Does not apply".* () None () Some, but less than half |
| ( ) About half ( ) More than half |
| ( ) All |
| ( ) Does not apply |
| ( / = ·· • |
| Shortname / Alias: peerawareness |
| ID: 104 |
| How many of your peers know about your sexual identity? "Peer" includes your friends, co-workers, and schoolmates.* () None () Some, but less than half () About half () More than half () All |
| Relationships |
| Shortname / Alias: relationship |
| ID: 118 |
| How do you define your primary relationship status?* ( ) Single, not currently dating ( ) Single, casually dating ( ) In a relationship ( ) Married or other legal commitment |

**Page entry logic:** This page will show when: #25 Question "How do you define your primary relationship status?" is one of the following answers ("In a relationship","Married or other legal commitment")

## **Sexual Health Priorities with Partner**

ID: 566

People have different sexual health priorities. For example, some people prioritize staying HIV-negative; others want to have as much fun as possible with their partners; others want to feel as close and connected to their partners as possible.

For these next questions, we are interested in you and your primary romantic partner's sexual health priorities.

Shortname / Alias: shpriorities scale

ID: 569

Thinking about you and your partner's sexual health priorities, please indicate the extent to

which you agree or disagree with the following statements.\*

| | Strongly<br>Agree | Agree | Disagree | Strongly<br>Disagree |
|---|---|---|---|---|
| I feel like my partner and I are "on the same page" in terms of the decisions we make about sexual health and risk | () | () | () | () |
| When it comes to sexual decision-making, I feel like my partner and I are "of the same mind" | () | () | () | () |
| Sometimes I<br>feel like my<br>priorities for<br>my sexual<br>health are | () | () | () | () |

| incompatible<br>with my<br>partner's<br>goals | | | | |
|---|---|---|---|---|
| I'm confident that my partner and I generally share the same priorities when it comes to sexual health | () | () | () | () |
| Making sexual health decisions with my partner can be difficult because we have different priorities | () | () | () | () |

| Ce | II P | hon | e. I | nteri | net | Use |
|--------------|------|-----|------|-------|-----|-----|
| $\mathbf{-}$ | | | | | 101 | |

ID: 120

Now, we'd like to ask you about your cell phone and internet use.

Logic: Show/hide trigger exists.

Shortname / Alias: techuse

ID: 121

## Which of the following devices do you own? (Check all that apply)\*

- [] Cell phone (basic mobile phone for calling or texting; does not have internet access, apps, or a touch screen)
- [] Smartphone (advanced mobile phone with internet access, apps, and a touch screen)

| [ ] Desktop computer | |
|---|---|
| [ ] Laptop computer | |
| [ ] Tablet computer | |
| [] E-book reader | |
| [] Fitness tracker or smart watch | |
| [] Another device, specify: | |
| Shortname / Alias: internetaccess | |
| ID: 122 | |
| How do you usually access the internet? (Check all that apply)* [] Smartphone | |
| [ ] Desktop computer | |
| [ ] Laptop computer | |
| [ ] Tablet computer | |
| [] E-book reader | |
| [] Another method, specify: | |
| Internet (cont.), Phone Plan | |
| Action: Custom Script: Script to count checkboxes and skip q if < 2 | |
| Shortname / Alias: accessrank | |
| ID: 123 | |
| Piping: Piped Values From Question 28. (How do you usually access the internet? (Check all that a | pply)) |
| How do you access the internet most frequently? (Rank your answers)*Smartphone | |
| Desktop computer | |
| Laptop computer | |
| Tablet computer | |
| E-book reader | |
| Another method, specify | |

**Page entry logic:** This page will show when: #27 Question "Which of the following devices do you own? (Check all that apply)" is one of the following answers ("Cell phone (basic mobile phone for calling or texting; does not have internet access, apps, or a touch screen)", "Smartphone (advanced mobile phone with internet access, apps, and a touch screen)")

## **Cellphone/ Smartphone Plan**

Logic: Hidden unless: #27 Question "Which of the following devices do you own? (Check all that apply)" is one of the following answers ("Smartphone (advanced mobile phone with internet access, apps, and a touch screen)")

Shortname / Alias: phoneplatform

ID: 125

| ( ) Apple (iOS) |
|---------------------|
| ( ) Android |
| ( ) Don't know |
| ( ) Other, specify: |

Logic: Hidden unless: #27 Question "Which of the following devices do you own? (Check all that apply)" is one of the following answers ("Cell phone (basic mobile phone for calling or texting; does not have internet access, apps, or a touch screen)", "Smartphone (advanced mobile phone with internet access, apps, and a touch screen)")

Shortname / Alias: phoneplan

ID: 126

#### What kind of cell phone or smartphone service do you have?\*

- () I have a prepaid account
- () I have a monthly contract
- () I'm on a shared plan
- () Don't know
- () None of the above

Logic: Hidden unless: #27 Question "Which of the following devices do you own? (Check all that apply)" is one of the following answers ("Cell phone (basic mobile phone for calling or texting; does not have internet access, apps, or a touch screen)", "Smartphone (advanced mobile phone with internet access, apps, and a touch screen)")

Shortname / Alias: phonepay

ID: 127

Who usually pays for your cell phone or smartphone plan?\*

() I do

() Someone else does

**Page entry logic:** This page will show when: #27 Question "Which of the following devices do you own? (Check all that apply)" is one of the following answers ("Cell phone (basic mobile phone for calling or texting; does not have internet access, apps, or a touch screen)", "Smartphone (advanced mobile phone with internet access, apps, and a touch screen)")

#### **Phone Disconnect**

Logic: Show/hide trigger exists

| Logic. Chewinde trigger exists. |
|---|
| Shortname / Alias: disconnect |
| ID: 128 |
| In the past year, did you ever not have access to your phone or phone service?* ( ) Yes |

Logic: Hidden unless: #33 Question "In the past year, did you ever not have access to your phone or phone service?" is one of the following answers ("Yes")

Shortname / Alias: disconnecttimes

ID: 129

How many times in the last year did you not have access to your phone or phone service?\*

- () Once
- () Twice
- () 3 to 5 times
- () More than 5 times

Logic: Hidden unless: #33 Question "In the past year, did you ever not have access to your phone or phone service?" is one of the following answers ("Yes")

Shortname / Alias: disconnectlength

ID: 130

The *last* time you did not have access to your phone or phone service, for how long did you know have access?\*

- () 1 day or less
- () 2 to 6 days
- () 1 to 4 weeks
- () More than 4 weeks

# **Internet Time, Frequency**

**Smartphone Sites** 

| Shortname / Alias: internettime ID: 131 |
|---|
| On average, how many hours per day do you spend on the internet (online) <u>outside of your school or work responsibilities</u> ?* ( ) No hours |
| ( ) Less than an hour |
| ( ) 1 to 3 hours |
| ( ) 4 to 6 hours |
| ( ) 7 to 9 hours |
| ( ) 10 to 12 hours |
| ( ) 13 to 15 hours |
| () 16 hours or more |
| Page entry logic: This page will show when: #27 Question "Which of the following devices do you own (Check all that apply)" is one of the following answers ("Smartphone (advanced mobile phone with internet access, apps, and a touch screen)") |
| Smartphone Apps |
| Shortname / Alias: phoneapps |
| Shortname / Alias: phoneapps ID: 132 |
| ID: 132 How often do you use apps on your smartphone (for example: Facebook, dating apps, banking apps, Snapchat)?* |
| How often do you use apps on your smartphone (for example: Facebook, dating apps, banking apps, Snapchat)?* ( ) More than once a day |
| How often do you use apps on your smartphone (for example: Facebook, dating apps, banking apps, Snapchat)?* ( ) More than once a day ( ) About once a day |
| How often do you use apps on your smartphone (for example: Facebook, dating apps, banking apps, Snapchat)?* ( ) More than once a day ( ) About once a day ( ) A few times a week |
| How often do you use apps on your smartphone (for example: Facebook, dating apps, banking apps, Snapchat)?* ( ) More than once a day ( ) About once a day ( ) A few times a week ( ) About once a week |

Shortname / Alias: phonesites

ID: 133

How often do you use websites or smartphone apps for the following reasons:

| Tiow often do y | Never | Rarely | Sometimes | Often |
|---|---|---|---|---|
| Make new friends | () | () | () | () |
| Chat with friends | () | () | () | () |
| Chat with family | () | () | () | () |
| Find a date | () | () | () | () |
| Meet partners for casual sex | () | () | () | () |
| Look for work opportunities | () | () | () | () |
| Track health behaviors (diet, exercise, medication management, etc.) | () | () | () | () |
| Get<br>information<br>about HIV or<br>other STIs | () | () | () | () |
| Get other<br>health or<br>medical<br>information | () | () | () | () |
| Create event reminders (take a daily pill, exercise, etc.) | () | () | () | () |

# **Internet Opinions**

Shortname / Alias: hi

ID: 145

Please indicate your agreement with the following statements:\*

| | Strongly | | | Strongly |
|---|---|---|---|---|
| | Disagree | Disagree | Agree | Agree |
| I know what health resources are available on the Internet. | () | () | () | () |
| I know how to find helpful health resources on the Internet. | () | () | () | () |
| I know how to use the Internet to answer my questions about health. | () | () | () | () |
| I know how to use the health information I find on the Internet to help me. | () | () | () | () |
| I have the<br>skills I<br>need to<br>evaluate<br>the health<br>resources I | () | () | () | () |

| - | | | | |
|---|---|---|---|---|
| find on the<br>Internet. | | | | |
| I can tell high quality health resources from low quality health resources on the Internet. | () | () | () | () |
| I feel confident in using information from the Internet to make health decisions. | () | () | () | () |
| I know where to find helpful health resources on the Internet. | () | () | () | () |

## **Health Providers**

ID: 157

Now, we are going to ask you about your health and health care decision making.

Logic: Show/hide trigger exists.

Shortname / Alias: pcp

ID: 158

| Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?* () Yes |
|---|
| ( ) No |
| Logic: Hidden unless: #40 Question "Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?" is one of the following answers ("Yes") |
| Shortname / Alias: pcpawareness |
| ID: 105 |
| How open are you about your sexual identity to your primary medical care provider?* ( ) Primary medical provider definitely does NOT know your sexual identity |
| ( ) Primary medical provider MIGHT know about your sexual identity |
| ( ) Primary medical provider PROBABLY knows about your sexual identity |
| ( ) Primary medical provider DEFINITELY knows about your sexual identity |
| Logic: Hidden unless: #40 Question "Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?" is one of the following answers ("Yes") |
| Shortname / Alias: pcptalksex |
| ID: 160 |
| How comfortable are you discussing your sexual behavior with your primary health care provider?* ( ) Very comfortable |
| ( ) Somewhat comfortable |
| ( ) Somewhat uncomfortable |
| ( ) Very uncomfortable |
| HIV Testing |
| Shortname / Alias: recenthivtest_mon |
| ID: 165 |
| When did you have your most recent HIV test? |
| Please enter the month and year. |
| Month:* ( ) January ( ) February ( ) March |

| () September |
|---|
| () October |
| ( ) November |
| () December |
| Validation: Min = 1980 Must be numeric Whole numbers only Positive numbers only Max character count = 4 |
| Shortname / Alias: recenthivtest_yr |
| ID: 166 |
| Year:* |
| Action: Custom Script: Check HIV test date not in future |
| STI Testing |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: lifetimestitest |
| ID: 170 |

Logic: Hidden unless: #45 Question "A sexually transmitted infection (STI) is an infection transmitted through sexual activity, such as syphilis, gonorrhea, chlamydia, herpes, or genital warts. Have you ever been tested for an STI that was not HIV?" is one of the following answers ("Yes")

A sexually transmitted infection (STI) is an infection transmitted through sexual activity, such as syphilis, gonorrhea, chlamydia, herpes, or genital warts. Have you ever been tested for an STI

Shortname / Alias: sti3mo

that was not HIV?\*

ID: 171

() Yes

() No

() April () May () June

() July

() August

| infections in the <u>past 3 months</u> . Please select all that apply.* |
|---|
| [] Chlamydia |
| [] Genital warts, anal warts, HPV |
| [] Gonorrhea |
| [] Hepatitis B |
| [ ] Hepatitis C |
| [] Herpes, HSV1/HSV2 |
| [ ] Syphilis |
| [ ] Urethritis |
| [] Other, please specify:: |
| [] None of these |
| PrEP Start |
| Shortname / Alias: startprep_why |
| ID: 943 |
| 15.010 |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ |
| Why have you decided to start taking PrEP? Select all that apply.* |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy [] I want to be safe and healthy |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy [] I want to be safe and healthy [] I want to have a better future |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy [] I want to be safe and healthy [] I want to have a better future [] I am having sex with multiple partners |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy [] I want to be safe and healthy [] I want to have a better future [] I am having sex with multiple partners [] I don't like to use condoms |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy [] I want to be safe and healthy [] I want to have a better future [] I am having sex with multiple partners [] I don't like to use condoms [] My partner won't use condoms |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy [] I want to be safe and healthy [] I want to have a better future [] I am having sex with multiple partners [] I don't like to use condoms [] My partner won't use condoms [] I had a previous HIV scare [] My health care provider recommended it |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy [] I want to be safe and healthy [] I want to have a better future [] I am having sex with multiple partners [] I don't like to use condoms [] My partner won't use condoms [] I had a previous HIV scare [] My health care provider recommended it [] I was recently diagnosed with an STI |
| Why have you decided to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ [] I'm having sex with or thinking about having sex with someone whose status HIV I don't know [] I want to be in control of my sexual health [] I want to reduce my anxiety around sex [] I want to increase my sexual satisfaction and intimacy [] I want to be safe and healthy [] I want to have a better future [] I am having sex with multiple partners [] I don't like to use condoms [] My partner won't use condoms [] I had a previous HIV scare [] My health care provider recommended it |

Please indicate whether you have been diagnosed with any of the following sexually transmitted
#### **PrEP Start**

Shortname / Alias: startprep primwhy

ID: 945

Piping: Piped Values From Question 47. (Why did you choose to start taking PrEP? Select all that apply.)

What was the main reason you have decided to start taking PrEP?\*

#### **PrEP Confidence**

ID: 907

We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident).

Validation: Min = 1 Max = 10

Shortname / Alias: keepappts

ID: 903

How confident are you that you will be able to...

**Keep your PrEP medical appointments:\*** 

1 \_\_\_\_\_\_ 10 or N/A

Validation: Min = 1 Max = 10

Shortname / Alias: followplan

ID: 904

Follow a plan for taking PrEP:\*

1 [ ] 10 or N/A

Validation: Min = 1 Max = 10

Shortname / Alias: atworkschool

ID: 905

| Take PrEP at work/school:* | [_] | 10 or N/A |
|---|---|---|
| Validation Min - 4 May - 40 | | |
| Validation: Min = 1 Max = 10 Shortname / Alias: onweekday | | |
| ID: 906 | | |
| Take PrEP on a weekday:* | | |
| | <u></u> | _ 10 or N/A |
| PrEP Confidence 2 | | |
| ID: 908 | | |
| We are interested in how we | u fact about the fallowing statemen | into Dioggo anguar hu |
| | ou feel about the following stateme<br>about each statement on a scale fi | |
| (totally confident). | | |
| Validation: Min = 1 Max = 10 | | |
| Shortname / Alias: onweekend | | |
| ID: 909 | | |
| How confident are you that yo | u will be able to | |
| Take PrEP on a weekend:* | | |
| 1 | | _ 10 or N/A |
| Validation: Min = 1 Max = 10 | | |
| Shortname / Alias: wfriends | | |
| ID: 910 | | |
| Take PrEP when I'm out with f | | |
| 1 | | _ 10 or N/A |
| Validation: Min = 1 Max = 10 | | |
| Shortname / Alias: prepdrinking | | |
| ID: 911 | | |
| Take PrEP when I'm drinking | | 40 |
| 1 | [] | _ 10 or N/A |

| Validation: Min = 1 Max = 10 | | |
|---|---|---|
| Shortname / Alias: schedulechan | ge | |
| ID: 912 | | |
| Take PrEP when my schedule of[ | changes:*<br>] | _ 10 or N/A |
| PrEP Confidence 3 | | |
| ID: 913 | | |
| | u feel about the following stateme<br>bout each statement on a scale fr | |
| Validation: Min = 1 Max = 10 | | |
| Shortname / Alias: whiletraveling | | |
| ID: 914 | | |
| How confident are you that you | u will be able to | |
| Take PrEP while traveling:* 1[ | ] | _ 10 or N/A |
| Validation: Min = 1 Max = 10 | | |
| Shortname / Alias: takewsideeffe | cts | |
| Take PrEP when you are havin 1[ | g medication side effects:* | _ 10 or N/A |
| Validation: Min = 1 Max = 10 | | |
| Shortname / Alias: havingcrisis ID: 916 | | |
| Take PrEP when you are havin | g a crisis:* | _ 10 or N/A |

### **PrEP Delivery**

Shortname / Alias: prep prefmode

ID: 597

Right now there are no other approved options for taking PrEP. However, if there were more than one option and each method was equally good at protecting you from getting HIV, which method would you most prefer?\*

- () Taking one pill, every day
- () Taking two pills before you had sex and a pill a day for the next two days
- () Taking one pill a day just on Tuesday, Thursday, Saturday, and Sunday
- () Getting an injection about every 2 to 3 months
- ( ) Putting medicated lubrication (lube) in your anus (and/or your partner's anus) both before and after having anal sex
- ( ) Douching with a medicated solution (microbicide) before having anal sex

Action: JavaScript: Hide General Error Message

**PrEP Beliefs** 

Shortname / Alias: prepbeliefs

ID: 598

Please rate your agreement with the following statements:\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| Men are less likely to use condoms for anal sex if they are using PrEP | () | () | () | () |

| I feel as if<br>starting to<br>take PrEP<br>will allow<br>me to have<br>more sex<br>partners | () | () | () | () |
|---|---|---|---|---|
| I feel as if<br>starting to<br>take PrEP<br>will allow<br>me to have<br>more<br>condomless<br>anal sex | () | () | () | () |

### **PrEP and People**

Shortname / Alias: prepppl

ID: 193

We are interested in how you feel about the following statements. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I worry people will assume I sleep around if they know I take PrEP | () | () | () | () |
| I worry people will assume that I am HIV- positive if they know I take PrEP | () | () | () | () |
| I worry<br>people will<br>think my<br>partner(s) | () | () | () | () |

| are HIV-<br>positive if<br>they know I<br>take PrEP | | | | |
|---|---|---|---|---|
| I worry about listing PrEP as one of my current medications during appointments such as at a dentist's or specialist's office | () | () | () | () |
| I feel<br>ashamed to<br>tell other<br>people that I<br>am taking<br>PrEP | () | () | () | () |
| I worry people will think I am a bad person if they know I take PrEP | () | () | () | () |
| I worry<br>people will<br>think I am<br>gay if they<br>know I take<br>PrEP | () | () | () | () |
| I worry my<br>friends will<br>find out that I<br>take PrEP | () | () | () | () |
| I worry my<br>family will<br>find out that I<br>take PrEP | () | () | () | () |
| I worry my<br>sexual<br>partners will<br>find out that I<br>take PrEP | () | () | () | () |

| I think people<br>will give me a<br>hard time if I<br>tell them I<br>take PrEP | () | () | () | () |
|---|---|---|---|---|
| I think people<br>will judge me<br>if they know I<br>am taking<br>PrEP | () | () | () | () |

### **PrEP Concerns**

Shortname / Alias: prepconc

ID: 210

We are interested in how you feel about the following statements. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| My family<br>does not<br>support me<br>taking PrEP | () | () | () | () |
| My friends<br>do not<br>support me<br>taking PrEP | () | () | () | () |
| People<br>taking PrEP<br>are<br>portrayed<br>poorly in the<br>media and<br>online | () | () | () | () |
| People in my<br>community<br>talk poorly<br>about people<br>taking PrEP | () | () | () | () |

| I feel<br>embarrassed<br>about taking<br>PrEP | () | () | () | () |
|---|---|---|---|---|
| I think I am<br>not following<br>the 'rules' of<br>my<br>community if<br>I take PrEP | () | () | () | () |

### **PrEP Difficulties**

Shortname / Alias: prepdifficulties

ID: 602

In making your decision to continue taking PrEP after you start, please rate how much the following items concern you.\*

| | Not at all concerned | A little concerned | Concerned | Very<br>concerned |
|---|---|---|---|---|
| Getting the costs of PrEP covered (including office visits or office visit copays, lab costs, transportation costs) | () | () | () | () |
| Using insurance to get coverage for PrEP costs (including office visits, lab costs) | () | () | () | () |
| Getting<br>transportation | () | () | () | () |

| to PrEP<br>appointments<br>and labs | | | | |
|---|---|---|---|---|
| Returning for<br>PrEP follow-<br>up<br>appointments<br>and labs | () | () | () | () |
| Getting PrEP prescription refilled | () | () | () | () |

### **PrEP Difficulties Continued**

Shortname / Alias: prepdifficulties2

ID: 649

In making your decision to start taking PrEP, please rate how much the following items concern

| you." | | | | |
|---|---|---|---|---|
| | Not at all concerned | A little concerned | Concerned | Very<br>concerned |
| The possibility that if I were to become HIV+, certain medications might no longer work or I might be resistant to them | () | () | () | () |
| The possibility that PrEP might not provide complete | () | () | () | () |

| protection<br>against HIV | | | | |
|---|---|---|---|---|
| Having to talk to a health care provider about PrEP | () | () | () | () |
| Having to talk to a health care provider about my sex life | () | () | () | () |
| Experiencing side effects from PrEP | () | () | () | () |
| The long-<br>term effects<br>of PrEP on<br>my health | () | () | () | () |
| Having to<br>remember to<br>take PrEP<br>every day | () | () | () | () |
| Friends<br>finding out<br>that I am on<br>PrEP | () | () | () | () |
| Family<br>members<br>finding out<br>that I am on<br>PrEP | () | () | () | () |
| Sexual partners finding out that I am on PrEP | () | () | () | () |

Logic: Hidden unless: Question "The possibility that PrEP might not provide complete protection against HIV" is one of the following answers ("Concerned", "Very concerned")

Shortname / Alias: prepworry

| Т | D | ) - ( | 6 | 8 | $\overline{}$ |
|---|---|-------|---|----|---------------|
| | ப | - | U | U. | |

| Why do you worry about the <b> </b> | oossibility that PrEP | might not provide | complete protection | against |
|---|---|---|---|---|
| HIV? (Check all that apply)* | | | | |

- [] I worry that the drug is not effective at preventing HIV
- [] Because I worry that I won't take PrEP every day consistently
- [] Because I feel I am at very high risk for becoming infected with HIV
- [] Other, please specify::

\_\_\_\_\_

### **HIV** perceptions

Shortname / Alias: hivthoughts

ID: 667

Imagine how you would feel if you became infected with HIV. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I would<br>be afraid<br>people<br>would<br>judge me<br>when<br>they<br>learn I<br>have HIV | () | () | () | () |
| If I got infected, people would not want to have sex with me | () | () | () | () |
| I would<br>feel<br>guilty if I<br>got HIV | () | () | () | () |

| I would<br>feel<br>ashamed<br>if I got<br>HIV | () | () | () | () | |
|---|---|---|---|---|---|
| Insurance | | | | | |
| | len unless: #' | | | | e health insurance or health care |
| _ | Alias: ins_typ | _ | | , | |
| What kind o | of health insu | rance or hea | Ith care co | overage do y | ou have? Select all that apply.* |
| [] National H<br>[] Private co<br>[] Private pe<br>[] Civil servi | ersonal insural<br>ce health cove<br>ersonal insural | ge<br>nce<br>erage | | | |
| PEP | | | | | |
| Shortname / | Alias: pep | | | | |
| ID: 229 | | | | | |
| | | | | | medicines <u>AFTER</u> a sexual or drug ed post-exposure prophylaxis, or |

| Logic: Show/hide trigger exists. |
|---|
| Shortname / Alias: lifetimepep |
| ID: 230 |
| Have you ever taken post-exposure prophylaxis (PEP) <u>AFTER</u> a sexual or drug use exposure to reduce the risk of getting HIV?* ( ) Yes |
| ( ) No |
| Logic: Hidden unless: #113 Question "Have you ever taken post-exposure prophylaxis (PEP) <u>AFTER</u> a sexual or drug use exposure to reduce the risk of getting HIV?" is one of the following answers ("Yes") |
| Shortname / Alias: lastyearpep |
| ID: 231 |
| In the past 12 months, have you taken PEP (post-exposure prophylaxis) AFTER a sexual or drug use exposure, to reduce the risk of getting HIV?* ( ) Yes ( ) No |
| PrEP On-demand |
| Shortname / Alias: heardprepod |
| ID: 673 |
| Some people choose to not take PrEP daily, but only around the time when they are planning to have sex. This is known as on-demand or episodic PrEP, where you take two pills before having sex, and one pill a day or two days after. It is not an approved method and has not been shown to be an effective method for preventing HIV. Before today, have you ever heard of on-demand PrEP?* () Yes |

## **Substances**

( ) No

() Decline to answer

#### ID: 232

Now we'd like to ask you a little bit about your experiences using alcohol, tobacco products, and other drugs. Please be assured that this information will be treated as strictly confidential.

The questions will concern your experiences with using these substances across your lifetime and in the past three months. These substances can be smoked, swallowed, snorted, inhaled, injected, or taken in the form of pills. Some of the substances may be prescribed by a doctor (like amphetamines, sedatives, or pain medications). For this survey, do not report on medications that are used as prescribed by your doctor. However, if you have taken such medications for reasons other than prescription, or taken them more frequently or at higher doses than prescribed, please report on this use. Once again, please remember that all information provided will be treated as *strictly confidential*.

Shortname / Alias: lifetimesubstanceuse

ID: 233

# Which of the following drugs have you used in your life? Please check all that apply.\*

- [] Tobacco (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)
- [] Alcohol (beer, wine, spirits, etc.)
- [] Cannabis (marijuana, pot, weed, grass, hash, synthetic cannabis, etc.)
- [] Cocaine (coke, crack, etc.)
- [] Amphetamines (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)
- [] Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)
- [] Sedatives, tranquilizers, or sleeping pills (valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)
- [] Hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)
- [ ] Opioids (heroin, morphine, methadone, codeine, Oxycotin, Percocet, Vicodin, etc.)
- [] None of these

**Page entry logic:** This page will show when: #118 Question "Which of the following drugs have you used in your life?

*Please check all that apply.*" is one of the following answers ("Tobacco (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)")

#### Tobacco

| Shortname / Alias: tobacco3months |
|---|
| ID: 234 |
| In the past 3 months, how often have you used tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccodesire |
| ID: 235 |
| During the past 3 months, how often have you had a desire to use tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccoproblems |
| ID: 236 |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccofailed |
| ID: 237 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, |

**etc.)?\*** ( ) Never

() Once or twice

() Monthly

| ( ) Daily or almost daily |
|---|
| Shortname / Alias: tobaccofriend |
| ID: 238 |
| Has a friend or relative or anyone else ever expressed concern about your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| Shortname / Alias: tobaccostop |
| ID: 239 |
| Have you ever tried and failed to control, cut down or stop using tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| <b>Page entry logic:</b> This page will show when: #118 Question "Which of the following drugs have you used in your life? Please check all that apply." is one of the following answers ("Alcohol (beer, wine, spirits, etc.)") |
| Alcohol |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: alcohol3months |
| ID: 240 |
| In the past 3 months, how often have you used alcoholic beverages (beer, wine, spirits, etc.)?* |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

Logic: Hidden unless: #125 Question "In the past 3 months, how often have you used alcoholic

beverages (beer, wine, spirits, etc.)?" is one of the following answers ("Once or

twice","Monthly","Weekly","Daily or almost daily","Decline to answer")

() Weekly

52

| Shortname / Alias: alcoholdaily |
|---|
| ID: 241 |
| How many drinks containing alcohol do you have on a typical day?* |
| ( ) 1 or 2 |
| () 3 or 4 |
| () 5 or 6 |
| () 7 to 9 |
| ( ) 10 or more |
| Shortname / Alias: alcoholbinge |
| ID: 242 |
| How often do you have 5 or more drinks on one occasion?* ( ) Never |
| ( ) Less than monthly |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholdesire |
| ID: 243 |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| ( ) Daily or almost daily |
| ( ) Daily or almost daily Shortname / Alias: alcoholproblems |
| Shortname / Alias: alcoholproblems |
| Shortname / Alias: alcoholproblems ID: 244 During the past 3 months, how often has your use of alcoholic beverages (beer, wine, spirits, etc.) led to health, social, legal or financial problems?* |
| Shortname / Alias: alcoholproblems ID: 244 During the past 3 months, how often has your use of alcoholic beverages (beer, wine, spirits, etc.) led to health, social, legal or financial problems?* ( ) Never |

| Shortname / Alias: alcoholfailed |
|---|
| ID: 245 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholfriend |
| ID: 246 |
| Has a friend or relative or anyone else ever expressed concern about your use of alcoholic beverages (beer, wine, spirits, etc.)?* ( ) No, never |
| beverages (beer, wine, spirits, etc.)?* |
| beverages (beer, wine, spirits, etc.)?* ( ) No, never |
| beverages (beer, wine, spirits, etc.)?* ( ) No, never ( ) Yes, in the past 3 months |
| beverages (beer, wine, spirits, etc.)?* ( ) No, never ( ) Yes, in the past 3 months |
| beverages (beer, wine, spirits, etc.)?* ( ) No, never ( ) Yes, in the past 3 months ( ) Yes, but not in the past 3 months |
| beverages (beer, wine, spirits, etc.)?* ( ) No, never ( ) Yes, in the past 3 months ( ) Yes, but not in the past 3 months Shortname / Alias: alcoholstop |
| beverages (beer, wine, spirits, etc.)?* () No, never () Yes, in the past 3 months () Yes, but not in the past 3 months Shortname / Alias: alcoholstop ID: 247 Have you ever tried and failed to control, cut down or stop using alcoholic beverages (beer, wine, spirits, etc.)?* |

**Page entry logic:** This page will show when: #118 Question "Which of the following drugs have you used in your life?

*Please check all that apply.*" is one of the following answers ("Cannabis (marijuana, pot, weed, grass, hash, synthetic cannabis, etc.)")

#### **Cannabis**

() Daily or almost daily

Shortname / Alias: cannabis3months

ID: 251

| In the past 3 months, how often have you used cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| <b>Page entry logic:</b> This page will show when: #135 Question "In the past 3 months, how often have you used cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?" is one of the following answers ("Once or twice", "Monthly", "Weekly", "Daily or almost daily") |
| Cannabis (cont.) |
| Shortname / Alias: cannabisdesire |
| ID: 252 |
| During the past 3 months, how often have you had a desire to use cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) One contains |
| ( ) Once or twice |
| ( ) Monthly |
| ( ) Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisproblems |
| ID: 253 |
| During the past 3 months, how often has your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisfailed |
| ID: 254 |

| because of your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
|---|
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisfriend |
| ID: 255 |
| Has a friend or relative or anyone else ever expressed concern about your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| Shortname / Alias: cannabisstop |
| ID: 256 |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) No, never |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) No, never |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) No, never ( ) Yes, in the past 3 months |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) No, never ( ) Yes, in the past 3 months |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) No, never ( ) Yes, in the past 3 months |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* () No, never () Yes, in the past 3 months () Yes, but not in the past 3 months Page entry logic: This page will show when: #118 Question "Which of the following drugs have you used in your life? Please check all that apply." is one of the following answers ("Cocaine (coke, crack, etc.)") |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) No, never ( ) Yes, in the past 3 months ( ) Yes, but not in the past 3 months Page entry logic: This page will show when: #118 Question "Which of the following drugs have you used in your life? |
| Have you ever tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* () No, never () Yes, in the past 3 months () Yes, but not in the past 3 months Page entry logic: This page will show when: #118 Question "Which of the following drugs have you used in your life? Please check all that apply." is one of the following answers ("Cocaine (coke, crack, etc.)") |

In the past 3 months, how often have you used cocaine (coke, crack, etc.)?\*

() Never

() Monthly () Weekly

() Once or twice

During the past 3 months, how often have you failed to do what was normally expected of you

| ( ) Daily or almost daily |
|---|
| <b>Page entry logic:</b> This page will show when: #141 Question "In the past 3 months, how often have you used cocaine (coke, crack, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Cocaine (cont.) |
| Shortname / Alias: cocainedesire ID: 258 |
| During the past 3 months, how often have you had a desire to use cocaine (coke, crack, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cocaineproblems |
| Shortname / Alias: cocaineproblems ID: 259 |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily Shortname / Alias: cocainefailed |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: cocainefailed ID: 260 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of cocaine (coke, crack, etc.)?* |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: cocainefailed ID: 260 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of cocaine (coke, crack, etc.)?* ( ) Never |

| ( ) Daily or almost daily |
|---|
| Shortname / Alias: cocainefriend |
| ID: 261 |
| Has a friend or relative or anyone else ever expressed concern about your use of cocaine (coke, crack, etc.)?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| Shortname / Alias: cocainestop |
| ID: 262 |
| Have you ever tried and failed to control, cut down or stop using cocaine (coke, crack, etc.)?* |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| Page entry logic: This page will show when: #118 Question "Which of the following drugs have you |
| used in your life? Please check all that apply." is one of the following answers ("Amphetamines (speed, meth, diet pills, |
| ecstasy, Ritalin, Adderall, etc.)") |
| Amphatamina |
| Amphetamine |
| Shortname / Alias: amphetamine3months |
| ID: 263 |
| In the past 3 months, how often have you used amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |

() Daily or almost daily

**Page entry logic:** This page will show when: #147 Question "In the past 3 months, how often have you used amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?" is one of the following answers ("Once or twice", "Monthly", "Weekly", "Daily or almost daily")

### **Amphetamine (cont.)**

| Shortname / Alias: amphetaminedesire |
|---|
| ID: 265 |
| During the past 3 months, how often have you had a desire to use amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetamineproblems |
| ID: 266 |
| During the past 3 months, how often has your use of amphetamine type stimulants (speed, methodiet pills, ecstasy, Ritalin, Adderall, etc.) led to health, social, legal or financial problems?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetaminefailed |
| ID: 267 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

| ID: 268 |
|---|
| Has a friend or relative or anyone else ever expressed concern about your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| Shortname / Alias: amphetaminestop |
| ID: 269 |
| Have you ever tried and failed to control, cut down or stop using amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| Page entry logic: This page will show when: #118 Question "Which of the following drugs have you used in your life? |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") Inhalants |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") Inhalants Shortname / Alias: inhalants3months |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") Inhalants |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") Inhalants Shortname / Alias: inhalants3months |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") Inhalants Shortname / Alias: inhalants3months ID: 271 In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") Inhalants Shortname / Alias: inhalants3months ID: 271 In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) Never |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") Inhalants Shortname / Alias: inhalants3months ID: 271 In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) Never ( ) Once or twice |
| used in your life? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") Inhalants Shortname / Alias: inhalants3months ID: 271 In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* () Never () Once or twice () Monthly |

Shortname / Alias: amphetaminefriend

**Page entry logic:** This page will show when: #153 Question "In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily")

# Inhalants (cont.)

| Shortname / Alias: inhalantsdesire |
|---|
| ID: 272 |
| During the past 3 months, how often have you had a desire to use inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsproblems |
| ID: 273 |
| During the past 3 months, how often has your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.) led to health, social, legal or financial problems?* |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsfailed |
| ID: 274 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsfriend |
| ID: 275 |
| Has a friend or relative or anyone else ever expressed concern about your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* () No, never |

| ( ) Yes, in the past 3 months |
|---|
| ( ) Yes, but not in the past 3 months |
| Shortname / Alias: inhalantsstop |
| ID: 276 |
| Have you ever tried and failed to control, cut down or stop using inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| <b>Page entry logic:</b> This page will show when: #118 Question "Which of the following drugs have you used in your life? |
| Please check all that apply." is one of the following answers ("Sedatives, tranquilizers, or sleeping pills (valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)") |
| Sedatives |
| Chartenana / Alian, and tive a 2 mountly a |
| Shortname / Alias: sedatives3months |
| ID: 277 |
| In the past 3 months, how often have you used sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| <b>Page entry logic:</b> This page will show when: #159 Question "In the past 3 months, how often have you used sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Sedatives (cont.) |

Shortname / Alias: sedativesdesire

ID: 279

62

| sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never |
|---|
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: sedativesproblems |
| ID: 280 |
| During the past 3 months, how often has your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.) led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: sedativesfailed |
| Shortname / Alias: sedativesfailed ID: 281 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never ( ) Once or twice |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily Shortname / Alias: sedativesfriend ID: 282 Has a friend or relative or anyone else ever expressed concern about your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* |

During the past 3 months, how often have you had a desire to use sedatives, tranquilizers, or

| ID: 283 |
|---|
| Have you ever tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| <b>Page entry logic:</b> This page will show when: #118 Question "Which of the following drugs have you used in your life? Please check all that apply." is one of the following answers ("Hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)") |
| Hallucinogens |
| Shortname / Alias: hallucinogens3months |
| ID: 285 |
| In the past 3 months, how often have you used hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

**Page entry logic:** This page will show when: #165 Question "In the past 3 months, how often have you used hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily")

### Hallucinogens (cont.)

Shortname / Alias: sedativesstop

Shortname / Alias: hallucinogensdesire

ID: 286

During the past 3 months, how often have you had a desire to use hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?\*

- () Never
- () Once or twice

| ( ) Monthly |
|---|
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensproblems |
| ID: 287 |
| During the past 3 months, how often has your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.) led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensfailed |
| ID: 288 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensfriend |
| ID: 289 |
| Has a friend or relative or anyone else ever expressed concern about your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) No, never |
| ( ) Yes, in the past 3 months |
| ( ) Yes, but not in the past 3 months |
| Shortname / Alias: hallucinogensstop |
| ID: 290 |
| Have you ever tried and failed to control, cut down or stop using hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) No, never |

| () Yes, in the past 3 months |
|--------------------------------------|
| () Yes, but not in the past 3 months |

**Page entry logic:** This page will show when: #118 Question "Which of the following drugs have you used in your life?

*Please check all that apply.*" is one of the following answers ("Opioids (heroin, morphine, methadone, codeine, Oxycotin, Percocet, Vicodin, etc.)")

### **Opioids**

Shortname / Alias: opioids3months

ID: 291

In the past 3 months, how often have you used opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?\*

- () Never
- () Once or twice
- () Monthly
- () Weekly
- () Daily or almost daily

**Page entry logic:** This page will show when: #171 Question "In the past 3 months, how often have you used opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?" is one of the following answers ("Once or twice", "Monthly", "Weekly", "Daily or almost daily")

### **Opioids (cont.)**

Logic: Show/hide trigger exists.

Shortname / Alias: opioidsheroin

ID: 299

In the past 3 months, has your opioid use included heroin?\*

- () Yes
- () No

Logic: Hidden unless: #172 Question "In the past 3 months, has your opioid use included heroin?" is one of the following answers ("Yes")

Shortname / Alias: heroinprimary

| ID: 300 |
|---|
| In the past 3 months, was heroin the most common opioid that you used?* ( ) Yes ( ) No |
| Shortname / Alias: opioidssdesire |
| ID: 293 |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: opioidsproblems |
| ID: 294 |
| During the past 3 months, how often has your use of opioids (heroin, morphine, methadone, |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily Shortname / Alias: opioidsfailed |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily Shortname / Alias: opioidsfailed ID: 295 |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: opioidsfailed ID: 295 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: opioidsfailed ID: 295 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: opioidsfailed ID: 295 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly |
| codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: opioidsfailed ID: 295 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice |

Shortname / Alias: opioidsfriend

#### ID: 296

Has a friend or relative or anyone else ever expressed concern about your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?\*

- () No, never
- () Yes, in the past 3 months
- () Yes, but not in the past 3 months

Shortname / Alias: opioidsstop

ID: 297

Have you ever tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?\*

- () No, never
- () Yes, in the past 3 months
- () Yes, but not in the past 3 months

#### **Sexual Behaviors**

**Page exit logic:** Skip / Disqualify Logic**IF:** #179 Question "In the past 3 months, how many people have you had anal sex with?" is exactly equal to "0" **THEN:** Jump to page 123 - Perceived HIV Risk

ID: 368

The next section of questions will ask about your sexual behaviors. We know that this can be a sensitive topic, so we would like to remind you that your answers will be kept completely confidential. Please be as honest as possible in order to ensure the success of the current study.

The following questions refer to your sexual behavior during the past 3 months. Our focus will be only on anal sex. Therefore, do not include references to people with whom you did not engage in anal sex.

For these questions, anal sex refers to sex where the other person's penis was in your rectum (you were the bottom) and to sex where your penis was in the other person's rectum (you were the top).

These questions only ask about people assigned male at birth, which includes cisgender men (men assigned male at birth) and transgender women (women assigned male at

birth). Therefore, do not include references to cisgender women (women assigned female at birth) or transgender men (men assigned female at birth).

| Validation: Min = 0 Max = 999 Must be numeric Whole numbers only Positive numbers only |
|---|
| Shortname / Alias: numsexpartner |
| ID: 302 |
| In the past 3 months, how many people have you had anal sex with?* |
| Page entry logic: This page will show when: #179 Question "In the past 3 months, how many people have you had anal sex with?" is greater than "0" |
| HIV Status of Sexual Partners |
| Logic: Hidden by default |
| ID: 677 |
| The total number must equal the number of people you had anal sex with in the last 3 months ([question('value'), id='302']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: partnerhivstatus |
| ID: 676 |
| Before you had sex, what did you know of the HIV status of your sexual partner(s)? |
| Enter numerical values. Numbers must add up to [question('value'), id='302'], the number of people you reported having anal sex within the last three months.* This person/these people told you they were HIV negative and you had no reason to doubt it |
| You knew this person/these people were HIV positive |
| You were not completely sure of this person/these people's HIV status |
| Action: Custom Script: Script to check the continuous sum totals |

Page entry logic: This page will show when: Num HIV Neg partners is greater than "0"

### **HIV Negative Partners**

ID: 690

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Shortname / Alias: hivneg\_timesbot

ID: 701

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom?\*

\_\_\_\_\_

Shortname / Alias: hivneg\_timestop

ID: 702

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the top?\*

**Page entry logic:** This page will show when: #181 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative <a href="where you were the bottom">where you were the bottom</a>?" is greater than "0"

**HIV Negative Partners - Condomless Receptive Al** 

Logic: Hidden by default

ID: 714

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='701']). Please correct this.

Shortname / Alias: hivneg timesbotunp

| In the past 3 months, how many of the [question('value'), id='701'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom were without a condom? * |
|---|
| Action: Custom Script: Check number condomless is not greater than total times |
| <b>Page entry logic:</b> This page will show when: #183 Question "In the past 3 months, how many of the [question('value'), id='701'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom were without a condom?" is greater than "0" |
| HIV Negative Partners - Condomless Receptive Al |
| ID: 721 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative |
| Logic: Hidden by default |
| ID: 999 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivneg_botunp_typ |
| ID: 711 |
| Regarding the partners who told you they were HIV negative who you had <u>condomless receptive</u> <u>anal sex with (where you were the bottom)</u> , how many were |
| Enter numerical values.* |

\_Casual hook-up(s) or one-night stand(s)

ID: 710

| etc. |
|---|
| Logic: Hidden by default |
| ID: 1002 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivneg_botunp_gender |
| ID: 964 |
| How many were |
| Enter numerical values.*MenTranswomenNon-binary, genderqueer, or gender non-conforming |
| Hidden Page of Script Action: Custom Script: Script to check continuous sum totals |
| Hidden Page of Script Action: Custom Script: Script to check continuous sum totals |

**Page entry logic:** This page will show when: #182 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the top?" is greater than "0"
The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 719

This number cannot be greater than the number of times you had anal sex where you were the top ([question('value'), id='702']). Please correct this.

Shortname / Alias: hivneg timestopunp

ID: 718

In the past 3 months, how many of the [question('value'), id='702'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the top were without a condom? \*

## **Hidden Page of Script**

Action: Custom Script: Script to check number condomless is not greater than the totals

**Page entry logic:** This page will show when: #186 Question "In the past 3 months, how many of the [question('value'), id='702'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the top were without a condom?" is greater than "0"

# **HIV Negative Partners - Condomless Insertive AI**

ID: 723

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this. |
|---|
| Validation: Must be numeric |
| Shortname / Alias: hivneg_topunp_typ |
| ID: 725 |
| Regarding the partners who told you they were HIV negative who you had <u>condomless insertive</u> anal sex with (where you were the top), how many were |
| Enter numerical values.* |
| Romantic partner(s), someone you are in a relationship with |
| Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, |
| etc. |
| Logic: Hidden by default |
| ID: 1005 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivneg_topunp_gender |
| ID: 965 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |

Action: Custom Script: Script to check continuous sum totals

Logic: Hidden by default

ID: 1004

74

Action: Custom Script: Script to check continuous sum totals

Page entry logic: This page will show when: Num HIV Neg partners is greater than "0"

### **HIV Negative Partners - PrEP and Alcohol and Drug Use**

ID: 992

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 732

This number cannot be greater than the number of partners who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Shortname / Alias: hivneg toldyouprep

ID: 729

How many of your sexual partners who told you they were HIV negative told you they were taking PrEP?

Number must be less than or equal to [question('option value'), id='676', option='12278'].\*

Logic: Hidden by default

ID: 733

This number cannot be greater than the number of partners who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Logic: Hidden unless: #190 Question "Regarding your sexual partners who told you they were HIV negative, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivneg youtoldprepnum

How many of your sexual partner(s) who told you they were HIV negative did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12278'].\*

\_\_\_\_\_

Shortname / Alias: hivneg\_timesdrunk

ID: 740

In the past 3 months, how many of the times you had anal sex with partners who told you they were HIV negative were you or this person under the influence of alcohol or drugs?\*

\_\_\_\_\_

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Page entry logic: This page will show when: Num HIV Pos partners is greater than "0"

#### **HIV Positive Partners**

ID: 770

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Shortname / Alias: hivpos\_timesbot

ID: 775

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom?\*

Shortname / Alias: hivpos\_timestop

| | | 7 | 7 | a |
|---|----|-----|---|---|
| - | ٠. | - 1 | • | u |

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the top?\*

\_\_\_\_\_

**Page entry logic:** This page will show when: #193 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom?" is greater than "0"

## **HIV Positive Partners - Condomless Receptive AI**

ID: 782

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 783

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='775']). Please correct this.

Shortname / Alias: hivpos timesbotunp

ID: 784

In the past 3 months, how many of the [question('value'), id='775'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom were without a condom? \*

Action: Custom Script: Check number condomless is not greater than total times

**Page entry logic:** This page will show when: #195 Question "In the past 3 months, how many of the [question('value'), id='775'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom were without a condom? " is greater than "0"

### **HIV Positive Partners - Condomless Receptive AI**

ID: 786

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 1008

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivpos botunp typ

ID: 788

Regarding the partners who told you they were HIV positive who you had <u>condomless receptive</u> <u>anal sex with (where you were the bottom)</u>, how many were...

Enter numerical values.\*

| F | _Romantic partner(s), someone you are in a relationship with |
|---|--------------------------------------------------------------|
| | _Casual hook-up(s) or one-night stand(s) |

\_\_\_\_\_A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc.

Logic: Hidden by default

ID: 1009

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivpos\_botunp\_gender

ID: 994

| How many were |
|---|
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, and gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| <b>Page entry logic:</b> This page will show when: #194 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the top?" is greater than "0" |
| HIV Pos Partners - Condomless Insertive Al |
| ID: 792 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive. |
| Logic: Hidden by default |
| ID: 793 |
| This number cannot be greater than the number of times you had anal sex where you were the top ([question('value'), id='776']). Please correct this. |
| Shortname / Alias: hivpos_timestopunp ID: 794 |

| In the past 3 months, how many of the [question('value'), id='776'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the top were without a condom? * |
|---|
| Action: Custom Script: Script to check number condomless is not greater than the totals |
| <b>Page entry logic:</b> This page will show when: #198 Question "In the past 3 months, how many of the [question('value'), id='776'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the top were without a condom? " is greater than "0" |
| HIV Positive Partners - Condomless Insertive Al |
| ID: 796 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive. |
| Logic: Hidden by default |
| ID: 1012 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivpos_topunp_typ ID: 798 |
| Regarding the partners who told you they were HIV positive who you had <u>condomless insertive</u> <u>anal sex with (where you were the top)</u> , how many were |
| Enter numerical values.*Romantic partner(s), someone you are in a relationship with |
| Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |

ID: 800

taking medication to treat HIV?

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivpos_topunp_gender |
| ID: 995 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: Num HIV Pos partners is greater than "0" |
| HIV Positive Partners - HIV Trt |
| Logic: Hidden by default |
| ID: 799 |
| This number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this. |
| Shortname / Alias: hivpos_toldyouhivmeds |

How many of your sexual partners who told you they were HIV positive told you they were

Number must be less than or equal to [question('option value'), id='676', option='12279'].

81

Logic: Hidden by default

ID: 920

The number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Shortname / Alias: hivpos\_toldyouundetect

ID: 918

How many of your sexual partners who told you they were HIV positive told you they were undetectable?

**Number must be less than or equal to** [question('option value'), id='676', option='12279'].

\_\_\_\_\_

Logic: Hidden by default

ID: 802

This number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Shortname / Alias: hivpos timesdrunk

ID: 807

In the past 3 months, how many of the times you had anal sex with partners who told you they were HIV positive were you or this person under the influence of alcohol or drugs?\*

Action: Custom Script: Script to check med number not greater than the total number of partners

Action: Custom Script: Script to check undetectable number not greater than the total number of partners

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Page entry logic: This page will show when: Num HIV Unk partners is greater than "0"

**HIV Status Unknown Partners** 

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Shortname / Alias: hivunk timesbot

ID: 815

In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom?\*

\_\_\_\_\_\_

Shortname / Alias: hivunk\_timestop

ID: 816

In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?\*

\_\_\_\_\_

**Page entry logic:** This page will show when: #206 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of <a href="where you were the bottom?">where you were the bottom?</a>" is greater than "0"

**HIV Status Unknown Partners - Condomless Receptive AI** 

ID: 822

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 823

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='815']). Please correct this.

Shortname / Alias: hivunk\_timesbotunp

ID: 824

In the past 3 months, how many of the [question('value'), id='815'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom were without a condom? \*

Action: Custom Script: Check number condomless is not greater than total times

**Page entry logic:** This page will show when: #208 Question "In the past 3 months, how many of the [question('value'), id='815'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom were without a condom? " is greater than "0"

### **HIV Status Unknown Partners - Condomless Receptive Al**

ID: 826

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 1016

The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivunk\_botunp\_typ

ID: 828

Regarding the partners whose HIV status you were not sure of who you had <u>condomless</u> <u>receptive anal sex with (where you were the bottom)</u>, how many were...

| Enter numerical values.* |
|---|
| Romantic partner(s), someone you are in a relationship with Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, |
| etc. |
| Logic: Hidden by default |
| ID: 1017 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivunk_botunp_gender |
| ID: 996 |
| How many were |
| Enter numerical values.* Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: #207 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" |
| you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the |

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 833

This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this.

Shortname / Alias: hivunk timestopunp

ID: 834

In the past 3 months, how many of the [question('value'), id='816'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top were without a condom?\*

Action: Custom Script: Script to check number condomless is not greater than the totals

**Page entry logic:** This page will show when: #211 Question "In the past 3 months, how many of the [question('value'), id='816'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top were without a condom?" is greater than "0"

**HIV Status Unknown Partners - Condomless Insertive AI** 

ID: 836

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 1020

The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivunk_topunp_typ |
| ID: 838 |
| Regarding the partners whose HIV status you were not sure of who you had <u>condomless</u> <u>insertive anal sex with (where you were the top)</u> , how many were |
| Enter numerical values.*Romantic partner(s), someone you are in a relationship with |
| Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |
| Logic: Hidden by default ID: 1021 |
| ID. 1021 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivunk_topunp_gender |
| ID: 997 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |

Page entry logic: This page will show when: Num HIV Unk partners is greater than "0"

#### **HIV Status Unknown Partners - PrEP**

Logic: Hidden by default

ID: 839

This number cannot be greater than the number of partners whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Shortname / Alias: hivunk\_toldyouprep

ID: 840

How many of your sexual partners whose HIV status you were not sure of told you they were taking PrEP?

Number must be less than or equal to [question('option value'), id='676', option='12280'].\*

\_\_\_\_\_

Logic: Hidden by default

ID: 842

This number cannot be greater than the number of partners whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Shortname / Alias: hivunk timesdrunk

ID: 847

In the past 3 months, how many of the times you had anal sex with partners whose HIV status you were not sure of were you or this person under the influence of alcohol or drugs?\*

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

### **Perceived HIV Risk**

| Shortname / Alias: perceivedrisk1 |
|---|
| ID: 762 |
| Based on your reported sexual activities over the last 3 months, how at risk do you think you were for contracting HIV in the last 3 months?* ( ) Not at all at risk for contracting HIV |
| ( ) Somewhat at risk for contracting HIV |
| ( ) High risk for contracting HIV |
| Shortname / Alias: perceivedrisk2 |
| ID: 763 |
| What is your gut feeling about how likely you are to get infected with HIV?* ( ) Extremely unlikely |
| () Very unlikely |
| ( ) Somewhat likely |
| ( ) Very likely |
| ( ) Extremely likely |
| Shortname / Alias: perceivedrisk3 |
| ID: 764 |
| I worry about getting infected with HIV:* ( ) None of the time |
| () Rarely |
| () Some of the time |
| ( ) A moderate amount of time |
| ( ) A lot of the time |
| ( ) All of the time |
| Perceived HIV Risk |
| Shortname / Alias: perceivedrisk4 |

Getting HIV is something I am...\*
( ) Not concerned about

() A little concerned about

| ( ) Moderately concerned about |
|---|
| ( ) Concerned about a lot |
| ( ) Extremely concerned about |
| Shortname / Alias: perceivedrisk5 |
| ID: 766 |
| There is a chance, no matter how small, I could get HIV:* ( ) Strongly Disagree |
| ( ) Disagree |
| ( ) Neither agree nor disagree |
| () Agree |
| ( ) Strongly Agree |
| Shortname / Alias: perceivedrisk6 |
| ID: 767 |
| I think my chances of getting infected with HIV are:* ( ) Zero |
| ( ) Almost zero |
| () Small |
| () Moderate |
| () Large |
| () Very large |
| PHQ-2/GAD-2 |
| ID: 760 |
| ID: 768 |
| Now we are going to ask you about your mental health and how you have been feeling recently. |
| recently. |

Shortname / Alias: mentalhealthscreener

ID: 388

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Little interest or pleasure in doing things | () | () | () | () |
| Feeling<br>down,<br>depressed,<br>or<br>hopeless | () | () | () | () |
| Feeling<br>nervous,<br>anxious or<br>on edge | () | () | () | () |
| Not being<br>able to<br>stop or<br>control<br>worrying | () | () | () | () |

# **Hidden Mental Health Screener Script**

Hidden Value: psychdistress1

Value:

Hidden Value: psychdistress2

Value:

**Action: Custom Script: Mental Health Script** 

Page entry logic: This page will show when: psychdistress1 is greater than or equal to "3"

# PHQ-8

Shortname / Alias: phq8

ID: 397

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| Over the past 2 | wooko, | | | |
|---|---|---|---|---|
| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
| Trouble falling or staying asleep, or sleeping too much | () | () | () | () |
| Feeling tired<br>or having<br>little energy | () | () | () | () |
| Poor appetite or overeating | () | () | () | () |
| Feeling bad<br>about<br>yourself - or<br>that you are<br>a failure or<br>have let<br>yourself or<br>your family<br>down | () | () | () | () |
| Trouble concentrating on things, such as reading the newspaper or watching television | () | () | () | () |
| Moving or<br>speaking so<br>slowly that<br>other people<br>could have<br>noticed, or | () | () | () | () |

| fidgety or restless that you have been moving around a lot more than usual |
|----------------------------------------------------------------------------|
|----------------------------------------------------------------------------|

Page entry logic: This page will show when: psychdistress2 is greater than or equal to "3"

### GAD-7

Shortname / Alias: gad7

ID: 404

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Worrying<br>too much<br>about<br>different<br>things | () | () | () | () |
| Trouble relaxing | () | () | () | () |
| Being so<br>restless<br>that it is<br>hard to sit<br>still | () | () | () | () |
| Becoming<br>easily<br>annoyed<br>or irritable | () | () | () | () |

| Feeling ( afraid as if something awful might happen | ) () | () | () |
|-----------------------------------------------------|------|----|----|
|-----------------------------------------------------|------|----|----|

## **Social Isolation**

Shortname / Alias: socialisolation

ID: 432

The following questions ask about your relationships with other people.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| I feel<br>left out. | () | () | () | () | () |
| I feel<br>that<br>people<br>barely<br>know<br>me. | () | () | () | () | () |
| I feel isolated from others. | () | () | () | () | () |
| I feel that people are around me but not with me. | () | () | () | () | () |

# **Emotional Support**

Shortname / Alias: emotionalsupport

ID: 411

The following questions ask about your relationships with other people.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| I have someone who will listen to me when I need to talk. | () | () | () | () | () |
| I have<br>someone to<br>confide in or<br>talk to about<br>myself or<br>my<br>problems. | () | () | () | () | () |
| I have<br>someone<br>who makes<br>me feel<br>appreciated. | () | () | () | () | () |
| I have<br>someone to<br>talk with<br>when I have<br>a bad day. | () | () | () | () | () |

# **Informational Support**

Shortname / Alias: informational support

ID: 417

The following questions ask about your relationships with other people.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| I have<br>someone to<br>give me<br>good | () | () | () | () | () |

| advice<br>about a<br>crisis if I<br>need it. | | | | | |
|---|---|---|---|---|---|
| I have someone to turn to for suggestions about how to deal with a problem. | () | () | () | () | () |
| I have someone to give me information if I need it. | () | () | () | () | () |
| I get useful<br>advice<br>about<br>important<br>things in<br>life. | () | () | () | () | () |

# **Instrumental Support**

Shortname / Alias: instrumentalsupport

ID: 422

The following questions ask about your relationships with other people.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| Do you have someone to help you if you are confined to bed? | () | () | () | () | () |

| Do you have someone to take you to the doctor if you need it? | () | () | () | () | () |
|---|---|---|---|---|---|
| Do you have someone to help with your daily chores if you are sick? | () | () | () | () | () |
| Do you have someone to run errands if you need it? | () | () | () | () | () |

# Companionship

Shortname / Alias: companionship

ID: 427

The following questions ask about your relationships with other people.

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| Do you have someone with whom to have fun? | () | () | () | () | () |
| Do you have someone with whom to relax? | () | () | () | () | () |

| Do you have someone with whom you can do something enjoyable? | () | () | () | () | () |
|---|---|---|---|---|---|
| Do you find companionship when you want it? | () | () | () | () | () |

# Thank You!

ID: 1

Thank you for taking this survey!

### P3-T RCT Month-3 Follow-up (P3-T Arm)

Shortname / Alias: studyarm

ID: 1071

Enter Study Arm for testing survey (will switch to staff login before launch):

- () P3-T Arm
- () Standard of Care Arm

ID: 93

Thank you for participating in the P3-T study! The purpose of the study is to test a PrEP adherence intervention for young men who have sex with men who are starting PrEP. As part of the P3-T study, there are three surveys: one when you enrolled, one at your follow up appointment today, and one at your follow up appointment in 3 months.

Try to answer every question as best you can. If you need help, please ask the study staff. Your answers will be used only for research purposes. Let's get started!

#### **Cell Phone**

ID: 120

Now, we'd like to ask you about your cell phone and internet use.

Logic: Show/hide trigger exists.

Shortname / Alias: paychange

ID: 1068

In the last 3 months, has who pays for your cellphone or smart phone changed?\*

- () Yes
- () No

Logic: Hidden unless: #2 Question "In the last 3 months, has who pays for your cellphone or smart phone changed?" is one of the following answers ("Yes")

Shortname / Alias: phonepay

| ID: 127 |
|---|
| Who usually pays for your cell phone or smartphone plan?* |
| ( ) Someone else does |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: disconnect |
| ID: 128 |
| In the last 3 months, did you ever not have access to your phone or phone service?* ( ) Yes |
| ( ) No |
| Logic: Hidden unless: #4 Question "In the last 3 months, did you ever not have access to your |
| phone or phone service?" is one of the following answers ("Yes") |
| Shortname / Alias: disconnecttimes |
| ID: 129 |
| How many times in the last 3 months did you not have access to your phone or phone service?* ( ) Once |
| () Twice |
| ( ) 3 to 5 times |
| ( ) More than 5 times |
| Logic: Hidden unless: #4 Question "In the last 3 months, did you ever not have access to your phone or phone service?" is one of the following answers ("Yes") |
| Shortname / Alias: disconnectlength |
| ID: 130 |
| The <i>last</i> time you did not have access to your phone or phone service, for how long did you not have access?* ( ) 1 day or less |
| ( ) 2 to 6 days |

( ) 1 to 4 weeks

() More than 4 weeks

| Logic: Show/hide trigger exists. |
|---|
| Shortname / Alias: employed |
| ID: 109 |
| Are you currently employed?* ( ) Yes |
| ( ) No |
| Logic: Hidden unless: #7 Question "Are you currently employed?" is one of the following answers ("Yes") |
| Shortname / Alias: employedhours |
| ID: 110 |
| Are you employed full-time or part-time? Part-time means that you work less than 35 hours per week during most weeks.* ( ) Full time |
| ( ) Part time |
| Shortname / Alias: income_30d |
| ID: 564 |
| How much money did you make altogether during the past 30 days?* |
| ( ) Don't know |
| Shortname / Alias: incomelevel |
| ID: 111 |
| How would you describe your income level?* ( ) Low income |
| ( ) Middle income |
| ( ) High income |
| ( ) Decline to answer |
| Food. Shelter |

Shortname / Alias: cutmeal

ID: 565

| In the past 3 months, how often did you or your family have to cut meal size or skip a meal because there was not enough money for food?* ( ) Almost every week |
|---|
| ( ) Several weeks but not every week |
| ( ) Only a few weeks |
| ( ) Did not have to skip or cut the size of meals |
| Shortname / Alias: shelter |
| ID: 113 |
| In the past 3 months, have you spent at least one night (check all that apply):* [] In a shelter? |
| [] In a public place not intended for sleeping (e.g., bus station, car, abandoned building)? |
| [] On the street or anywhere outside (e.g., park, sidewalk)? |
| [] Temporarily doubled up with a friend or family member? |
| [] In a temporary housing program? |
| [] In a welfare or voucher hotel/motel? |
| [] In jail, prison, or a halfway house? |
| [] In drug treatment, a detox unit, or drug program housing? |
| [] In a hospital, nursing home, or hospice? |
| [] I have not spent a night in any of the above places. |
| Insurance |
| Shortname / Alias: insurance |
| ID: 206 |
| Do you currently have health insurance or health care coverage? ( ) Yes |
| ( ) No |
| ( ) I don't know |
| Sexual Identity, Relationships |

The following questions ask about your sexual identity and relationship status.

Please answer to the best of your ability.

| Shortname / Alias: sexualid | |
|---|---|
| ID: 102 | |
| What is your current sexual identity?* ( ) Gay, homosexual, same gender loving | |
| ( ) Bisexual | |
| () Queer | |
| ( ) Straight or heterosexual | |
| ( ) Other, specify:: | * |

Shortname / Alias: relationship

ID: 118

How do you define your primary relationship status?\*

- () Single, not currently dating
- () Single, casually dating
- () In a relationship
- () Married or other legal commitment

**Page entry logic:** This page will show when: #20 Question "How do you define your primary relationship status?" is one of the following answers ("In a relationship","Married or other legal commitment")

#### **Sexual Health Priorities with Partner**

ID: 566

People have different sexual health priorities. For example, some people prioritize staying HIV-negative; others want to have as much fun as possible with their partners; others want to feel as close and connected to their partners as possible.

For these next questions, we are interested in you and your primary romantic partner's sexual health priorities.

Shortname / Alias: shpriorities\_scale

ID: 569

Thinking about you and your partner's sexual health priorities, please indicate the extent to which you agree or disagree with the following statements.\*

| | Strongly<br>Agree | Agree | Disagree | Strongly<br>Disagree |
|---|---|---|---|---|
| I feel like my<br>partner and<br>I are "on the<br>same page"<br>in terms of<br>the<br>decisions<br>we make<br>about<br>sexual<br>health and<br>risk | () | () | () | () |
| When it comes to sexual decision-making, I feel like my partner and I are "of the same mind" | () | () | () | () |
| Sometimes I feel like my priorities for my sexual health are incompatible with my partner's goals | () | () | () | () |
| I'm confident that my partner and I generally share the same priorities when it comes to sexual health | () | () | () | () |

| Making sexual health decisions with my partner can be difficult because we | () | () | () | () |
|---|---|---|---|---|
| different<br>priorities | | | | |

#### **Health Providers**

ID: 157

Now, we are going to ask you about your health care and health care decision making.

Logic: Show/hide trigger exists.

Shortname / Alias: pcp

ID: 158

Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?\*

() Yes

() No

Logic: Hidden unless: #22 Question "Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?" is one of the following answers ("Yes")

Shortname / Alias: pcpawareness

ID: 105

How open are you about your sexual identity to your primary medical care provider?\*

- ( ) Primary medical provider definitely does NOT know your sexual identity
- ( ) Primary medical provider MIGHT know about your sexual identity
- ( ) Primary medical provider PROBABLY knows about your sexual identity
- ( ) Primary medical provider DEFINITELY knows about your sexual identity

| Logic: Hidden unless: #22 Question "Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?" is one of the following answers ("Yes") |
|---|
| Shortname / Alias: pcptalksex |
| ID: 160 |
| How comfortable are you discussing your sexual behavior with your primary health care provider?* ( ) Very comfortable ( ) Somewhat comfortable ( ) Somewhat uncomfortable ( ) Very uncomfortable |
| STI Testing |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: stitest3m |
| ID: 170 |
| A sexually transmitted infection (STI) is an infection transmitted through sexual activity, such as syphilis, gonorrhea, chlamydia, herpes, or genital warts. In the past 3 months, have you been tested for an STI that was not HIV?* () Yes () No |
| Logic: Hidden unless: #25 Question "A sexually transmitted infection (STI) is an infection transmitted through sexual activity, such as syphilis, gonorrhea, chlamydia, herpes, or genital warts. In the past 3 months, have you been tested for an STI that was not HIV?" is one of the following answers ("Yes") |
| Shortname / Alias: sti3mo |
| ID: 171 |
| Please indicate whether you have been diagnosed with any of the following sexually transmitted infections in the past 3 months. Please select all that apply.* [] Chlamydia |
| [] Genital warts, anal warts, HPV |
| [] Gonorrhea |
| [] Hepatitis B |
| [] Hepatitis C<br>[] Herpes, HSV1/HSV2 |

| [] Syphilis [] Urethritis [] Other, please specify:: [] None of these |
|---|
| HIV Testing |
| Shortname / Alias: recenthivtest_mon ID: 165 |
| When did you have your most recent HIV test? |
| Please enter the month and year. |
| Month:* () January () February () March () April () May () June () July () August () September () October () November () December |
| Validation: Min = 1980 Must be numeric Whole numbers only Positive numbers only Max character coun = 4 |
| Shortname / Alias: recenthivtest_yr ID: 166 |
| Year:* |

| Page entry logic: This page will show when: (#27 Question "When did you have your most recent HIV test? |
|---|
| Please enter the month and year. |
| Month:" AND #28 Question "Year:" ) |
| Action: Custom Script: Check HIV test date not in future |
| PrEP Use |
| Shortname / Alias: prepstartafterP3-T ID: 1201 |
| Did you start taking PrEP after you started the P3-T study?* ( ) Yes ( ) No |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: nowprep |
| ID: 1202 |
| Are you taking PrEP right now?* ( ) Yes ( ) No |
| Lawier Hidden unless. Fin lawie If we to Did you stout toking DuFD often you awalled in D2 T |
| Logic: Hidden unless: Fix logic- If no to Did you start taking PrEP after you enrolled in P3-T |
| Shortname / Alias: noprep_why ID: 1203 |
| Why did you decide not to start PrEP? Select all of the factors below that were related to why you didn't start PrEP.* [] I couldn't afford it |
| [] I was not having sex |
| [] I was no longer having sex with a person living with HIV |
| [] I was only having sex with one person and they were undetectable or HIV negative |
| [1] I didn't want to take a nill every day |
| [ ] My parent(s) or guardian(s) found out and wouldn't let me start |
|---|
| [] I kept forgetting to take my pill |
| [] I could no longer see my PrEP provider and haven't found another PrEP provider |
| [] I was worried about experiencing side effects |
| [] I was worried about the long term effects of PrEP on my health |
| [] It was medically unsafe for me to take PrEP (due to kidney/renal function, bone density, or another medical issue) |
| [] I was worried that if I were to become HIV-positive certain medications may no longer work or I might be resistant to them |
| [] I was worried that PrEP might not provide complete protection against HIV |
| [] I started using condoms all of the time |
| [] I was worried that the medication would taste bad and/or the pill would be too big |
| [] Other, please specify:: |

**Page entry logic:** This page will show when: #32 Question "Why did you decide not to take PrEP? Select all of the factors below that were related to why you didn't take PrEP."

### PrEP Use, why didn't start

Action: Custom Script: Script to count checkboxes and skip if q <2

ID: 1204

Piping: Piped Values From Question 32. (Why did you decide not to take PrEP? Select all of the factors below that were related to why you didn't take PrEP.)

Please rank the reasons you did not start taking PrEP in order of importance.\*

Page entry logic: Fix logic- If yes to Did you start taking PrEP after you enrolled in P3-T

#### **PrEP Start**

Shortname / Alias: startprep why

ID: 943

### Why did you choose to start taking PrEP? Select all that apply.\*

[] I'm having sex with or thinking about having sex with someone who is HIV+

[] I'm having sex with or thinking about having sex with someone whose HIV status I don't know

| [] I want to be in control of my sexual health |
|-----------------------------------------------------------|
| [] I want to reduce my anxiety around sex |
| [] I want to increase my sexual satisfaction and intimacy |
| [] I want to be safe and healthy |
| [] I want to have a better future |
| [] I am having sex with multiple partners |
| [] I don't like to use condoms |
| [ ] My partner won't use condoms |
| [] I had a previous HIV scare |
| [] My health care provider recommended it |
| [] I was recently diagnosed with an STI |
| [] Many people in my community take PrEP |
| [ ] Other, please specify:: |

#### **PrEP Start**

Action: Custom Script: Script to count checkboxes and skip q if < 2

Shortname / Alias: startprep\_primwhy

ID: 945

Piping: Piped Values From Question 34. (Why did you choose to start taking PrEP? Select all that apply.)

What was the main reason you started PrEP?\*

**Page entry logic:** This page will show when: (#30 Question "Did you start taking PrEP after you started the P3-T study?" is one of the following answers ("Yes") OR #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes"))

### **PrEP Start and Stop**

Validation: %s format expected

Logic: Hidden unless: #30 Question "Did you start taking PrEP after you started the P3-T study?"

is one of the following answers ("Yes")

Shortname / Alias: prep firststart

#### ID: 947

When did you start taking PrEP after enrolling in P3-T?

If you do not know the exact day of the month, please give your best estimate. \*

\_\_\_\_\_\_

Logic: Hidden unless: #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes")

Shortname / Alias: prepstoP3-Tmo

ID: 576

Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?\*

() Yes

() No

Action: Custom Script: Check date not in future

Action: Custom Script: Script to populate - 3 months date

Hidden Value: Date for prompt - today minus 3 months

Value:

**Page entry logic:** This page will show when: #37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes")

### PrEP Stop, last 3 months

Logic: Show/hide trigger exists.

Shortname / Alias: timesprepstoP3-Tmo

ID: 950

How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?\*

- ()0
- ()1
- ()2
- ()3
- ()4

| ()6 |
|---|
| ()7 |
| ()8 |
| ()9 |
| ()10 |
| ( ) 11 |
| ( ) 12 or more |
| Logic: Hidden by default |
| ID: 1159 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("1") |
| Shortname / Alias: time1_dates |
| ID: 1027 |
| Please enter the dates you were off PrEP (from [question('value'), id='1026'] to today): |
| Please enter the dates you were off PrEP (from [question('value'), id='1026'] to today): Validation: %s format expected |
| Validation: %s format expected |
| Validation: %s format expected ID: 1028 |
| Validation: %s format expected ID: 1028 Date stopped:*: |
| Validation: %s format expected ID: 1028 Date stopped:*: Validation: %s format expected |
| Validation: %s format expected ID: 1028 Date stopped:*: Validation: %s format expected ID: 1029 |
| Validation: %s format expected ID: 1028 Date stopped:*: Validation: %s format expected ID: 1029 |
| Validation: %s format expected ID: 1028 Date stopped:*: Validation: %s format expected ID: 1029 Date re-started:*: |
| Validation: %s format expected ID: 1028 Date stopped:*: Validation: %s format expected ID: 1029 Date re-started:*: Logic: Hidden by default |

()5

Shortname / Alias: timefirst\_dates

112

| | ID: 1030 |
|---|---|
| | Please enter the dates you were off PrEP for the first time (from [question('value'), id='1026'] to today): |
| | Validation: %s format expected |
| | ID: 1031 |
| | Date stopped:*: |
| | Validation: %s format expected |
| | ID: 1032 |
| | Date re-started:*: |
| Ī | |
| | Logic: Hidden by default |
| | ID: 1161 |
| | The date re-started is before the date stopped. Please correct this. |
| Ī | |
| | Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("2","3","4","5","6","7","8","9","10","11","12 or more") |
| | Shortname / Alias: timesecond_dates |
| | ID: 1033 |
| | Please enter the dates you were off PrEP for the second time (from [question('value'), id='1026'] to today): |
| | Validation: %s format expected |
| | ID: 1034 |
| | Date stopped:*: |
| | Validation: %s format expected |
| | ID: 1035 |
| | Date re-started:*: |

Logic: Hidden by default

ID: 1162

The date re-started is before the date stopped. Please correct this.

| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("3","4","5","6","7","8","9","10","11","12 or more") |
|---|
| Shortname / Alias: timethird_dates |
| ID: 1036 |
| Please enter the dates you were <u>off</u> PrEP for the <u>third</u> time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1037 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1038 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1163 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates ID: 1039 Please enter the dates you were off PrEP for the fourth time (from [question('value'), |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates ID: 1039 Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates ID: 1039 Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates ID: 1039 Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates ID: 1039 Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 Date stopped:*: |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates ID: 1039 Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 Date stopped:*: |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates ID: 1039 Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 Date stopped:*: Validation: %s format expected ID: 1041 |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefourth_dates ID: 1039 Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 Date stopped:*: Validation: %s format expected ID: 1041 |

| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") |
|---|
| Shortname / Alias: timefifth_dates |
| ID: 1042 |
| Please enter the dates you were off PrEP for the fifth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1043 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1044 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1165 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you <u>stop taking PrEP for 7 days in a row or more</u> in the last three months ( <i>from [question('value'), id='1026'] to today)</i> ?" is one of the following answers ("6","7","8","9","10","11","12 or more") |
| Shortname / Alias: timesixth_dates |
| ID: 1045 |
| Please enter the dates you were off PrEP the sixth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1046 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1047 |
| Date re-started:*: |

| ID: 1166 |
|---|
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("7","8","9","10","11","12 or more") |
| Shortname / Alias: timeseventh_dates |
| ID: 1048 |
| Please enter the dates you were off PrEP for the seventh time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1049 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1050 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1167 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("8","9","10","11","12 or more") |
| Shortname / Alias: timeeighth_dates |
| ID: 1051 |
| Please enter the dates you were <u>off</u> PrEP for the <u>eighth</u> time (from [question('value'), id='1026'] to today): |
| id='1026'] to today): |
| id='1026'] to today): Validation: %s format expected |
| id='1026'] to today): Validation: %s format expected ID: 1052 |
| <pre>id='1026'] to today): Validation: %s format expected ID: 1052 Date stopped:*:</pre> |

Logic: Hidden by default

| Logic: Hidden by default |
|---|
| ID: 1168 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("9","10","11","12 or more") |
| Shortname / Alias: timeninth_dates |
| ID: 1054 |
| Please enter the dates you were off PrEP for the ninth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1055 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1056 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1169 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a |

Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("10","11","12 or more")

Shortname / Alias: timetenth\_dates

Date re-started:\*:

ID: 1057

Please enter the dates you were off PrEP for the tenth time (from [question('value'), id='1026'] to today):\*

Validation: %s format expected

ID: 1058

| Validation: %s format expected |
|---|
| ID: 1059 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1170 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("11","12 or more") |
| Shortname / Alias: timeeleventh_dates |
| ID: 1060 |
| Please enter the dates you were off PrEP for the eleventh time (from [question('value'), id='1026'] to today):* |
| id='1026'] to today):* |
| id='1026'] to today):* Validation: %s format expected |
| id='1026'] to today):* Validation: %s format expected ID: 1061 |
| <pre>id='1026'] to today):*</pre> Validation: %s format expected ID: 1061 Date stopped:*: |
| <pre>id='1026'] to today):*</pre> Validation: %s format expected ID: 1061 Date stopped:*: Validation: %s format expected |
| <pre>id='1026'] to today):*</pre> Validation: %s format expected ID: 1061 Date stopped:*: Validation: %s format expected ID: 1062 |
| <pre>id='1026'] to today):*</pre> Validation: %s format expected ID: 1061 Date stopped:*: Validation: %s format expected ID: 1062 |
| <pre>id='1026'] to today):*</pre> Validation: %s format expected ID: 1061 Date stopped:*: Validation: %s format expected ID: 1062 |
| id='1026'] to today):* Validation: %s format expected ID: 1061 Date stopped:*: |
| id='1026'] to today):* Validation: %s format expected ID: 1061 Date stopped:*: Validation: %s format expected ID: 1062 Date re-started:*: Logic: Hidden by default ID: 1171 |
| id='1026'] to today):* Validation: %s format expected ID: 1061 Date stopped:*: Validation: %s format expected ID: 1062 Date re-started:*: Logic: Hidden by default |

Date stopped:\*:

Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("12 or more")

Shortname / Alias: timetwelfth\_dates

ID: 1063

Please enter the dates you were off PrEP for the twelfth time (from [question('value'), id='1026'] to today):\*

| Validation: %s format expected |
|--------------------------------|
| ID: 1064 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1065 |
| Date re-started:*: |

**Page entry logic:** This page will show when: ((#37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes") OR (#29 Question "When you started the P3-T study, were you taking PrEP?" is one of the following answers ("Yes") AND #31 Question "Are you taking PrEP right now?" is one of the following answers ("No"))) OR (#30 Question "Did you start taking PrEP after you started the P3-T study?" is one of the following answers ("Yes") AND #31 Question "Are you taking PrEP right now?" is one of the following answers ("No")))

### **PrEP Stop**

Logic: Hidden by default

ID: 1206

This number cannot be greater than the number of times you stopped taking PrEP for 7 days in a row or more in the last 3 months ([question('value'), id='950']). Please correct this.

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("1","2","3","4","5","6","7","8","9","10","11","12 or more")

Shortname / Alias: prepstop drconsult

ID: 578

Of the [question("value"), id="950"] times you stopped taking PrEP, how many did you talk with your medical provider about before you stopped taking PrEP?\*

\_\_\_\_\_\_

Shortname / Alias: stopprep why

ID: 581

Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP.\*

[] I couldn't afford it anymore

| [] I was not having sex |
|---|
| [] I was no longer having sex with a person living with HIV |
| [] I was only having sex with one person and they were undetectable or HIV negative |
| [] I didn't want to keep taking a pill every day |
| [] My parent(s) or guardian(s) found out and made me stop |
| [] I kept forgetting to take my pill |
| [] I haven't been able to make it to my follow-up appointments |
| [] I could no longer see my PrEP provider and haven't found another PrEP provider |
| [] I experienced side effects |
| [] I was worried about the long term effects of PrEP on my health |
| [] It was medically unsafe for me to continue taking PrEP (due to kidney/renal function, bone density, or another medical issue) |
| [] I was worried that if I were to become HIV-positive certain medications may no longer work or I might be resistant to them |
| [] I was worried that PrEP might not provide complete protection against HIV |
| [] I started using condoms all of the time |
| [] The medication tastes bad and/or the pill is too big |
| [] Other, please specify:: |

**Page entry logic:** This page will show when: #38 Question "How many times did you <u>stop taking PrEP for 7 days in a row or more</u> in the last three months (*from [question('value'), id='1026'] to today)*?" is one of the following answers ("1","2","3","4","5","6","7","8","9","10","11")

Action: Custom Script: Script to check number of times off PrEP

**Page entry logic:** This page will show when: #53 Question "Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP."

### **PrEP Stop Continued**

Action: Custom Script: Script to count checkboxes and skip if q <2

Shortname / Alias: stopprep primwhy

ID: 582

Piping: Piped Values From Question 53. (Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP.)

Please rank the reasons you stopped taking PrEP in order of importance.\*

**Page entry logic:** This page will show when: #37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes")

### PrEP Restart, current users

Shortname / Alias: restart\_why

| ID: 956 |
|---|
| Why did you choose to restart taking PrEP the last time? Select all that apply.* [] I was able to start seeing my PrEP provider again |
| [] I found a new PrEP provider |
| [] I was having issues with side effects, but I found a way to deal with them |
| [] I was having issues taking my pill every day, but I found a way to deal with it |
| [] I'm having sex with or thinking about having sex with someone who is HIV+ |
| [] I'm having sex with or thinking having sex with someone whose status HIV I don't know |
| [] I want to be in control of my sexual health |
| [] I want to reduce my anxiety around sex |
| [] I want to increase my sexual satisfaction and intimacy |
| [] I want to be safe and healthy |
| [] I want to have a better future |
| [] I am having sex with multiple partners |
| [] I don't like to use condoms |
| [] My partner won't use condoms |
| [] I had a previous HIV scare |
| [] My health care provider recommended it |
| [] I was recently diagnosed with an STI |
| [] Many people in my community take PrEP |
| [] Other, please specify:: |

**Page entry logic:** This page will show when: #55 Question "Why did you choose to restart taking PrEP the last time? Select all that apply."

### Restart reason, current users

Action: Custom Script: Script to count checkboxes and skip if q <2

Shortname / Alias: restart primwhy

ID: 957

Piping: Piped Values From Question 55. (Why did you choose to restart taking PrEP the last time? Select all that apply.)

What was the main reason you decided to restart PrEP?\*

#### **Healthcare Visits**

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Show/hide trigger exists.

Shortname / Alias: numdrvisits3m

ID: 584

In the last 3 months, how many times did you go to the doctor for any reason?\*

Logic: Hidden by default

ID: 940

This number cannot be greater than the total number of doctor's visits entered above.

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Show/hide trigger exists. Hidden unless: #57 Question "In the last 3 months, how many times did you go to the doctor for any reason?" is greater than "0"

Shortname / Alias: numprepvisits3m

ID: 586

Out of all these visits, how many were routine/scheduled PrEP appointments?\*

\_\_\_\_\_

Logic: Hidden by default

ID: 988

### This number cannot be greater than the total number of routine PrEP appointments.

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Hidden unless: #58 Question "Out of all these visits, how many were routine/scheduled PrEP appointments?" is greater than "0"

Shortname / Alias: missedprepvisits3m

ID: 587

In the last 3 months, how many of your scheduled PrEP appointments did you miss because you didn't show or forgot?

By scheduled appointments, we mean routine PrEP appointments, not walk-in or urgent care appointments for acute/urgent issues. \*

\_\_\_\_\_

Action: Custom Script: Script to check number of visits

Action: Custom Script: Script to check number of days

#### **PrEP Adherence**

Logic: Hidden unless: #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes")

Shortname / Alias: preplastweek

ID: 177

How many of the last 7 days did you take your PrEP medication?\*

- () 0 days
- () 1 day
- () 2 days
- () 3 days
- () 4 days
- () 5 days
- () 6 days
- () 7 days

Validation: Min = 0 Max = 100

Logic: Show/hide trigger exists.

| ID: 178 |
|---|
| In the last month, what percent of the time did you take your PrEP as prescribed (once a day)? Use the scale below. 0% would mean 'NONE' of the time and 100% would mean 'ALL' of the time. If you are unsure, make a guess. |
| % medication taken:* |
| 0 100 |
| PrEP Dose Barriers |
| Shortname / Alias: dose_ |
| ID: 959 |
| What has gotten in the way of you taking your PrEP on a daily basis? Please select all that apply.* [] I have not had any trouble taking PrEP on a daily basis |
| [] I get tired of taking a pill every day |
| [] I forget to take it |
| [] I don't always have my pills with me |
| [] My work/school schedule |
| [] My social life |
| [] I'm around people I don't want to take it in front of |
| [] I experience side effects |
| [] I was drinking or using drugs and I didn't take it |
| Action: Custom Script: Script to count checkboxes and skip if q <2 |
| Shortname / Alias: does_rank |
| ID: 960 |
| Piping: Piped Values From Question 62. (What has gotten in the way of you taking your PrEP on a daily basis? Please select all that apply.) |
| Please rank the things that have gotten in the way of you taking your PrEP on a daily basis.* |

### **PrEP Adherence Continued**

Shortname / Alias: prepmonth

Logic: Hidden unless: #61 Question "In the last month, what percent of the time did you take your PrEP as prescribed (once a day)? Use the scale below.

0% would mean 'NONE' of the time and 100% would mean 'ALL' of the time. If you are unsure, make a guess.

% medication taken:"

Shortname / Alias: prepadher protection

ID: 588

You said you took your PrEP [question("value"), id="178"] percent of the time in the last month. Based on this adherence level, how protected do you think you were from HIV in the last month?\*

- () Not protected at all
- () Somewhat protected
- () Mostly protected
- () Fully protected
- () Decline to answer

Shortname / Alias: prepadher\_decisionbot

ID: 589

In the last month, how much did your adherence to PrEP (if you took it every day or not) affect how often you used a condom during anal sex when you bottom?\*

- ( ) My decision about condom use when I bottom <u>was not</u> influenced by whether or not I took my pill every day
- ( ) My decision about condom use when I bottom <u>was somewhat</u> influenced by whether or not I took my pill every day
- ( ) My decision about condom use when I bottom <u>was</u> influenced by whether or not I took my pill every day

Shortname / Alias: prepadher decisiontop

ID: 590

In the last month, how much did your adherence to PrEP (if you took it every day or not) affect how often you used a condom during anal sex when you top?\*

- ( ) My decision about condom use when I top <u>was not</u> influenced by whether or not I took my pill every day
- ( ) My decision about condom use when I top <u>was somewhat</u> influenced by whether or not I took my pill every day
- ( ) My decision about condom use when I top was influenced by whether or not I took my pill every day
- () I did not top in the last month

#### **PrEP Confidence**

ID: 907

We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident).

| Validation: Min = 1 Max = 10 | |
|---------------------------------------------|------|
| Shortname / Alias: keepappts | |
| ID: 903 | |
| How confident are you that you can | |
| Keep your PrEP medical appointments:* 1[_] | _ 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: followplan ID: 904 | |
| Follow a plan for taking PrEP:* 1[_] | _ 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: atworkschool | |
| ID: 905 | |
| Take PrEP at work/school:* 1[_] | _ 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: onweekday | |
| ID: 906 | |
| Take PrEP on a weekday:* 1[_] | _ 10 |

Action: JavaScript: Hide General Error Message

# PrEP Confidence 2

| ID: 908 | |
|---|---|
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). | |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: onweekend | |
| ID: 909 | |
| How confident are you that you can | |
| Take PrEP on a weekend:* 1[_] | 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: wfriends ID: 910 | |
| Take PrEP when I'm out with friends:* 1[_] | 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: prepdrinking ID: 911 | |
| Take PrEP when I'm drinking or using drugs:* 1[_] | 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: schedulechange | |
| ID: 912 | |
| Take PrEP when my schedule changes:* | |

### **PrEP Confidence 3**

| i | ח | 9 | 1 | 3 |
|---|---|---|---|---|

ID: 597

We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident).

Right now there are no other approved options for taking PrEP. However, if there were more than one option and each method was equally good at protecting you from getting HIV, which method would you most prefer?\*

- () Taking one pill, every day
- ( ) Taking two pills before you had sex and a pill a day for the next two days
- ( ) Taking one pill a day just on Tuesday, Thursday, Saturday, and Sunday
- () Getting an injection about every 2 to 3 months
- ( ) Putting medicated lubrication (lube) in your anus (and/or your partner's anus) before having anal sex
- ( ) Douching with a medicated solution (microbicide) before having anal sex

#### **PrEP Beliefs**

Shortname / Alias: prepbeliefs

ID: 598

Please rate your agreement with the following statements:\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| People are<br>less likely<br>to use<br>condoms<br>for anal sex<br>if they are<br>using PrEP | () | () | () | () |
| I feel as if<br>starting to<br>take PrEP<br>would allow<br>me to have<br>more sex<br>partners | () | () | () | () |
| I feel as if<br>starting to<br>take PrEP<br>would allow<br>me to have<br>more<br>condomless<br>anal sex | () | () | () | () |

# **PrEP and People**

Shortname / Alias: prepppl

ID: 193

We are interested in how you feel about the following statements. Read each statement carefully

and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I worry people will assume I sleep around if they know I take PrEP | () | () | () | () |
| I worry people will assume that I am HIV- positive if they know I take PrEP | () | () | () | () |
| I worry people will think my partner(s) are HIV- positive if they know I take PrEP | () | () | () | () |
| I worry about listing PrEP as one of my current medications during appointments such as at a dentist's or specialist's office | () | () | () | () |
| I feel<br>ashamed to<br>tell other | () | () | () | () |

| | | | 1 | |
|---|---|---|---|---|
| people that I<br>am taking<br>PrEP | | | | |
| I worry people will think I am a bad person if they know I take PrEP | () | () | () | () |
| I worry people will think I am gay if they know I take PrEP | () | () | () | () |
| I worry my<br>friends will<br>find out that I<br>take PrEP | () | () | () | () |
| I worry my<br>family will<br>find out that I<br>take PrEP | () | () | () | () |
| I worry my<br>sexual<br>partners will<br>find out that I<br>take PrEP | () | () | () | () |
| I think people<br>will give me a<br>hard time if I<br>tell them I<br>take PrEP | () | () | () | () |
| I think people<br>will judge me<br>if they know I<br>am taking<br>PrEP | () | () | () | () |

# **PrEP Concerns**

Shortname / Alias: prepconc

ID: 210

We are interested in how you feel about the following statements. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| My family<br>does not<br>support me<br>taking PrEP | () | () | () | () |
| My friends<br>do not<br>support me<br>taking PrEP | () | () | () | () |
| People<br>taking PrEP<br>are<br>portrayed<br>poorly in the<br>media and<br>online | () | () | () | () |
| People in my<br>community<br>talk poorly<br>about people<br>taking PrEP | () | () | () | () |
| I feel<br>embarrassed<br>about taking<br>PrEP | () | () | () | () |
| I think I am<br>not following<br>the 'rules' of<br>my<br>community if<br>I take PrEP | () | () | () | () |
| I have been blamed by people in my community for spreading HIV through PrEP use | () | () | () | () |

| I have been | () | () | () | () |
|---|---|---|---|---|
| blamed by<br>people in my<br>community<br>for spreading<br>sexually<br>transmitted<br>infections<br>through not<br>using<br>condoms | • | | | |
| I have been<br>rejected<br>romantically<br>because I<br>take PrEP | () | () | () | () |
| I have been slut-shamed because I take PrEP (or told that I am a "Truvada-slut/whore") | () | () | () | () |
| I have been judged by a health care provider for taking PrEP | () | () | () | () |
| I don't think<br>that I need to<br>take PrEP<br>anymore | () | () | () | () |
| I have been told by a health care provider that I don't need PrEP or I shouldn't take PrEP | () | () | () | () |
| I have been<br>yelled at or<br>scolded<br>because I<br>take PrEP | () | () | () | () |

| I have been unfairly discriminated against because I take PrEP | () | () | () | () |
|---|---|---|---|---|
| I have experienced physical violence because I am taking PrEP | () | () | () | () |

Logic: Hidden unless: Question "I don't think that I need to take PrEP anymore" is one of the following answers ("Agree", "Strongly Agree")

Shortname / Alias: whydontneed

ID: 1067

| Why do you think that you do not need t | o take PrEP anymore | ?? Select all that apply.* |
|---|---|---|
|---|---|---|

- [] My relationship status changed -- I became single
- [ ] My relationship status changed -- I became monogamous (only having sex with one person)
- [] I stopped having sex with an HIV-positive person
- [] I am having less sex
- [] I am sexually inactive (I haven't been having sex for a period of time)
- [] I have started using condoms every time I have sex
- [] Other, please specify:: \_\_\_\_

#### **PrEP Difficulties**

Shortname / Alias: prepdifficulties

ID: 602

In making your decision to continue taking PrEP, please rate how much the following items

concern you.\*

| | Not at all concerned | A little<br>concerned | Concerned | Very<br>concerned |
|---|---|---|---|---|
| Getting the costs of PrEP covered (including | () | () | () | () |

| office visits or office visit copays, lab costs, transportation costs) | | | | |
|---|---|---|---|---|
| Using insurance to get coverage for PrEP costs (including office visits, lab costs) | () | () | () | () |
| Getting<br>transportation<br>to PrEP<br>appointments<br>and labs | () | () | () | () |
| Returning for PrEP follow-<br>up appointments and labs | () | () | () | () |
| Getting PrEP prescription refilled | () | () | () | () |

### **PrEP Difficulties Continued**

Shortname / Alias: prepdifficulties2

ID: 649

In making your decision to continue taking PrEP, please rate how much the following items concern you.\*

| | Not at all concerned | A little concerned | Concerned | Very<br>concerned |
|---|---|---|---|---|
| The possibility that if I were to become | () | () | () | () |

| HIV+,<br>certain<br>medications<br>might no<br>longer work<br>or I might be<br>resistant to<br>them | | | | |
|---|---|---|---|---|
| The possibility that PrEP might not provide complete protection against HIV | () | () | () | () |
| Having to talk to a health care provider about PrEP | () | () | () | () |
| Having to talk to a health care provider about my sex life | () | () | () | () |
| Experiencing side effects from PrEP | () | () | () | () |
| The long-<br>term effects<br>of PrEP on<br>my health | () | () | () | () |
| Having to<br>remember to<br>take PrEP<br>every day | () | () | () | () |
| Friends<br>finding out<br>that I am on<br>PrEP | () | () | () | () |
| Family<br>members<br>finding out | () | () | () | () |

| that I am on<br>PrEP | | | | |
|-----------------------------------------------|----|----|----|----|
| Sexual partners finding out that I am on PrEP | () | () | () | () |

Logic: Hidden unless: Question "The possibility that PrEP might not provide complete protection against HIV" is one of the following answers ("Concerned", "Very concerned")

Shortname / Alias: prepworry

ID: 665

| Why d | lo you worry | y about the | possibility that | : PrEP might | not provide | complete | protection | against |
|---|---|---|---|---|---|---|---|---|
| HIV? ( | Check all th | nat apply)* | | | | | | |

- [] I worry that the drug is not effective at preventing HIV
- [] Because I don't take PrEP every day consistently
- [] Because I feel I am at very high risk for becoming infected with HIV

| г. | O41 | | :£ |
|----|----------|--------|-----------|
| 1 | i Other. | blease | specify:: |
| | ,, | | , |

### **HIV** perceptions

Shortname / Alias: hivthoughts

ID: 667

Imagine how you would feel if you became infected with HIV. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I would<br>be afraid<br>people<br>would<br>judge me<br>when<br>they<br>learn I<br>have HIV | () | () | () | () |

| If I got infected, people would not want to have sex with me | () | () | () | () |
|---|---|---|---|---|
| I would<br>feel<br>guilty if I<br>got HIV | () | () | () | () |
| I would<br>feel<br>ashamed<br>if I got<br>HIV | () | () | () | () |

#### PEP and PrEP On-Demand

| Shortname / A | lias: pepi | 3m |
|---------------|------------|----|
|---------------|------------|----|

ID: 230

In the past 3 months, have you taken post-exposure prophylaxis (PEP) <u>AFTER</u> a sexual or drug use exposure to reduce the risk of getting HIV?\*

() Yes

() No

Shortname / Alias: prepondemand3m

ID: 674

In the past 3 months, have you taken PrEP on-demand (taking two pills before you had sex and a pill a day for the next two days)?

It is not an approved method and has not been shown to be an effective method for preventing HIV.\*

() Yes

() No

#### **Substances**

#### ID: 232

Now we'd like to ask you a little bit about your experiences using alcohol, tobacco products, and other drugs. Please be assured that this information will be treated as *strictly confidential*.

The questions will concern your experiences with using these substances in the past three months. These substances can be smoked, swallowed, snorted, inhaled, injected, or taken in the form of pills. Some of the substances may be prescribed by a doctor (like amphetamines, sedatives, or pain medications). For this survey, do not report on medications that are used as prescribed by your doctor. However, if you have taken such medications for reasons other than prescription, or taken them more frequently or at higher doses than prescribed, please report on this use. Once again, please remember that all information provided will be treated as *strictly confidential*.

Shortname / Alias: substanceuse3m

ID: 233

# Which of the following drugs have you used in the last 3 months? Please check all that apply.\*

- [] Tobacco (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)
- [] Alcohol (beer, wine, spirits, etc.)
- [] Cannabis (marijuana, pot, weed, grass, hash, synthetic cannabis, etc.)
- [] Cocaine (coke, crack, etc.)
- [] Amphetamines (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)
- [] Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)
- [] Sedatives, tranquilizers, or sleeping pills (valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)
- [] Hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)
- [ ] Opioids (heroin, morphine, methadone, codeine, Oxycotin, Percocet, Vicodin, etc.)
- [] None of these

**Page entry logic:** This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

*Please check all that apply.*" is one of the following answers ("Tobacco (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)")

### **Tobacco**

Shortname / Alias: tobacco3months

ID: 234

| cigars, e-cigarettes, etc.)?* |
|---|
| () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccodesire |
| ID: 235 |
| During the past 3 months, how often have you had a desire to use tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccoproblems |
| Shortname / Alias: tobaccoproblems ID: 236 |
| · |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* ( ) Never |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily Shortname / Alias: tobaccofailed ID: 237 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily Shortname / Alias: tobaccofailed ID: 237 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () Never |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily Shortname / Alias: tobaccofailed ID: 237 During the past 3 months, how often have you failed to do what was normally expected of you because of your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () Never () Once or twice |

| Shortname / Alias: tobaccofriend |
|---|
| ID: 238 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use o tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () No |
| () Yes |
| Shortname / Alias: tobaccostop |
| ID: 239 |
| In the last 3 months, have you tried and failed to control, cut down or stop using tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* ( ) No |
| () Yes |
| <b>Page entry logic:</b> This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? Please check all that apply." is one of the following answers ("Alcohol (beer, wine, spirits, etc.)") |
| Alcohol |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: alcohol3months |
| ID: 240 |
| In the past 3 months, how often have you used alcoholic beverages (beer, wine, spirits, etc.)?* |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

Logic: Hidden unless: #97 Question "In the past 3 months, how often have you used alcoholic beverages (beer, wine, spirits, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily","Decline to answer")

Shortname / Alias: alcoholdaily

() Daily or almost daily

| ID: 241 |
|---|
| How many drinks containing alcohol do you have on a typical day?* |
| ( ) 1 or 2 |
| () 3 or 4 |
| () 5 or 6 |
| () 7 to 9 |
| ( ) 10 or more |
| Shortname / Alias: alcoholbinge |
| ID: 242 |
| How often do you have 5 or more drinks on one occasion?* ( ) Never |
| ( ) Less than monthly |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholdesire |
| ID: 243 |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* () Never |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: alcoholproblems |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: alcoholproblems ID: 244 During the past 3 months, how often has your use of alcoholic beverages (beer, wine, spirits, etc.) led to health, social, legal or financial problems?* |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* () Never () Once or twice () Monthly () Weekly () Daily or almost daily Shortname / Alias: alcoholproblems ID: 244 During the past 3 months, how often has your use of alcoholic beverages (beer, wine, spirits, etc.) led to health, social, legal or financial problems?* () Never |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: alcoholproblems ID: 244 During the past 3 months, how often has your use of alcoholic beverages (beer, wine, spirits, etc.) led to health, social, legal or financial problems?* ( ) Never ( ) Once or twice |

| Shortname / Alias: alcoholfailed |
|---|
| ID: 245 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of alcoholic beverages (beer, wine, spirits, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholfriend |
| ID: 246 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of alcoholic beverages (beer, wine, spirits, etc.)?* () No |
| () Yes |
| Shortname / Alias: alcoholstop |
| ID: 247 |
| In the last 3 months, have you tried and failed to control, cut down or stop using alcoholic beverages (beer, wine, spirits, etc.)?* () No |
| () Yes |
| Action: JavaScript: Hide General Error Message |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? |

Please check all that apply." is one of the following answers ("Cannabis (marijuana, pot, weed, grass,

### **Cannabis**

Shortname / Alias: cannabis3months

hash, synthetic cannabis, etc.)")

# ID: 251

ID: 254

| In the past 3 months, how often have you used cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| <b>Page entry logic:</b> This page will show when: #107 Question "In the past 3 months, how often have you used cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Cannabis (cont.) |
| Shortname / Alias: cannabisdesire |
| ID: 252 |
| During the past 3 months, how often have you had a desire to use cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisproblems |
| ID: 253 |
| During the past 3 months, how often has your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisfailed |

144
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisfriend |
| ID: 255 |
| In the past 3 months, has a friend or relative or anyone else expressed concern about your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) No |
| () Yes |
| Shortname / Alias: cannabisstop |
| ID: 256 |
| In the last 3 months, have you tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* |
| () Yes |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? Please check all that apply." is one of the following answers ("Cocaine (coke, crack, etc.)") |
| Cocaine |
| Shortname / Alias: cocaine3months |
| ID: 257 |
| In the past 3 months, how often have you used cocaine (coke, crack, etc.)?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

Action: JavaScript: Hide General Error Message

**Page entry logic:** This page will show when: #113 Question "In the past 3 months, how often have you used cocaine (coke, crack, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily")

### Cocaine (cont.)

| Shortname / Alias: cocainedesire ID: 258 |
|---|
| During the past 3 months, how often have you had a desire to use cocaine (coke, crack, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cocaineproblems |
| ID: 259 |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cocainefailed |
| ID: 260 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of cocaine (coke, crack, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

| Shortname / Alias: cocainefriend |
|---|
| ID: 261 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of cocaine (coke, crack, etc.)?* () No () Yes |
| Shortname / Alias: cocainestop |
| ID: 262 |
| In the last 3 months, have you tried and failed to control, cut down or stop using cocaine (coke, crack, etc.)?* ( ) No ( ) Yes |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you use in the last 3 months? Please check all that apply." is one of the following answers ("Amphetamines (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)") |
| Amphetamine |
| Shortname / Alias: amphetamine3months |
| ID: 263 |
| In the past 3 months, how often have you used amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |

**Page entry logic:** This page will show when: #119 Question "In the past 3 months, how often have you used amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?" is one of the following answers ("Once or twice", "Monthly", "Weekly", "Daily or almost daily")

# **Amphetamine (cont.)**

| Shortname / Alias: amphetaminedesire |
|---|
| ID: 265 |
| During the past 3 months, how often have you had a desire to use amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetamineproblems |
| ID: 266 |
| During the past 3 months, how often has your use of amphetamine type stimulants (speed, methodiet pills, ecstasy, Ritalin, Adderall, etc.) led to health, social, legal or financial problems?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetaminefailed |
| ID: 267 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

| 1 | ١- | 2 | A | Q |
|---|----|---|-----|---|
| | , | | ( ) | n |

| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* |
|---|
| ( ) No |
| () Yes |

Shortname / Alias: amphetaminestop

ID: 269

In the last 3 months, have you tried and failed to control, cut down or stop using amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?\*

( ) No

() Yes

Action: JavaScript: Hide General Error Message

**Page entry logic:** This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

*Please check all that apply.*" is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)")

#### **Inhalants**

Shortname / Alias: inhalants3months

ID: 271

In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?\*

() Never

() Once or twice

() Monthly

() Weekly

() Daily or almost daily

**Action: JavaScript: Hide General Error Message** 

**Page entry logic:** This page will show when: #125 Question "In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily")

# Inhalants (cont.)

Shortname / Alias: inhalantsfriend

| Shortname / Alias: inhalantsdesire |
|---|
| ID: 272 |
| During the past 3 months, how often have you had a desire to use inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsproblems |
| ID: 273 |
| During the past 3 months, how often has your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.) led to health, social, legal or financial problems?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsfailed |
| ID: 274 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

#### ID: 275

| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of | of |
|---|---|
| inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* | |
| ( ) No | |

()Yes

### Shortname / Alias: inhalantsstop

ID: 276

In the last 3 months, have you tried and failed to control, cut down or stop using inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?\*

() No

() Yes

Action: JavaScript: Hide General Error Message

**Page entry logic:** This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

*Please check all that apply.*" is one of the following answers ("Sedatives, tranquilizers, or sleeping pills (valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)")

#### **Sedatives**

Shortname / Alias: sedatives3months

ID: 277

In the past 3 months, how often have you used sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?\*

() Never

() Once or twice

() Monthly

() Weekly

() Daily or almost daily

**Action: JavaScript: Hide General Error Message** 

**Page entry logic:** This page will show when: #131 Question "In the past 3 months, how often have you used sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily")

# **Sedatives (cont.)**

| Shortname / Alias: sedativesdesire |
|---|
| ID: 279 |
| During the past 3 months, how often have you had a desire to use sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: sedativesproblems |
| ID: 280 |
| During the past 3 months, how often has your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.) led to health, social, legal or financial problems?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: sedativesfailed |
| ID: 281 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

| Shortname / Alias: sedativesfriend |
|---|
| ID: 282 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* () No () Yes |
| Shortname / Alias: sedativesstop |
| ID: 283 |
| In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) No |
| () Yes |
| <b>Page entry logic:</b> This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? Please check all that apply." is one of the following answers ("Hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)") |
| Hallucinogens |
| Shortname / Alias: hallucinogens3months ID: 285 |
| In the past 3 months, how often have you used hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |

**Page entry logic:** This page will show when: #137 Question "In the past 3 months, how often have you used hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily")

# Hallucinogens (cont.)

| Shortname / Alias: hallucinogensdesire |
|---|
| ID: 286 |
| During the past 3 months, how often have you had a desire to use hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensproblems |
| ID: 287 |
| During the past 3 months, how often has your use of hallucinogens (LSD, acid, mushrooms, PC Ketamine, etc.) led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensfailed |
| ID: 288 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

| Shortname / Alias: hallucinogensfriend |
|---|
| ID: 289 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* |
| () Yes |
| Shortname / Alias: hallucinogensstop |
| ID: 290 |
| In the last 3 months, have you tried and failed to control, cut down or stop using hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* |
| () Yes |
| Action: JavaScript: Hide General Error Message |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used |
| in the last 3 months? Please check all that apply." is one of the following answers ("Opioids (heroin, morphine, methadone, codeine, Oxycotin, Percocet, Vicodin, etc.)") |
| Opioids |
| Shortname / Alias: opioids3months |
| ID: 291 |
| In the past 3 months, how often have you used opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |

**Page entry logic:** This page will show when: #143 Question "In the past 3 months, how often have you used opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?" is one of the following answers ("Once or twice", "Monthly", "Weekly", "Daily or almost daily")

# **Opioids (cont.)**

ID: 299

() Never

() Once or twice

Logic: Show/hide trigger exists.

Shortname / Alias: opioidsheroin

| 13.120 |
|---|
| In the past 3 months, has your opioid use included heroin?* () Yes |
| ( ) No |
| Logic: Hidden unless: #144 Question "In the past 3 months, has your opioid use included heroin?" is one of the following answers ("Yes") |
| Shortname / Alias: heroinprimary |
| ID: 300 |
| In the past 3 months, was heroin the most common opioid that you used?* () Yes |
| ( ) No |
| Shortname / Alias: opioidssdesire |
| ID: 293 |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: opioidsproblems |
| ID: 294 |
| During the past 3 months, how often has your use of opioids (heroin, morphine, methadone, |

| ( ) Monthly |
|---|
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: opioidsfailed |
| ID: 295 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: opioidsfriend |
| ID: 296 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* |
| ( ) No |
| ( ) No<br>( ) Yes |
| · · |
| · · |
| · · |
| · · |
| () Yes |
| ( ) Yes Shortname / Alias: opioidsstop |
| Shortname / Alias: opioidsstop ID: 297 In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* |
| Shortname / Alias: opioidsstop ID: 297 In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) No |
| Shortname / Alias: opioidsstop ID: 297 In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* () No () Yes |
| Shortname / Alias: opioidsstop ID: 297 In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) No |
| Shortname / Alias: opioidsstop ID: 297 In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* () No () Yes |
| Shortname / Alias: opioidsstop ID: 297 In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* () No () Yes |
| Shortname / Alias: opioidsstop ID: 297 In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* () No () Yes |

**Page exit logic:** Skip / Disqualify Logic**IF:** #151 Question "In the past 3 months, how many people have you had anal sex with?" is exactly equal to "0" **THEN:** Jump to page 120 - Perceived HIV Risk

ID: 368

The next section of questions will ask about your sexual behaviors. We know that this can be a sensitive topic, so we would like to remind you that your answers will be kept completely confidential. Please be as honest as possible in order to ensure the success of the current study.

The following questions refer to your sexual behavior during the past 3 months. Our focus will be only on anal sex. Therefore, do not include references to people with whom you did not engage in anal sex.

For these questions, anal sex refers to sex where the other person's penis was in your rectum (you were the bottom) and to sex where your penis was in the other person's rectum (you were the top).

These questions only ask about people assigned male at birth, which includes cisgender men (men assigned male at birth) and transgender women (women assigned male at birth). Therefore, do not include references to cisgender women (women assigned female at birth) or transgender men (men assigned female at birth).

Validation: Min = 0 Max = 999 Must be numeric Whole numbers only Positive numbers only

Shortname / Alias: numsexpartner

ID: 302

In the past 3 months, how many people have you had anal sex with?\*

\_\_\_\_\_

Action: JavaScript: Hide General Error Message

**Page entry logic:** This page will show when: #151 Question "In the past 3 months, how many people have you had anal sex with?" is greater than "0"

#### **HIV Status of Sexual Partners**

Logic: Hidden by default

ID: 677

The total number must equal the number of people you had anal sex with in the last 3 months ([question('value'), id='302']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: partnerhivstatus |
| ID: 676 |
| Before you had sex, what did you know of the HIV status of your sexual partner(s)? |
| Enter numerical values. Numbers must add up to [question('value'), id='302'], the number of people you reported having anal sex within the last three months.* This person/these people told you they were HIV negative and you had no reason to doubt it |
| You knew this person/these people were HIV positive |
| You were not completely sure of this person/these people's HIV status |
| Actions Contain Conints Conint to about the continuous commetatele |
| Action: Custom Script: Script to check the continuous sum totals |
| Hidden Value: Num HIV Neg partners |
| Value: [question("option value"), id="676", option="12278"] |
| Hidden Value: Num HIV Pos partners |
| Value: [question("option value"), id="676", option="12279"] |
| Hidden Value: Num HIV Unk partners |
| Value: [question("option value"), id="676", option="12280"] |
| Page entry logic: This page will show when: Num HIV Neg partners is greater than "0" |
| HIV Negative Partners |

ID: 690

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Shortname / Alias: hivneg timesbot

ID: 701

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom?\*

Shortname / Alias: hivneg\_timestop

ID: 702

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the top?\*

\_\_\_\_\_\_

**Page entry logic:** This page will show when: #153 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative <a href="https://www.where.negative-where-you were the-bottom">where you were the bottom</a>?" is greater than "0"

**HIV Negative Partners - Condomless Receptive AI** 

Logic: Hidden by default

ID: 714

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='701']). Please correct this.

Shortname / Alias: hivneg\_timesbotunp

ID: 710

In the past 3 months, how many of the [question('value'), id='701'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom were without a condom? \*

Action: Custom Script: Check number condomless is not greater than total times

**Page entry logic:** This page will show when: #155 Question "In the past 3 months, how many of the [question('value'), id='701'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom were without a condom? " is greater than "0"

# **HIV Negative Partners - Condomless Receptive Al**

ID: 721

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 999

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivneg botunp typ

ID: 711

Regarding the partners who told you they were HIV negative who you had <u>condomless receptive</u> <u>anal sex with (where you were the bottom)</u>, how many were...

| –ntor | numerical | I VAIIIDE ^ |
|-------|-------------|-------------|
| | Hulliciicai | values. |

\_\_\_\_\_Romantic partner(s), someone you are in a relationship with

\_\_\_Casual hook-up(s) or one-night stand(s)

\_\_\_\_\_A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc.

Logic: Hidden by default

ID: 1002

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivneg_botunp_gender |
| ID: 964 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |
| Astions Contain Conint Conint to also also antiques a sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| <b>Page entry logic:</b> This page will show when: #154 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the top?" is greater than "0" |
| HIV Negative Partners - Condomless Insertive Al |
| ID: 722 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative. |
| Logic: Hidden by default |
| ID: 719 |

This number cannot be greater than the number of times you had anal sex where you were the top ([question('value'), id='702']). Please correct this.

Shortname / Alias: hivneg timestopunp

ID: 718

In the past 3 months, how many of the [question('value'), id='702'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the top were without a condom? \*

Action: Custom Script: Script to check number condomless is not greater than the totals

**Page entry logic:** This page will show when: #158 Question "In the past 3 months, how many of the [question('value'), id='702'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the top were without a condom?" is greater than "0"

**HIV Negative Partners - Condomless Insertive AI** 

ID: 723

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 1004

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivneg\_topunp\_typ

ID: 725

Regarding the partners who told you they were HIV negative who you had <u>condomless insertive</u> anal sex with (where you were the top), how many were...

| Romantic partner(s), someone you are in a relationship with |
|---|
| Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, |
| etc. |
| Logic: Hidden by default |
| ID: 1005 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivneg_topunp_gender |
| ID: 965 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: Num HIV Neg partners is greater than "0" |
| HIV Negative Partners - PrEP and Alcohol and Drug Use |
| ID: 992 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative. |

Logic: Hidden by default

ID: 732

This number cannot be greater than the number of partners who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Shortname / Alias: hivneg toldyouprep

ID: 729

How many of your sexual partners who told you they were HIV negative told you they were taking PrEP?

Number must be less than or equal to [question('option value'), id='676', option='12278'].\*

\_\_\_\_\_

Logic: Show/hide trigger exists.

Shortname / Alias: hivneg\_youtoldprep

ID: 730

Regarding your sexual partners who told you they were HIV negative, did you tell any of them that you were taking PrEP?\*

- () Yes
- () No
- () I was not taking PrEP at this time

Logic: Hidden by default

ID: 733

This number cannot be greater than the number of partners who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Logic: Hidden unless: #162 Question "Regarding your sexual partners who told you they were HIV negative, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivneg youtoldprepnum

ID: 731

How many of your sexual partner(s) who told you they were HIV negative did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12278'].\*

\_\_\_\_\_

| ID: 740 |
|---|
| In the past 3 months, how many of the times you had anal sex with partners who told you they were HIV negative were you or this person under the influence of alcohol or drugs?* |
| Action: Custom Script: Script to check PrEP number not greater than the total number of partners |
| Action: Custom Script: Script to check PrEP number not greater than the total number of partners |
| Page entry logic: This page will show when: Num HIV Pos partners is greater than "0" |
| HIV Positive Partners |
| ID: 770 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive. |
| Shortname / Alias: hivpos_timesbot ID: 775 |
| In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom?* |
| Shortname / Alias: hivpos_timestop |

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the top?\*

\_\_\_\_\_

**Page entry logic:** This page will show when: #165 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom?" is greater than "0"

# **HIV Positive Partners - Condomless Receptive AI**

ID: 782

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 783

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='775']). Please correct this.

Shortname / Alias: hivpos timesbotunp

ID: 784

In the past 3 months, how many of the [question('value'), id='775'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom were without a condom? \*

\_\_\_\_\_

Action: Custom Script: Check number condomless is not greater than total times

**Page entry logic:** This page will show when: #167 Question "In the past 3 months, how many of the [question('value'), id='775'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom were without a condom? " is greater than "0"

| ID: 786 |
|---------|
|---------|

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 1008

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivpos\_botunp\_typ

ID: 788

Regarding the partners who told you they were HIV positive who you had <u>condomless receptive</u> <u>anal sex with (where you were the bottom)</u>, how many were...

#### Enter numerical values.\*

\_\_\_\_\_Romantic partner(s), someone you are in a relationship with \_\_\_\_\_Casual hook-up(s) or one-night stand(s)

\_\_\_\_A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc.

#### Logic: Hidden by default

ID: 1009

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivpos botunp gender

ID: 994

How many were...

#### Enter numerical values.\*

\_\_\_Men

| TranswomenNon-binary, genderqueer, and gender non-conforming |
|---|
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| <b>Page entry logic:</b> This page will show when: #166 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the top?" is greater than "0" |
| HIV Pos Partners - Condomless Insertive Al |
| ID: 792 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive. |
| Logic: Hidden by default |
| ID: 793 |
| This number cannot be greater than the number of times you had anal sex where you were the top ([question('value'), id='776']). Please correct this. |
| Shortname / Alias: hivpos_timestopunp ID: 794 |
| In the past 3 months, how many of the [question('value'), id='776'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the top were without a condom? * |

Action: Custom Script: Script to check number condomless is not greater than the totals

**Page entry logic:** This page will show when: #170 Question "In the past 3 months, how many of the [question('value'), id='776'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the top were without a condom? " is greater than "0"

### **HIV Positive Partners - Condomless Insertive AI**

ID: 796

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 1012

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivpos\_topunp\_typ

ID: 798

Regarding the partners who told you they were HIV positive who you had <u>condomless insertive</u> anal sex with (where you were the top), how many were...

| ⊨nter | numeri | ical v | /alıı | ac * |
|-------|--------|--------|-------|------|

| | Romantic partner(s), someone you are in a relationship with |
|---|---|
| | Casual hook-up(s) or one-night stand(s) |
| | A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, |
| oto | |

Logic: Hidden by default

ID: 1013

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivpos_topunp_gender |
| ID: 995 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action. Oustoin Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: Num HIV Pos partners is greater than "0" |
| age entry logic. This page will show when. Num this is greater than o |
| HIV Positive Partners - HIV Trt and PrEP |
| Logic: Hidden by default |
| ID: 799 |
| This number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this. |
| Shortname / Alias: hivpos_toldyouhivmeds |
| ID: 800 |
| How many of your sexual partners who told you they were HIV positive told you they were taking medication to treat HIV? Number must be less than or equal to [question('option value'), id='676', option='12279']. |
| Logic: Hidden by default |
| ID: 920 |

The number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Shortname / Alias: hivpos toldyouundetect

ID: 918

How many of your sexual partners who told you they were HIV positive told you they were undetectable?

Number must be less than or equal to [question('option value'), id='676', option='12279'].

Logic: Show/hide trigger exists.

Shortname / Alias: hivpos youtoldprep

ID: 801

Regarding your sexual partners who told you they were HIV positive, did you tell any of them that you were taking PrEP?\*

- ()Yes
- () No
- () I was not taking PrEP at this time

Logic: Hidden by default

ID: 802

This number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Logic: Hidden unless: #175 Question "Regarding your sexual partners who told you they were HIV positive, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivpos youtoldprepnum

ID: 803

How many of your sexual partner(s) who told you they were HIV positive did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12279'].

\_\_\_\_\_\_

Shortname / Alias: hivpos\_timesdrunk

| ID: 807 |
|---|
| In the past 3 months, how many of the times you had anal sex with partners who told you they were HIV positive were you or this person under the influence of alcohol or drugs?* |
| Action: JavaScript: Hide General Error Message |
| Action: Custom Script: Script to check med number not greater than the total number of partners |
| Action: Custom Script: Script to check undetectable number not greater than the total number of partners |
| Action: Custom Script: Script to check PrEP number not greater than the total number of partners |

Page entry logic: This page will show when: Num HIV Unk partners is greater than "0"

### **HIV Status Unknown Partners**

ID: 810

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Shortname / Alias: hivunk timesbot

ID: 815

In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom?\*

Shortname / Alias: hivunk timestop

ID: 816

In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?\*

\_\_\_\_\_

**Page entry logic:** This page will show when: #178 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of <a href="where you were the">where you were the</a> bottom?" is greater than "0"

# **HIV Status Unknown Partners - Condomless Receptive AI**

ID: 822

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 823

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='815']). Please correct this.

Shortname / Alias: hivunk timesbotunp

ID: 824

In the past 3 months, how many of the [question('value'), id='815'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom were without a condom? \*

Action: Custom Script: Check number condomless is not greater than total times

**Page entry logic:** This page will show when: #180 Question "In the past 3 months, how many of the [question('value'), id='815'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom were without a condom? " is greater than "0"

# **HIV Status Unknown Partners - Condomless Receptive Al**

ID: 826

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 1016

The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivunk botunp typ

ID: 828

Regarding the partners whose HIV status you were not sure of who you had <u>condomless</u> receptive anal sex with (where you were the bottom), how many were...

| Entar | numorical | 1 ./~! | <br>* |
|-------|-----------|--------|-------|

\_\_\_\_\_Romantic partner(s), someone you are in a relationship with
\_\_\_\_\_Casual hook-up(s) or one-night stand(s)

A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs,

Logic: Hidden by default

ID: 1017

etc.

The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Validation: Must be numeric

| Shortname / Alias: hivunk_botunp_gender ID: 996 How many were Enter numerical values.* MenTranswomenNon-binary, genderqueer, or gender non-conforming Action: Custom Script: Script to check continuous sum totals Action: Custom Script: Script to check continuous sum totals Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive Al ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
|---|---|
| How many were Enter numerical values.* Men Transwomen Non-binary, genderqueer, or gender non-conforming Action: Custom Script: Script to check continuous sum totals Action: Custom Script: Script to check continuous sum totals Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | Shortname / Alias: hivunk_botunp_gender |
| Enter numerical values.* MenTranswomenNon-binary, genderqueer, or gender non-conforming Action: Custom Script: Script to check continuous sum totals Action: Custom Script: Script to check continuous sum totals Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s), whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | ID: 996 |
| Men | How many were |
| Transwomen Non-binary, genderqueer, or gender non-conforming Action: Custom Script: Script to check continuous sum totals Action: Custom Script: Script to check continuous sum totals Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| Action: Custom Script: Script to check continuous sum totals Action: Custom Script: Script to check continuous sum totals Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| Action: Custom Script: Script to check continuous sum totals Action: Custom Script: Script to check continuous sum totals Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | Non-binary, genderqueer, or gender non-comorming |
| Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | Action: Custom Script: Script to check continuous sum totals |
| you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0" HIV Status Unknown Partners - Condomless Insertive AI ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the |
| ID: 832 The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | HIV Status Unknown Partners - Condomiess Insertive Al |
| The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | ID: 832 |
| option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. Logic: Hidden by default ID: 833 This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | 10.002 |
| This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure |
| This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | Logic: Hidden by default |
| whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | ID: 833 |
| whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this. | |
| Shortname / Alias: hivunk timestopunp | whose HIV status you were not sure of where you were the top ([question('value'), id='816']). |
| Shortname / Alias: hivunk timestopunp | |
| | Shortname / Alias: hivunk timestopunp |

ID: 834

| In the past 3 months, how many of the [question('value'), id='816'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top were without a condom?* |
|---|
| Action: Custom Script: Script to check number condomless is not greater than the totals |
| <b>Page entry logic:</b> This page will show when: #183 Question "In the past 3 months, how many of the [question('value'), id='816'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top were without a condom?" is greater than "0" |
| HIV Status Unknown Partners - Condomless Insertive Al |
| ID: 836 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. |
| Logic: Hidden by default |
| ID: 1020 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivunk_topunp_typ |
| ID: 838 |
| Regarding the partners whose HIV status you were not sure of who you had <u>condomless</u> <u>insertive anal sex with (where you were the top)</u> , how many were |
| Enter numerical values.* Romantic partner(s), someone you are in a relationship with |
| Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, |
| etc |

Logic: Hidden by default ID: 1021 The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. Validation: Must be numeric Shortname / Alias: hivunk topunp gender ID: 997 How many were... Enter numerical values.\* Men Transwomen Non-binary, genderqueer, or gender non-conforming Action: Custom Script: Script to check continuous sum totals **Action: Custom Script: Script to check continuous sum totals** Page entry logic: This page will show when: Num HIV Unk partners is greater than "0"

### **HIV Status Unknown Partners - PrEP**

Logic: Hidden by default

ID: 839

This number cannot be greater than the number of partners whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Shortname / Alias: hivunk\_toldyouprep

ID: 840

How many of your sexual partners whose HIV status you were not sure of told you they were taking PrEP?

Number must be less than or equal to [question('option value'), id='676', option='12280'].\*

Logic: Show/hide trigger exists.

Shortname / Alias: hivunk\_youtoldprep

ID: 841

Regarding your sexual partners whose HIV status you were not sure of, did you tell any of them that you were taking PrEP?\*

- () Yes
- () No
- () I was not taking PrEP at this time

Logic: Hidden by default

ID: 842

This number cannot be greater than the number of partners whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Logic: Hidden unless: #187 Question "Regarding your sexual partners whose HIV status you were not sure of, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivunk youtoldprepnum

ID: 843

How many of your sexual partner(s) whose HIV status you were not sure of did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12280'].\*

\_\_\_\_\_

Shortname / Alias: hivunk timesdrunk

ID: 847

In the past 3 months, how many of the times you had anal sex with partners whose HIV status you were not sure of were you or this person under the influence of alcohol or drugs?\*

\_\_\_\_\_\_

| <b>Action: Custom Script: Script to che</b> | ck PrEP number not greater than the | total number of partners |
|---|---|---|
|---|---|---|

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

#### **Perceived HIV Risk**

Shortname / Alias: perceivedrisk1

ID: 762

Based on your reported sexual activities over the last 3 months, how at risk do you think you were for contracting HIV in the last 3 months?\*

- () Not at all at risk for contracting HIV
- () Somewhat at risk for contracting HIV
- () High risk for contracting HIV

Shortname / Alias: perceivedrisk2

ID: 763

What is your gut feeling about how likely you are to get infected with HIV?\*

- () Extremely unlikely
- () Very unlikely
- () Somewhat likely
- () Very likely
- () Extremely likely

Shortname / Alias: perceivedrisk3

ID: 764

### I worry about getting infected with HIV:\*

- () None of the time
- () Rarely
- () Some of the time
- () A moderate amount of time
- () A lot of the time
- () All of the time
# Perceived HIV Risk

ID: 768

| PHQ-2/GAD-2 |
|---|
| () Very large |
| () Large |
| ( ) Moderate |
| () Small |
| ( ) Almost zero |
| I think my chances of getting infected with HIV are:* ( ) Zero |
| ID: 767 |
| Shortname / Alias: perceivedrisk6 |
| ( ) Strongly Agree |
| () Agree |
| () Disagree |
| There is a chance, no matter how small, I could get HIV:* ( ) Strongly Disagree |
| ID: 766 |
| Shortname / Alias: perceivedrisk5 |
| ( ) Extremely concerned about |
| ( ) Concerned about a lot |
| ( ) Moderately concerned about |
| ( ) A little concerned about |
| ( ) Not concerned about |
| Getting HIV is something I am* |
| ID: 765 |
| Shortname / Alias: perceivedrisk4 |

Now we are going to ask you about your mental health and how you have been feeling recently.

Shortname / Alias: mentalhealthscreener

ID: 388

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Little interest or pleasure in doing things | () | () | () | () |
| Feeling<br>down,<br>depressed,<br>or<br>hopeless | () | () | () | () |
| Feeling<br>nervous,<br>anxious or<br>on edge | () | () | () | () |
| Not being<br>able to<br>stop or<br>control<br>worrying | () | () | () | () |

Page entry logic: This page will show when: psychdistress1 is greater than or equal to "3"

### PHQ-8

Shortname / Alias: phq8

ID: 397

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Trouble falling or staying asleep, or sleeping too much | () | () | () | () |
| Feeling tired<br>or having<br>little energy | () | () | () | () |
| Poor appetite or overeating | () | () | () | () |
| Feeling bad<br>about<br>yourself - or<br>that you are<br>a failure or<br>have let<br>yourself or<br>your family<br>down | () | () | () | () |
| Trouble concentrating on things, such as reading the newspaper or watching television | () | () | () | () |
| Moving or speaking so slowly that other people could have noticed, or the opposite - being so fidgety or restless that you have been moving around a lot | () | () | () | () |

| more than<br>usual |
|--------------------|
|--------------------|

Page entry logic: This page will show when: psychdistress2 is greater than or equal to "3"

### GAD-7

Shortname / Alias: gad7

ID: 404

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Worrying<br>too much<br>about<br>different<br>things | () | () | () | () |
| Trouble relaxing | () | () | () | () |
| Being so<br>restless<br>that it is<br>hard to sit<br>still | () | () | () | () |
| Becoming<br>easily<br>annoyed<br>or irritable | () | () | () | () |
| Feeling<br>afraid as if<br>something<br>awful<br>might<br>happen | () | () | () | () |

### **Social Isolation**

Shortname / Alias: socialisolation

ID: 432

Please respond to each item by marking one circle per row.\*

| | i lease respond to each item by marking one circle per row. | | | | |
|---|---|---|---|---|---|
| | Never | Rarely | Sometimes | Usually | Always |
| I feel<br>left out. | () | () | () | () | () |
| I feel<br>that<br>people<br>barely<br>know<br>me. | () | () | () | () | () |
| I feel<br>isolated<br>from<br>others. | () | () | () | () | () |
| I feel<br>that<br>people<br>are<br>around<br>me but<br>not with<br>me. | () | () | () | () | () |

# **Emotional Support**

Shortname / Alias: emotional support

ID: 411

| 1 loads respond to such item by marking one on ole per row. | | | | | |
|---|---|---|---|---|---|
| - | Never | Rarely | Sometimes | Usually | Always |
| | 110101 | itaioiy | Comounio | Codding | muyo |

| I have someone who will listen to me when I need to talk. | () | () | () | () | () |
|---|---|---|---|---|---|
| I have someone to confide in or talk to about myself or my problems. | () | () | () | () | () |
| I have<br>someone<br>who makes<br>me feel<br>appreciated. | () | () | () | () | () |
| I have<br>someone to<br>talk with<br>when I have<br>a bad day. | () | () | () | () | () |

# **Informational Support**

Shortname / Alias: informationalsupport

ID: 417

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| I have someone to give me good advice about a crisis if I need it. | () | () | () | () | () |
| I have someone to | () | () | () | () | () |

| turn to for<br>suggestions<br>about how<br>to deal with<br>a problem. | | | | | |
|---|---|---|---|---|---|
| I have someone to give me information if I need it. | () | () | () | () | () |
| I get useful<br>advice<br>about<br>important<br>things in<br>life. | () | () | () | () | () |

# **Instrumental Support**

Shortname / Alias: instrumentalsupport

ID: 422

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| Do you have someone to help you if you are confined to bed? | () | () | () | () | () |
| Do you have someone to take you to the doctor if you need it? | () | () | () | () | () |

| Do you have someone to help with your daily chores if you are sick? | () | () | () | () | () |
|---|---|---|---|---|---|
| Do you have someone to run errands if you need it? | () | () | () | () | () |

# Companionship

Shortname / Alias: companionship

ID: 427

| riease respond to each item by marking one circle per row. | | | | | |
|---|---|---|---|---|---|
| | Never | Rarely | Sometimes | Usually | Always |
| Do you have someone with whom to have fun? | () | () | () | () | () |
| Do you have someone with whom to relax? | () | () | () | () | () |
| Do you have someone with whom you can do something enjoyable? | () | () | () | () | () |
| Do you find companionship when you want it? | () | () | () | () | () |

**Page entry logic:** This page will show when: #1 Question "Enter Study Arm for testing survey (will switch to staff login before launch):" is one of the following answers ("P3 Intervention", "P3-T+ (WITH COUNSELOR) Intervention")

### **P3-T App Questions, Content**

Shortname / Alias: P3-T\_1

ID: 1072

The following questions ask about the content in P3-T. Please rate how strongly you agree or

disagree with the following statements:\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I trust the information in P3-T | () | () | () | () |
| The information in P3-T is easy to understand | () | () | () | () |
| The information in P3-T is accurate | () | () | () | () |

Page entry logic: Fix

## P3-T App Questions, Experience

Shortname / Alias: P3-T\_2

ID: 1076

The following questions ask about the content in P3-T. Please rate how strongly you agree or

disagree with the following statements:\*

| | tile lollowill | | <u>-</u> | |
|---|---|---|---|---|
| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
| P3-T helps<br>me to<br>quickly find<br>information<br>and<br>support for<br>healthy<br>living | () | () | () | () |
| P3-T helps<br>me make<br>healthier<br>choices in<br>my life | () | () | () | () |
| P3-T helps<br>me deal<br>with health<br>challenges<br>that might<br>come up | () | () | () | () |
| P3-T is<br>useful to<br>me | () | () | () | () |

Page entry logic: Fix

## P3-T App Questions, Satisfaction

Shortname / Alias: P3-T\_3

ID: 1081

The following questions ask about the content in P3-T. Please rate how strongly you agree or

disagree with the following statements:\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| Overall, I<br>am very | () | () | () | () |

| satisfied<br>with P3-T | | | | |
|-----------------------------------------------|----|----|----|----|
| Using P3-T is very frustrating | () | () | () | () |
| I would<br>recommend<br>P3-T to my<br>friends | () | () | () | () |

Page entry logic: Fix

### **P3-T App Questions, Opinions**

Validation: Max. answers = 2 (if answered)

Shortname / Alias: leastP3-T

ID: 1089

#### Which two things did you like <u>least</u> about P3-T?\*

[] Medication tracker

[] Quests

[] Social wall

[] Knowledge center

[] Collections (written stories)

[] Collections (video)

[] Adherence counselor

[] Decline to answer

Validation: Max. answers = 2 (if answered)

Shortname / Alias: bestP3-T

ID: 1090

#### Which two things did you like <u>best</u> about P3-T?\*

[] Medication tracker

[] Quests

[] Social wall

| [] Knowledge center | |
|----------------------------------|-----|
| [] Collections (written stories) | |
| [] Collections (video) | |
| [] Adherence counselor | |
| [] Decline to answer | |
| OL / /All DO TL II | |
| Shortname / Alias: P3-Tbetter | |
| ID: 1093 | |
| | ·?* |
| ID: 1093 | ·?* |
| ID: 1093 | ·?* |

**Page entry logic:** This page will show when: #1 Question "Enter Study Arm for testing survey (will switch to staff login before launch):" is one of the following answers ("P3-T Intervention","P3-T+ (WITH COUNSELOR) Intervention")

## **P3-T Opinions**

Shortname / Alias: P3-T\_4

ID: 1094

Please indicate your agreement with the following statements:\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I think that I<br>would like to<br>use P3-T<br>frequently | () | () | () | () |
| I found P3-T<br>unnecessarily<br>complex | () | () | () | () |
| I thought P3-<br>T was easy<br>to use | () | () | () | () |

| I think that I would need the support of a technical person to be able to use P3-T | () | () | () | () |
|---|---|---|---|---|
| I found the various functions in P3-T were well integrated | () | () | () | () |
| I thought<br>there was too<br>much<br>inconsistency<br>in P3-T | () | () | () | () |
| I imagine that<br>most people<br>would learn<br>to use P3-T<br>very quickly | () | () | () | () |
| I found P3-T<br>very<br>cumbersome<br>to use | () | () | () | () |
| I felt very<br>confident<br>using P3-T | () | () | () | () |
| I needed to learn a lot of things before I could get going with P3-T | () | () | () | () |
| I would use<br>P3-T in the<br>future if it<br>were<br>available. | | | | |

If P3-T were available in the app store, how much would you be willing to pay for it?

| Dage | | | . r: |
|------|-------|-------|-------|
| raye | entry | logic | . PIX |

### **P3-T Opinions**

Shortname / Alias: qualityP3-T

ID: 1107

How would you rate the quality of the help you have received from P3-T?\*

- () Excellent
- () Good
- () Fair
- () Poor

Shortname / Alias: appwanted

ID: 1108

Did you get the kind of help and/or support you wanted from P3-T?\*

- () No, definitely not
- () No, not really
- () Yes, generally
- () Yes, definitely

Shortname / Alias: metneeds

ID: 1109

To what extent has P3-T met your needs related to improving taking your meds?\*

- () Almost all of my needs have been met
- () Most of my needs have been met
- () Only a few of my needs have been met
- () None of my needs have been met

Shortname / Alias: recommendP3-T

ID: 1110

If a friend were in need of similar help, would you recommend P3-T to them?\*

() No, definitely not

| ( ) Yes, I think so |
|---|
| () Yes, definitely |
| Page entry logic: Fix |
| P3-T Opinions |
| Shortname / Alias: satisfiedhelp |
| ID: 1111 |
| How satisfied are you with the amount of help taking your meds you have received from P3-T?* ( ) Quite dissatisfied |
| ( ) Indifferent or mildly dissatisfied |
| ( ) Mostly satisfied |
| () Very satisfied |
| Shortname / Alias: effectiveP3-T |
| ID: 1112 |
| Has P3-T helped you to deal with the challenges you've faced taking PrEP?* |
| ( ) Yes, they helped a great deal |
| () Yes, they helped |
| ( ) No, they really didn't help |
| ( ) No, they seemed to make things worse |
| Shortname / Alias: satisfiedP3-T |
| ID: 1113 |
| In an overall, general sense, how satisfied are you with P3-T?* ( ) Very satisfied |
| ( ) Mostly satisfied |
| ( ) Indifferent or mildly dissatisfied |
| Shortname / Alias: returnP3-T |
| ID: 1114 |

() No, I don't think so

| greement witl | h the followin | ıg stateme | ents: |
|---|---|---|---|
| Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
| () | () | () | () |
| () | () | () | () |
| () | () | () | () |
| () | () | () | () |
| () | () | () | () |
| () | () | () | () |
| () | () | () | () |
| | Strongly Disagree () () () () () | Strongly Disagree Disagree () () () () () () () () () () () () | Disagree Agree () () () () () () () () () () () () () () |

If you were having trouble taking your meds in the future, would you use P3-T again?\* ( ) No, definitely not

( ) No, I don't think so

( ) Yes, I think so( ) Yes, definitely

Please indicate your agreement with the following statement:

| | f | | | |
|---|---|---|---|---|
| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
| I understand how to use all the features in P3-T. | () | () | () | () |
| I think P3-T would be<br>a positive addition for<br>young people on<br>PrEP. | () | () | () | () |
| It is easy to navigate within P3-T. | () | () | () | () |
| I like the look of P3-<br>T. | () | () | () | () |
| Everyone on PrEP should have P3-T. | () | () | () | () |

If to "everyone on PrEP should have P3-T" answers strongly agree-undecided, then ask,

| Who would | P3-T be | best for? | Check all | that apply. |
|-----------|---------|-----------|-----------|-------------|
|-----------|---------|-----------|-----------|-------------|

| ( | , | ) F | 'eo | ple | star | tina | PrEP |
|---|---|-----|-----|-----|------|------|------|

- () People who have been on PrEP more than 6 monghts
- () People having trouble taking PrEP
- () People who are taking PrEP regularly

| ( | ) Other: |
|---|----------|
|---|----------|

If to "everyone on PrEP should have P3-T" answers disagree-strongly disagree, then ask,

#### Who would P3-T not be good for? Check all the apply.

- () People starting PrEP
- () People who have been on PrEP more than 6 months

| Page entry logic: Fix |
|------------------------------------------|
| ( ) Other: |
| ( ) People who are taking PrEP regularly |

## **P3-T Informational Support**

() People having trouble taking PrEP

Shortname / Alias: P3-Tinformationalsupport

ID: 1122

Please respond to each item by marking one circle per row.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| The P3-T<br>app gives<br>me good<br>advice<br>about a<br>crisis if I<br>need it | () | () | () | () | () |
| The P3-T app gives me suggestions about how to deal with a problem | () | () | () | () | () |
| The P3-T app gives me information if I need it | () | () | () | () | () |
| The P3-T app gives me useful advice about important things in life | () | () | () | () | () |

Action: JavaScript: Hide General Error Message

Page entry logic: Fix

### **P3-T Social Isolation**

Shortname / Alias: P3-Tisolation

ID: 1131

Please respond to each item by marking one circle per row.\*

| i icase respond | lo cacii | | irking one circle | | 1 |
|---|---|---|---|---|---|
| | Never | Rarely | Sometimes | Usually | Always |
| In P3-T, I<br>feel left out | () | () | () | () | () |
| In P3-T, I<br>feel that<br>people<br>barely know<br>me | () | () | () | () | () |
| In P3-T, I<br>feel isolated<br>from others | () | () | () | () | () |
| In P3-T, I<br>feel that<br>people are<br>around me<br>but not with<br>me | () | () | () | () | () |

| | Strongl<br>y<br>Disagre<br>e | Disagre<br>e | Agre<br>e | Strongl<br>y Agree |
|---|---|---|---|---|
| It was easy to schedule with the adherence counselor. | () | () | () | () |

| The adherence counselor helped me take PrEP more regularly. | () | () | () | () |
|---|---|---|---|---|
| The adherence counselor helped me solve problems I had taking PrEP. | | | | |
| Talking to the adherence counselor was useful. | | | | |
| I trusted the information and advice from the adherence counselor. | | | | |
| The adherence counselor was responsive and reliable. | | | | |

Page entry logic: Fix

## **P3-T Virtual Community**

ID: 1186

The following questions regard your experience with other users of the P3-T app. Group refers to

the community of users on the P3-T app.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I think this<br>group is a<br>good<br>place for<br>me to be a<br>member. | () | () | () | () |

| I feel at<br>home in<br>this group. | () | () | () | () |
|---|---|---|---|---|
| It is very important to me to be a member of this group. | () | () | () | () |
| I anticipate how some members will react to certain questions or issues in this group. | () | () | () | () |
| I get a lot<br>out of<br>being in<br>this group. | () | () | () | () |
| l've had<br>questions<br>that have<br>been<br>answered<br>by this<br>group. | () | () | () | () |
| I've gotten<br>support<br>from this<br>group. | () | () | () | () |
| Some members of this group seem to have friendships with each other. | () | () | () | () |
| I have<br>friends in<br>this group. | () | () | () | () |

| Some members of this group can be counted on to help others by providing support or answering questions. | () | () | () | () |
|---|---|---|---|---|
| I feel obligated to help others in this group by providing support or answering questions. | () | () | () | () |
| I really like<br>this group. | () | () | () | () |
| This group<br>means a<br>lot to me. | () | () | () | () |

## Thank You!

ID: 1

Thank you for taking this survey and for participating! We greatly appreciate your involvement!

### P3-T RCT Month-3 Follow-up (SOC Arm)

Shortname / Alias: studyarm

ID: 1071

Enter Study Arm for testing survey (will switch to staff login before launch):

- () P3-T Arm
- () Standard of Care Arm

ID: 93

Thank you for participating in the P3-T study! The purpose of the study is to test a PrEP adherence intervention for young men who have sex with men who are starting PrEP. As part of the P3-T study, there are three surveys: one when you enrolled, one at your follow up appointment today, and one at your follow up appointment in 3 months.

Try to answer every question as best you can. If you need help, please ask the study staff. Your answers will be used only for research purposes. Let's get started!

#### **Cell Phone**

ID: 120

Now, we'd like to ask you about your cell phone and internet use.

Logic: Show/hide trigger exists.

Shortname / Alias: paychange

ID: 1068

In the last 3 months, has who pays for your cellphone or smart phone changed?\*

- () Yes
- () No

Logic: Hidden unless: #2 Question "In the last 3 months, has who pays for your cellphone or smart phone changed?" is one of the following answers ("Yes")

Shortname / Alias: phonepay

ID: 127

| Who usually pays for your cell phone or smartphone plan?* ( ) I do |
|---|
| () Someone else does |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: disconnect |
| ID: 128 |
| In the last 3 months, did you ever not have access to your phone or phone service?* ( ) Yes |
| ( ) No |
| Logic: Hidden unless: #4 Question "In the last 3 months, did you ever not have access to your phone or phone service?" is one of the following answers ("Yes") |
| Shortname / Alias: disconnecttimes |
| ID: 129 |
| How many times in the last 3 months did you not have access to your phone or phone service?* ( ) Once |
| () Twice |
| ( ) 3 to 5 times |
| () More than 5 times |
| Logic: Hidden unless: #4 Question "In the last 3 months, did you ever not have access to your phone or phone service?" is one of the following answers ("Yes") |
| Shortname / Alias: disconnectlength |
| ID: 130 |
| The <i>last</i> time you did not have access to your phone or phone service, for how long did you not have access?* ( ) 1 day or less |
| ( ) 2 to 6 days |
| () 1 to 4 weeks |
| () More than 4 weeks |

| Logic: Show/hide trigger exists. |
|---|
| Shortname / Alias: employed |
| ID: 109 |
| Are you currently employed?* ( ) Yes ( ) No |
| Logic: Hidden unless: #7 Question "Are you currently employed?" is one of the following answers ("Yes") |
| Shortname / Alias: employedhours |
| ID: 110 |
| Are you employed full-time or part-time? Part-time means that you work less than 35 hours per week during most weeks.* ( ) Full time ( ) Part time |
| Shortname / Alias: income_30d |
| ID: 564 |
| How much money did you make altogether during the past 30 days?* |
| ( ) Don't know |
| Shortname / Alias: incomelevel |
| ID: 111 |
| How would you describe your income level?* ( ) Low income ( ) Middle income ( ) High income |
| Food, Shelter |

# Shortname / Alias: cutmeal

| ID: 112 |
|---|
| In the past 3 months, how often did you or your family have to cut meal size or skip a meal because there was not enough money for food?* ( ) Almost every week |
| ( ) Several weeks but not every week |
| ( ) Only a few weeks |
| ( ) Did not have to skip or cut the size of meals |
| Shortname / Alias: shelter |
| ID: 113 |
| In the past 3 months, have you spent at least one night (check all that apply):* [] In a shelter? |
| [] In a public place not intended for sleeping (e.g., bus station, car, abandoned building)? |
| [] On the street or anywhere outside (e.g., park, sidewalk)? |
| [] Temporarily doubled up with a friend or family member? |
| [ ] In a temporary housing program? |
| [] In a welfare or voucher hotel/motel? |
| [] In jail, prison, or a halfway house? |
| [] In drug treatment, a detox unit, or drug program housing? |
| [] In a hospital, nursing home, or hospice? |
| [] I have not spent a night in any of the above places. |
| Insurance |
| Shortname / Alias: insurance |
| ID: 206 |
| Do you currently have health insurance or health care coverage? () Yes |

# Sexual Identity, Relationships

( ) No

() I don't know

#### ID: 565

The following questions ask about your sexual identity and relationship status.

Please answer to the best of your ability.

Shortname / Alias: sexualid

ID: 102

#### What is your current sexual identity?\*

- () Gay, homosexual, same gender loving
- () Bisexual
- () Queer
- () Straight or heterosexual
- ( ) Other, specify:: \_\_\_\_\_\_\_\*

Shortname / Alias: relationship

ID: 118

### How do you define your primary relationship status?\*

- () Single, not currently dating
- () Single, casually dating
- () In a relationship
- () Married or other legal commitment

**Page entry logic:** This page will show when: #20 Question "How do you define your primary relationship status?" is one of the following answers ("In a relationship","Married or other legal commitment")

#### **Sexual Health Priorities with Partner**

ID: 566

People have different sexual health priorities. For example, some people prioritize staying HIV-negative; others want to have as much fun as possible with their partners; others want to feel as close and connected to their partners as possible.

For these next questions, we are interested in you and your primary romantic partner's sexual health priorities.

Shortname / Alias: shpriorities\_scale

ID: 569

Thinking about you and your partner's sexual health priorities, please indicate the extent to which you agree or disagree with the following statements.\*

| | Strongly<br>Agree | Agree | Disagree | Strongly<br>Disagree |
|---|---|---|---|---|
| I feel like my partner and I are "on the same page" in terms of the decisions we make about sexual health and risk | () | () | () | () |
| When it comes to sexual decision-making, I feel like my partner and I are "of the same mind" | () | () | () | () |
| Sometimes I feel like my priorities for my sexual health are incompatible with my partner's goals | () | () | () | () |
| I'm confident that my partner and I generally share the same priorities when it comes to sexual health | () | () | () | () |

| Making sexual health decisions with my partner can be difficult because we | () | () | () | () |
|---|---|---|---|---|
| different<br>priorities | | | | |

#### **Health Providers**

ID: 157

Now, we are going to ask you about your health care and health care decision making.

Logic: Show/hide trigger exists.

Shortname / Alias: pcp

ID: 158

Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?\*

() Yes

() No

Logic: Hidden unless: #22 Question "Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?" is one of the following answers ("Yes")

Shortname / Alias: pcpawareness

ID: 105

How open are you about your sexual identity to your primary medical care provider?\*

- ( ) Primary medical provider definitely does NOT know your sexual identity
- ( ) Primary medical provider MIGHT know about your sexual identity
- ( ) Primary medical provider PROBABLY knows about your sexual identity
- ( ) Primary medical provider DEFINITELY knows about your sexual identity

| Logic: Hidden unless: #22 Question "Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?" is one of the following answers ("Yes") |
|---|
| Shortname / Alias: pcptalksex |
| ID: 160 |
| How comfortable are you discussing your sexual behavior with your primary health care provider?* ( ) Very comfortable ( ) Somewhat comfortable ( ) Somewhat uncomfortable ( ) Very uncomfortable |
| STI Testing |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: stitest3m |
| ID: 170 |
| A sexually transmitted infection (STI) is an infection transmitted through sexual activity, such as syphilis, gonorrhea, chlamydia, herpes, or genital warts. In the past 3 months, have you been tested for an STI that was not HIV?* () Yes () No |
| Logic: Hidden unless: #25 Question "A sexually transmitted infection (STI) is an infection transmitted through sexual activity, such as syphilis, gonorrhea, chlamydia, herpes, or genital warts. In the past 3 months, have you been tested for an STI that was not HIV?" is one of the following answers ("Yes") |
| Shortname / Alias: sti3mo |
| ID: 171 |
| Please indicate whether you have been diagnosed with any of the following sexually transmitted infections in the past 3 months. Please select all that apply.* [] Chlamydia |
| [] Genital warts, anal warts, HPV |
| [] Gonorrhea |
| [] Hepatitis B |
| [] Hepatitis C |
| [] Herpes, HSV1/HSV2 |

| [] Syphilis |
|---|
| [ ] Urethritis |
| [] Other, please specify:: |
| [] None of these |
| HIV Testing |
| Shortname / Alias: recenthistest mon |
| Shortname / Alias: recenthivtest_mon ID: 165 |
| When did you have your most recent HIV test? |
| Please enter the month and year. |
| Month:* |
| ( ) January |
| () February |
| () March |
| ( ) April |
| () May |
| () June |
| ( ) July |
| ( ) August |
| () September |
| ( ) October |
| () November |
| ( ) December |
| Validation: Min = 1980 Must be numeric Whole numbers only Positive numbers only Max character count = 4 |
| Shortname / Alias: recenthivtest_yr |
| ID: 166 |
| Year:* |
| <del></del> |

Action: JavaScript: Hide General Error Message

| Page entry logic: This page will show when: (#27 Question "When did you have your most recent HIV test? |
|---|
| Please enter the month and year. |
| Month:" AND #28 Question "Year:" ) |
| Action: Custom Script: Check HIV test date not in future |
| PrEP Use |
| Shortname / Alias: prepstartafterP3-T |
| ID: 1201 |
| Did you start taking PrEP after you started the P3-T study?* ( ) Yes |
| ( ) No |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: nowprep |
| ID: 1202 |
| Are you taking PrEP right now?* () Yes |
| ( ) No |
| Logic: Hidden unless: Fix logic- If no to Did you start taking PrEP after you enrolled in P3-T |
| Shortname / Alias: noprep_why |
| ID: 1203 |
| Why did you decide not to start PrEP? Select all of the factors below that were related to why you didn't take PrEP.* [] I couldn't afford it |
| [] I was not having sex |
| [] I was no longer having sex with a person living with HIV |
| [] I was only having sex with one person and they were undetectable or HIV negative |
| [ ] I didn't want to take a pill every day |
| • |

| [] I kept forgetting to take my pill |
|---|
| [] I could no longer see my PrEP provider and haven't found another PrEP provider |
| [] I was worried about experiencing side effects |
| [] I was worried about the long term effects of PrEP on my health |
| [] It was medically unsafe for me to take PrEP (due to kidney/renal function, bone density, or another medical issue) |
| [] I was worried that if I were to become HIV-positive certain medications may no longer work or I might be resistant to them |
| [] I was worried that PrEP might not provide complete protection against HIV |
| [] I started using condoms all of the time |
| [] I was worried that the medication would taste bad and/or the pill would be too big |
| [ ] Other, please specify:: |

**Page entry logic:** This page will show when: #32 Question "Why did you decide not to take PrEP? Select all of the factors below that were related to why you didn't take PrEP."

### PrEP Use, why didn't start

Action: Custom Script: Script to count checkboxes and skip if q <2

ID: 1204

Piping: Piped Values From Question 32. (Why did you decide not to take PrEP? Select all of the factors below that were related to why you didn't take PrEP.)

Please rank the reasons you did not start taking PrEP in order of importance.\*

Page entry logic: Fix logic- If yes to Did you start taking PrEP after you enrolled in P3-T

#### **PrEP Start**

Shortname / Alias: startprep\_why

ID: 943

### Why did you choose to start taking PrEP? Select all that apply.\*

- [] I'm having sex with or thinking about having sex with someone who is HIV+
- [] I'm having sex with or thinking about having sex with someone whose HIV status I don't know
- [] I want to be in control of my sexual health

| [ ] I want to reduce my anxiety around sex |
|-----------------------------------------------------------|
| [] I want to increase my sexual satisfaction and intimacy |
| [] I want to be safe and healthy |
| [] I want to have a better future |
| [] I am having sex with multiple partners |
| [] I don't like to use condoms |
| [] My partner won't use condoms |
| [] I had a previous HIV scare |
| [] My health care provider recommended it |
| [] I was recently diagnosed with an STI |
| [] Many people in my community take PrEP |
| [] Other, please specify:: |
| [ ] Decline to answer |

#### **PrEP Start**

Action: Custom Script: Script to count checkboxes and skip q if < 2

Shortname / Alias: startprep primwhy

ID: 945

Piping: Piped Values From Question 34. (Why did you choose to start taking PrEP? Select all that apply.)

What was the main reason you started PrEP?\*

**Page entry logic:** This page will show when: (#30 Question "Did you start taking PrEP after you started the P3-T-T study?" is one of the following answers ("Yes") OR #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes"))

### **PrEP Start and Stop**

Validation: %s format expected

Logic: Hidden unless: #30 Question "Did you start taking PrEP after you started the P3-T-T

study?" is one of the following answers ("Yes")

Shortname / Alias: prep\_firststart

#### ID: 947

When did you start taking after enrolling in P3-T?

If you do not know the exact day of the month, please give your best estimate. \*

\_\_\_\_\_\_

Logic: Hidden unless: #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes")

Shortname / Alias: prepstoP3-T-Tmo

ID: 576

Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?\*

() Yes

() No

Action: Custom Script: Check date not in future

Action: Custom Script: Script to populate - 3 months date

Hidden Value: Date for prompt - today minus 3 months

Value:

**Page entry logic:** This page will show when: #37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes")

## PrEP Stop, last 3 months

Logic: Show/hide trigger exists.

Shortname / Alias: timesprepstoP3-Tmo

ID: 950

How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?\*

- ()0
- ()1
- ()2
- ()3
- ()4

| ()6 |
|---|
| ()7 |
| ()8 |
| ()9 |
| ()10 |
| ()11 |
| ( ) 12 or more |
| Logic: Hidden by default |
| ID: 1159 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("1") |
| Shortname / Alias: time1_dates |
| ID: 1027 |
| Please enter the dates you were off PrEP (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1028 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1029 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1160 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the |

()5

Shortname / Alias: timefirst\_dates
| ID: 1030 |
|---|
| Please enter the dates you were <u>off</u> PrEP for the <u>first</u> time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1031 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1032 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1161 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("2","3","4","5","6","7","8","9","10","11","12 or more") |
| Shortname / Alias: timesecond_dates |
| ID: 1033 |
| Please enter the dates you were off PrEP for the second time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1034 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1035 |

Logic: Hidden by default

Date re-started:\*:

ID: 1162

The date re-started is before the date stopped. Please correct this.

| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("3","4","5","6","7","8","9","10","11","12 or more") |
|---|
| Shortname / Alias: timethird dates |
| ID: 1036 |
| Please enter the dates you were <u>off</u> PrEP for the <u>third</u> time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1037 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1038 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1163 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") |
| Shortname / Alias: timefourth_dates |
| ID: 1039 |
| Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): |
| Please enter the dates you were off PrEP for the fourth time (from [question('value'), |
| Please enter the dates you were <u>off</u> PrEP for the <u>fourth</u> time (from [question('value'), id='1026'] to today): |
| Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected |
| Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 |
| Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 Date stopped:*: |
| Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 Date stopped:*: Validation: %s format expected |
| Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 Date stopped:*: Validation: %s format expected ID: 1041 |
| Please enter the dates you were off PrEP for the fourth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1040 Date stopped:*: Validation: %s format expected ID: 1041 |

| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") |
|---|
| Shortname / Alias: timefifth_dates |
| ID: 1042 |
| Please enter the dates you were off PrEP for the fifth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1043 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1044 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1165 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("6","7","8","9","10","11","12 or more") |
| Shortname / Alias: timesixth_dates |
| ID: 1045 |
| Please enter the dates you were off PrEP the sixth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1046 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1047 |
| Date re-started:*: |

| ID: 1166 |
|---|
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("7","8","9","10","11","12 or more") |
| Shortname / Alias: timeseventh_dates |
| ID: 1048 |
| Please enter the dates you were off PrEP for the seventh time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1049 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1050 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1167 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("8","9","10","11","12 or more") |
| Shortname / Alias: timeeighth_dates |
| ID: 1051 |
| Please enter the dates you were off PrEP for the eighth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1052 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1053 |

Logic: Hidden by default

| Logic: Hidden by default |
|---|
| ID: 1168 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("9","10","11","12 or more") |
| Shortname / Alias: timeninth_dates |
| ID: 1054 |
| Please enter the dates you were off PrEP for the ninth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1055 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1056 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1169 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a |

row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("10","11","12 or more")

Shortname / Alias: timetenth\_dates

Date re-started:\*:

ID: 1057

Please enter the dates you were off PrEP for the tenth time (from [question('value'), id='1026'] to today):\*

Validation: %s format expected

| Validation: %s format expected |
|---|
| ID: 1059 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1170 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("11","12 or more") |
| Shortname / Alias: timeeleventh_dates |
| ID: 1060 |
| Please enter the dates you were off PrEP for the eleventh time (from [question('value'), id='1026'] to today):* |
| id='1026'] to today):* |
| id='1026'] to today):* Validation: %s format expected |
| id='1026'] to today):* Validation: %s format expected ID: 1061 |
| <pre>id='1026'] to today):* Validation: %s format expected ID: 1061 Date stopped:*:</pre> |
| Validation: %s format expected ID: 1061 Date stopped:*: Validation: %s format expected ID: 1062 Date re-started:*: |
| id='1026'] to today):* Validation: %s format expected ID: 1061 Date stopped:*: Validation: %s format expected ID: 1062 Date re-started:*: Logic: Hidden by default ID: 1171 |
| id='1026'] to today):* Validation: %s format expected ID: 1061 Date stopped:*: |

Date stopped:\*:

Logic: Hidden unless: #38 Question "How many times did you <u>stop taking PrEP for 7 days in a row or more</u> in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("12 or more")

Shortname / Alias: timetwelfth\_dates

Please enter the dates you were <u>off</u> PrEP for the <u>twelfth</u> time (from [question('value'), id='1026'] to today):\*

| Validation: %s format expected |
|--------------------------------|
| ID: 1064 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1065 |
| Date re-started:*: |

**Page entry logic:** This page will show when: ((#37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes") OR (#29 Question "When you started the P3-T study, were you taking PrEP?" is one of the following answers ("Yes") AND #31 Question "Are you taking PrEP right now?" is one of the following answers ("No"))) OR (#30 Question "Did you start taking PrEP after you started the P3-T study?" is one of the following answers ("Yes") AND #31 Question "Are you taking PrEP right now?" is one of the following answers ("No")))

## **PrEP Stop**

Logic: Hidden by default

ID: 1206

This number cannot be greater than the number of times you stopped taking PrEP for 7 days in a row or more in the last 3 months ([question('value'), id='950']). Please correct this.

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("1","2","3","4","5","6","7","8","9","10","11","12 or more")

Shortname / Alias: prepstop\_drconsult

ID: 578

Of the [question("value"), id="950"] times you stopped taking PrEP, how many did you talk with your medical provider about before you stopped taking PrEP?\*

Shortname / Alias: stopprep why

ID: 581

Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP.\*

[] I couldn't afford it anymore

| [] I was not having sex |
|---|
| [] I was no longer having sex with a person living with HIV |
| [] I was only having sex with one person and they were undetectable or HIV negative |
| [] I didn't want to keep taking a pill every day |
| [] My parent(s) or guardian(s) found out and made me stop |
| [] I kept forgetting to take my pill |
| [] I haven't been able to make it to my follow-up appointments |
| [] I could no longer see my PrEP provider and haven't found another PrEP provider |
| [] I experienced side effects |
| [] I was worried about the long term effects of PrEP on my health |
| [] It was medically unsafe for me to continue taking PrEP (due to kidney/renal function, bone density, or another medical issue) |
| [] I was worried that if I were to become HIV-positive certain medications may no longer work or I might be resistant to them |
| [] I was worried that PrEP might not provide complete protection against HIV |
| [] I started using condoms all of the time |
| [] The medication tastes bad and/or the pill is too big |
| [] Other, please specify:: |

**Page entry logic:** This page will show when: #38 Question "How many times did you <u>stop taking PrEP for 7 days in a row or more</u> in the last three months (*from [question('value'), id='1026'] to today)*?" is one of the following answers ("1","2","3","4","5","6","7","8","9","10","11")

Action: Custom Script: Script to check number of times off PrEP

**Page entry logic:** This page will show when: #53 Question "Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP."

# **PrEP Stop Continued**

Action: Custom Script: Script to count checkboxes and skip if q < 2

Shortname / Alias: stopprep primwhy

ID: 582

Piping: Piped Values From Question 53. (Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP.)

Please rank the reasons you stopped taking PrEP in order of importance.\*

**Page entry logic:** This page will show when: #37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes")

# PrEP Restart, current users

Shortname / Alias: restart\_why

| ID: 956 |
|---|
| Why did you choose to restart taking PrEP the last time? Select all that apply.* [] I was able to start seeing my PrEP provider again |
| [] I found a new PrEP provider |
| [] I was having issues with side effects, but I found a way to deal with them |
| [] I was having issues taking my pill every day, but I found a way to deal with it |
| [] I'm having sex with or thinking about having sex with someone who is HIV+ |
| [] I'm having sex with or thinking having sex with someone whose status HIV I don't know |
| [] I want to be in control of my sexual health |
| [] I want to reduce my anxiety around sex |
| [] I want to increase my sexual satisfaction and intimacy |
| [] I want to be safe and healthy |
| [] I want to have a better future |
| [] I am having sex with multiple partners |
| [] I don't like to use condoms |
| [] My partner won't use condoms |
| [] I had a previous HIV scare |
| [] My health care provider recommended it |
| [] I was recently diagnosed with an STI |
| [] Many people in my community take PrEP |
| [] Other, please specify:: |

Action: JavaScript: Hide General Error Message

**Page entry logic:** This page will show when: #55 Question "Why did you choose to restart taking PrEP the last time? Select all that apply."

Action: Custom Script: Script to count checkboxes and skip if q <2

Shortname / Alias: restart\_primwhy

ID: 957

Piping: Piped Values From Question 55. (Why did you choose to restart taking PrEP the last time?

Select all that apply.)

What was the main reason you decided to restart PrEP?\*

#### **Healthcare Visits**

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Show/hide trigger exists.

Shortname / Alias: numdrvisits3m

ID: 584

In the last 3 months, how many times did you go to the doctor for any reason?\*

\_\_\_\_\_

Logic: Hidden by default

ID: 940

This number cannot be greater than the total number of doctor's visits entered above.

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Show/hide trigger exists. Hidden unless: #57 Question "In the last 3 months, how many times did you go to the doctor for any reason?" is greater than "0"

Shortname / Alias: numprepvisits3m

ID: 586

Out of all these visits, how many were routine/scheduled PrEP appointments?\*

Logic: Hidden by default

## This number cannot be greater than the total number of routine PrEP appointments.

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Hidden unless: #58 Question "Out of all these visits, how many were routine/scheduled PrEP appointments?" is greater than "0"

Shortname / Alias: missedprepvisits3m

ID: 587

In the last 3 months, how many of your scheduled PrEP appointments did you miss because you didn't show or forgot?

By scheduled appointments, we mean routine PrEP appointments, not walk-in or urgent care appointments for acute/urgent issues. \*

Action: Custom Script: Script to check number of visits

Action: Custom Script: Script to check number of days

#### **PrEP Adherence**

Logic: Hidden unless: #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes")

Shortname / Alias: preplastweek

ID: 177

How many of the last 7 days did you take your PrEP medication?\*

- () 0 days
- () 1 day
- () 2 days
- () 3 days
- () 4 days
- () 5 days
- () 6 days
- () 7 days

Validation: Min = 0 Max = 100

| Shortname / Alias: prepmonth |
|---|
| ID: 178 |
| In the last month, what percent of the time did you take your PrEP as prescribed (once a day)? Use the scale below. 0% would mean 'NONE' of the time and 100% would mean 'ALL' of the time. If you are unsure, make a guess. |
| % medication taken:* 0 100 |
| PrEP Dose Barriers |
| Shortname / Alias: dose_ |
| ID: 959 |
| What has gotten in the way of you taking your PrEP on a daily basis? Please select all that apply.* [] I have not had any trouble taking PrEP on a daily basis [] I get tired of taking a pill every day [] I forget to take it [] I don't always have my pills with me [] My work/school schedule [] My social life [] I'm around people I don't want to take it in front of [] I experience side effects [] I was drinking or using drugs and I didn't take it |
| Hidden Page of Script Action: Custom Script: Script to count checkboxes and skip if q <2 |

Logic: Show/hide trigger exists.

Shortname / Alias: does\_rank

Piping: Piped Values From Question 62. (What has gotten in the way of you taking your PrEP on a daily basis? Please select all that apply.)

Please rank the things that have gotten in the way of you taking your PrEP on a daily basis.\*

#### **PrEP Adherence Continued**

Logic: Hidden unless: #61 Question "In the last month, what percent of the time did you take your PrEP as prescribed (once a day)? Use the scale below.

0% would mean 'NONE' of the time and 100% would mean 'ALL' of the time. If you are unsure, make a guess.

% medication taken:"

Shortname / Alias: prepadher protection

ID: 588

You said you took your PrEP [question("value"), id="178"] percent of the time in the last month. Based on this adherence level, how protected do you think you were from HIV in the last month?\*

- () Not protected at all
- () Somewhat protected
- () Mostly protected
- () Fully protected

Shortname / Alias: prepadher\_decisionbot

ID: 589

In the last month, how much did your adherence to PrEP (if you took it every day or not) affect how often you used a condom during anal sex when you bottom?\*

- ( ) My decision about condom use when I bottom <u>was not</u> influenced by whether or not I took my pill every day
- ( ) My decision about condom use when I bottom <u>was somewhat</u> influenced by whether or not I took my pill every day
- ( ) My decision about condom use when I bottom <u>was</u> influenced by whether or not I took my pill every day
- () I did not bottom in the last month

Shortname / Alias: prepadher decisiontop

ID: 590

In the last month, how much did your adherence to PrEP (if you took it every day or not) affect how often you used a condom during anal sex when you top?\*

- ( ) My decision about condom use when I top <u>was not</u> influenced by whether or not I took my pill every day
- ( ) My decision about condom use when I top <u>was somewhat</u> influenced by whether or not I took my pill every day
- ( ) My decision about condom use when I top was influenced by whether or not I took my pill every day
- () Decline to answer

# **PrEP Confidence**

Take PrEP on a weekday:\*

| Т | D | ٠. | 9 | U | 7 |
|---|---|----|---|---|---|
| | ட | 4 | ~ | w | • |

We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident).

| Validation: Min = 1 Max = 10 | |
|---------------------------------------|------|
| Shortname / Alias: keepappts | |
| ID: 903 | |
| How confident are you that you can | |
| Keep your PrEP medical appointments:* | |
| 1 | _ 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: followplan | |
| ID: 904 | |
| Follow a plan for taking PrEP:* | |
| 1 | _ 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: atworkschool | |
| ID: 905 | |
| Take PrEP at work/school:* | |
| 1 | _ 10 |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: onweekday | |
| ID: 906 | |

| Action: JavaScript: Hide General Error Message |
|---|
| PrEP Confidence 2 |
| ID: 908 |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). |
| Validation: Min = 1 Max = 10 |
| Shortname / Alias: onweekend |
| ID: 909 |
| How confident are you that you can |
| Take PrEP on a weekend:* 1 10 |
| Validation: Min = 1 Max = 10 |
| Shortname / Alias: wfriends |
| ID: 910 |
| Take PrEP when I'm out with friends:* 1 10 |
| Validation: Min = 1 Max = 10 |
| Shortname / Alias: prepdrinking |
| ID: 911 |
| Take PrEP when I'm drinking or using drugs:* 1 10 |
| · 'V |
| Validation: Min = 1 Max = 10 |

Shortname / Alias: schedulechange

| ID: 912 |
|---|
| Take PrEP when my schedule changes:* 1 10 |
| Action: JavaScript: Hide General Error Message |
| PrEP Confidence 3 |
| ID: 913 |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). |
| Validation: Min = 1 Max = 10 |
| Shortname / Alias: whiletraveling |
| ID: 914 |
| How confident are you that you can |
| Take PrEP while traveling:* 1 10 |
| Validation: Min = 1 Max = 10 |
| Shortname / Alias: takewsideeffects |
| ID: 915 |
| Take PrEP when you are having medication side effects:* 1 10 |
| Validation: Min = 1 Max = 10 |
| Shortname / Alias: havingcrisis |
| ID: 916 |
| Take PrEP when you are having a crisis:* 1 10 |

## **PrEP Delivery**

Shortname / Alias: prep prefmode

ID: 597

Right now there are no other approved options for taking PrEP. However, if there were more than one option and each method was equally good at protecting you from getting HIV, which method would you most prefer?\*

- () Taking one pill, every day
- ( ) Taking two pills before you had sex and a pill a day for the next two days
- ( ) Taking one pill a day just on Tuesday, Thursday, Saturday, and Sunday
- () Getting an injection about every 2 to 3 months
- ( ) Putting medicated lubrication (lube) in your anus (and/or your partner's anus) before having anal sex
- ( ) Douching with a medicated solution (microbicide) before having anal sex

## **PrEP Beliefs**

Shortname / Alias: prepbeliefs

ID: 598

Please rate your agreement with the following statements:\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| People are<br>less likely<br>to use<br>condoms<br>for anal sex<br>if they are<br>using PrEP | () | () | () | () |
| I feel as if<br>starting to<br>take PrEP<br>would allow<br>me to have<br>more sex<br>partners | () | () | () | () |

| I feel as if starting to take PrEP would allow me to have more condomless anal sex | () | () | () |
|---|---|---|---|
|---|---|---|---|

# **PrEP and People**

Shortname / Alias: prepppl

ID: 193

We are interested in how you feel about the following statements. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I worry people will assume I sleep around if they know I take PrEP | () | () | () | () |
| I worry people will assume that I am HIV- positive if they know I take PrEP | () | () | () | () |
| I worry people will think my partner(s) are HIV- positive if they know I take PrEP | () | () | () | () |
| I worry about<br>listing PrEP<br>as one of my | () | () | () | () |

| current medications during appointments such as at a dentist's or specialist's office | | | | |
|---|---|---|---|---|
| I feel<br>ashamed to<br>tell other<br>people that I<br>am taking<br>PrEP | () | () | () | () |
| I worry people will think I am a bad person if they know I take PrEP | () | () | () | () |
| I worry people will think I am gay if they know I take PrEP | () | () | () | () |
| I worry my<br>friends will<br>find out that I<br>take PrEP | () | () | () | () |
| I worry my<br>family will<br>find out that I<br>take PrEP | () | () | () | () |
| I worry my<br>sexual<br>partners will<br>find out that I<br>take PrEP | () | () | () | () |
| I think people<br>will give me a<br>hard time if I<br>tell them I<br>take PrEP | () | () | () | () |

| I think people<br>will judge me<br>if they know I | () | () | () | () |
|---------------------------------------------------|----|----|----|----|
| am taking<br>PrEP | | | | |

# **PrEP Concerns**

Shortname / Alias: prepconc

ID: 210

We are interested in how you feel about the following statements. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| My family<br>does not<br>support me<br>taking PrEP | () | () | () | () |
| My friends<br>do not<br>support me<br>taking PrEP | () | () | () | () |
| People<br>taking PrEP<br>are<br>portrayed<br>poorly in the<br>media and<br>online | () | () | () | () |
| People in my<br>community<br>talk poorly<br>about people<br>taking PrEP | () | () | () | () |
| I feel<br>embarrassed<br>about taking<br>PrEP | () | () | () | () |

| I think I am<br>not following<br>the 'rules' of<br>my<br>community if<br>I take PrEP | () | () | () | () |
|---|---|---|---|---|
| I have been<br>blamed by<br>people in my<br>community<br>for spreading<br>HIV through<br>PrEP use | () | () | () | () |
| I have been blamed by people in my community for spreading sexually transmitted infections through not using condoms | () | () | () | () |
| I have been rejected romantically because I take PrEP | () | () | () | () |
| I have been slut-shamed because I take PrEP (or told that I am a "Truvada-slut/whore") | () | () | () | () |
| I have been judged by a health care provider for taking PrEP | () | () | () | () |
| I don't think<br>that I need to<br>take PrEP<br>anymore | () | () | () | () |

| I have been told by a health care provider that I don't need PrEP or I shouldn't take PrEP | () | () | () | () |
|---|---|---|---|---|
| I have been<br>yelled at or<br>scolded<br>because I<br>take PrEP | () | () | () | () |
| I have been unfairly discriminated against because I take PrEP | () | () | () | () |
| I have experienced physical violence because I am taking PrEP | () | () | () | () |

Logic: Hidden unless: Question "I don't think that I need to take PrEP anymore" is one of the following answers ("Agree", "Strongly Agree")

Shortname / Alias: whydontneed

| Why do you think that you do not need to take PrEP anymore? Select all that apply.* [] My relationship status changed I became single |
|---|
| [] My relationship status changed I became monogamous (only having sex with one person) |
| [] I stopped having sex with an HIV-positive person |
| [] I am having less sex |
| [] I am sexually inactive (I haven't been having sex for a period of time) |
| [] I have started using condoms every time I have sex |
| [1 Other please specify: |

Shortname / Alias: prepdifficulties

ID: 602

In making your decision to continue taking PrEP, please rate how much the following items

concern you.\*

| | Not at all concerned | A little concerned | Concerned | Very<br>concerned |
|---|---|---|---|---|
| Getting the costs of PrEP covered (including office visits or office visit copays, lab costs, transportation costs) | () | () | () | () |
| Using insurance to get coverage for PrEP costs (including office visits, lab costs) | () | () | () | () |
| Getting<br>transportation<br>to PrEP<br>appointments<br>and labs | () | () | () | () |
| Returning for<br>PrEP follow-<br>up<br>appointments<br>and labs | () | () | () | () |
| Getting PrEP prescription refilled | () | () | () | () |

Shortname / Alias: prepdifficulties2

ID: 649

In making your decision to continue taking PrEP, please rate how much the following items concern you.\*

| | Not at all concerned | A little concerned | Concerned | Very<br>concerned |
|---|---|---|---|---|
| The possibility that if I were to become HIV+, certain medications might no longer work or I might be resistant to them | () | () | () | () |
| The possibility that PrEP might not provide complete protection against HIV | () | () | () | () |
| Having to talk to a health care provider about PrEP | () | () | () | () |
| Having to talk to a health care provider about my sex life | () | () | () | () |
| Experiencing side effects from PrEP | () | () | () | () |
| The long-<br>term effects<br>of PrEP on<br>my health | () | () | () | () |

| Having to remember to take PrEP every day | () | () | () | () |
|---|---|---|---|---|
| Friends<br>finding out<br>that I am on<br>PrEP | () | () | () | () |
| Family<br>members<br>finding out<br>that I am on<br>PrEP | () | () | () | () |
| Sexual<br>partners<br>finding out<br>that I am on<br>PrEP | () | () | () | () |

| Logic: Hidden unless: Question " | The possibility that PrEF | might not provide o | complete protection |
|---|---|---|---|
| against HIV" is one of the followi | ng answers ("Concerned | l","Very concerned" | |

Shortname / Alias: prepworry

ID: 665

# Why do you worry about the possibility that PrEP might not provide complete protection against HIV? (Check all that apply)\*

| г п | l 4 la | -44 | ــا بــا بــا اـــ | | - cc1: | _4 | _ 1: | 1 111 / |
|---|---|---|---|---|---|---|---|---|
| | i worry in | at the | arua is | not | effective | at breve | ntina | HIV |

| г | 1 December 1 | 1 4 - 6 4 - 6 - 6 | DrED avant | 40,400 | برالمرملمنمص |
|---|--------------|-------------------|------------|--------|--------------|
| | i because | i don i take | PrEP everv | gav co | ınsıstentiv |

| | _ | | | | 1 1 1 | | | | | 14.1 | 1 111 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ı | Because | I teel | i am at | Verv | hidh | rick | tor r | necomina | intected | with | HIV |
| | | 1 1001 | ı amı at | VOIV | HIGH | 1131 | 101 L | | 111100104 | VVILII | |

| I I ( )thar blace chacity |
|-----------------------------|
| [ ] Other, please specify:: |

Action: JavaScript: Hide General Error Message

# **HIV** perceptions

Shortname / Alias: hivthoughts

Imagine how you would feel if you became infected with HIV. Read each statement carefully and

indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I would<br>be afraid<br>people<br>would<br>judge me<br>when<br>they<br>learn I<br>have HIV | () | () | () | () |
| If I got infected, people would not want to have sex with me | () | () | () | () |
| I would<br>feel<br>guilty if I<br>got HIV | () | () | () | () |
| I would<br>feel<br>ashamed<br>if I got<br>HIV | () | () | () | () |

## PEP and PrEP On-Demand

Shortname / Alias: peP3-Tm

ID: 230

In the past 3 months, have you taken post-exposure prophylaxis (PEP) <u>AFTER</u> a sexual or drug use exposure to reduce the risk of getting HIV?\*

- () Yes
- () No
- () Decline to answer

Shortname / Alias: prepondemand3m ID: 674

In the past 3 months, have you taken PrEP on-demand (taking two pills before you had sex and a pill a day for the next two days)?

It is not an approved method and has not been shown to be an effective method for preventing HIV.\*

() Yes

() No

() Decline to answer

#### **Substances**

ID: 232

Now we'd like to ask you a little bit about your experiences using alcohol, tobacco products, and other drugs. Please be assured that this information will be treated as *strictly confidential*.

The questions will concern your experiences with using these substances in the past three months. These substances can be smoked, swallowed, snorted, inhaled, injected, or taken in the form of pills. Some of the substances may be prescribed by a doctor (like amphetamines, sedatives, or pain medications). For this survey, do not report on medications that are used as prescribed by your doctor. However, if you have taken such medications for reasons other than prescription, or taken them more frequently or at higher doses than prescribed, please report on this use. Once again, please remember that all information provided will be treated as *strictly confidential*.

Shortname / Alias: substanceuse3m

ID: 233

Which of the following drugs have you used in the last 3 months? *Please check all that apply.*\*

[ ] Tobacco (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)

[] Alcohol (beer, wine, spirits, etc.)

[ ] Cannabis (marijuana, pot, weed, grass, hash, synthetic cannabis, etc.)

[] Cocaine (coke, crack, etc.)

[] Amphetamines (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)

[] Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)

[] Sedatives, tranquilizers, or sleeping pills (valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)

| [] Hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.) |
|---|
| [] Opioids (heroin, morphine, methadone, codeine, Oxycotin, Percocet, Vicodin, etc.) |
| [] None of these |
| Action: JavaScript: Hide General Error Message |
| Page entry legic. This negativill above when #00 Outsetien "Which of the following drugs have you used |
| <b>Page entry logic:</b> This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? |
| Please check all that apply." is one of the following answers ("Tobacco (cigarettes, chewing tobacco, |
| cigars, e-cigarettes, etc.)") |
| Tobacco |
| Tobacco |
| Shortname / Alias: tobacco3months |
| ID: 234 |
| In the past 3 months, how often have you used tobacco products (cigarettes, chewing tobacco, |
| cigars, e-cigarettes, etc.)?* |
| () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccodesire |
| ID: 235 |
| During the past 3 months, how often have you had a desire to use tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* |
| () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccoproblems |
| ID: 236 |

| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* ( ) Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccofailed |
| ID: 237 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| ( ) Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccofriend |
| ID: 238 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* ( ) No ( ) Yes |
| Shortname / Alias: tobaccostop |
| ID: 239 |
| In the last 3 months, have you tried and failed to control, cut down or stop using tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () No |
| () Yes |

**Page entry logic:** This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

Please check all that apply." is one of the following answers ("Alcohol (beer, wine, spirits, etc.)")

# **Alcohol**

| Logic: Show/hide trigger exists. |
|---|
| Shortname / Alias: alcohol3months |
| ID: 240 |
| In the past 3 months, how often have you used alcoholic beverages (beer, wine, spirits, etc.)?* |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Logic: Hidden unless: #97 Question "In the past 3 months, how often have you used alcoholic beverages (beer, wine, spirits, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily","Decline to answer") |
| Shortname / Alias: alcoholdaily |
| ID: 241 |
| How many drinks containing alcohol do you have on a typical day?* |
| ()0 |
| () 1 or 2 |
| ( ) 1 or 2 |
| ( ) 1 or 2<br>( ) 3 or 4 |
| ( ) 1 or 2<br>( ) 3 or 4<br>( ) 5 or 6 |
| () 1 or 2<br>() 3 or 4<br>() 5 or 6<br>() 7 to 9 |
| () 1 or 2<br>() 3 or 4<br>() 5 or 6<br>() 7 to 9 |
| () 1 or 2<br>() 3 or 4<br>() 5 or 6<br>() 7 to 9 |
| () 1 or 2<br>() 3 or 4<br>() 5 or 6<br>() 7 to 9 |
| () 1 or 2<br>() 3 or 4<br>() 5 or 6<br>() 7 to 9<br>() 10 or more |
| () 1 or 2 () 3 or 4 () 5 or 6 () 7 to 9 () 10 or more Shortname / Alias: alcoholbinge |
| () 1 or 2 () 3 or 4 () 5 or 6 () 7 to 9 () 10 or more Shortname / Alias: alcoholbinge ID: 242 How often do you have 5 or more drinks on one occasion?* |
| () 1 or 2 () 3 or 4 () 5 or 6 () 7 to 9 () 10 or more Shortname / Alias: alcoholbinge ID: 242 How often do you have 5 or more drinks on one occasion?* () Never |
| () 1 or 2 () 3 or 4 () 5 or 6 () 7 to 9 () 10 or more Shortname / Alias: alcoholbinge ID: 242 How often do you have 5 or more drinks on one occasion?* () Never () Less than monthly |

| Shortname / Alias: alcoholdesire |
|---|
| ID: 243 |
| During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholproblems |
| ID: 244 |
| During the past 3 months, how often has your use of alcoholic beverages (beer, wine, spirits, etc.) led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholfailed |
| ID: 245 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholfriend |
| SHORMATILE / Alias, alconomieno |

| ()Yes |
|---|
| Shortname / Alias: alcoholstop |
| ID: 247 |
| In the last 3 months, have you tried and failed to control, cut down or stop using alcoholic beverages (beer, wine, spirits, etc.)?* () No |
| () Yes |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used |
| in the last 3 months? Please check all that apply." is one of the following answers ("Cannabis (marijuana, pot, weed, grass, hash, synthetic cannabis, etc.)") |
| Cannabis |
| Shortname / Alias: cannabis3months |
| ID: 251 |
| In the past 3 months, how often have you used cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Page entry logic: This page will show when: #107 Question "In the past 3 months, how often have you used cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?" is one of the following answers ("Once or twice", "Monthly", "Weekly", "Daily or almost daily") |
| Cannabis (cont.) |

In the last 3 months, has a friend or relative or anyone else expressed concern about your use of alcoholic beverages (beer, wine, spirits, etc.)?\*

() No

Shortname / Alias: cannabisdesire

| ID: 252 |
|---|
| During the past 3 months, how often have you had a desire to use cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisproblems |
| ID: 253 |
| During the past 3 months, how often has your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisfailed |
| ID: 254 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisfriend |

ID: 255

In the past 3 months, has a friend or relative or anyone else expressed concern about your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?\*

() No

() Yes

Shortname / Alias: cannabisstop

| - | $\overline{}$ | <br>$\Omega \Gamma C$ |
|---|---------------|-----------------------|
| ı | | 256 |

| In the last 3 months, have you tried and failed to control, cut down or stop using cannabis |
|---|
| (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* |
| ( ) No |

() Yes

**Page entry logic:** This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

Please check all that apply." is one of the following answers ("Cocaine (coke, crack, etc.)")

## Cocaine

Shortname / Alias: cocaine3months

ID: 257

In the past 3 months, how often have you used cocaine (coke, crack, etc.)?\*

- () Never
- () Once or twice
- () Monthly
- () Weekly
- () Daily or almost daily

**Page entry logic:** This page will show when: #113 Question "In the past 3 months, how often have you used cocaine (coke, crack, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily")

# Cocaine (cont.)

Shortname / Alias: cocainedesire

ID: 258

During the past 3 months, how often have you had a desire to use cocaine (coke, crack, etc.)?\*

- () Never
- () Once or twice
- () Monthly
- () Weekly
- () Daily or almost daily

| Shorthame / Alias. Cocalheproblems |
|---|
| ID: 259 |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cocainefailed |
| ID: 260 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of cocaine (coke, crack, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cocainefriend |
| ID: 261 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of cocaine (coke, crack, etc.)?* ( ) No |
| () Yes |
| Shortname / Alias: cocainestop |
| ID: 262 |
| In the last 3 months, have you tried and failed to control, cut down or stop using cocaine (coke, crack, etc.)?* ( ) No |
| () Yes |

**Page entry logic:** This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

*Please check all that apply.*" is one of the following answers ("Amphetamines (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)")

# **Amphetamine**

Shortname / Alias: amphetamineproblems

| Shortname / Alias: amphetamine3months |
|---|
| ID: 263 |
| In the past 3 months, how often have you used amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Page entry logic: This page will show when: #119 Question "In the past 3 months, how often have you used amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?" is one of th following answers ("Once or twice", "Monthly", "Weekly", "Daily or almost daily") |
| Amphetamine (cont.) |
| Shortname / Alias: amphetaminedesire |
| ID: 265 |
| During the past 3 months, how often have you had a desire to use amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| During the past 3 months, how often has your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.) led to health, social, legal or financial problems?* () Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetaminefailed |
| ID: 267 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetaminefriend |
| ID: 268 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) No |
| ()Yes |
| Shortname / Alias: amphetaminestop |
| ID: 269 |
| In the last 3 months, have you tried and failed to control, cut down or stop using amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) No |
| () Yes |

Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

*Please check all that apply.*" is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)")

#### **Inhalants**

() Never

() Monthly

() Once or twice

| Shortname / Alias: inhalants3months |
|---|
| ID: 271 |
| In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| <b>Page entry logic:</b> This page will show when: #125 Question "In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?" is one of the following answers ("One or twice","Monthly","Weekly","Daily or almost daily") |
| Inhalants (cont.) |
| Shortname / Alias: inhalantsdesire |
| ID: 272 |
| During the past 3 months, how often have you had a desire to use inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsproblems |
| ID: 273 |
| During the past 3 months, how often has your use of inhalants (poppers, nitrous, glue, petrol, |

paint thinner, etc.) led to health, social, legal or financial problems?\*

| () Weekly |
|---|
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsfailed |
| ID: 274 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsfriend |
| ID: 275 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* () No |
| () Yes |
| Shortname / Alias: inhalantsstop |
| ID: 276 |
| In the last 3 months, have you tried and failed to control, cut down or stop using inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* |
| ( ) No |
| ()Yes |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used |
| in the last 3 months? |

**Sedatives** 

Shortname / Alias: sedatives3months

Shortname / Alias: sedativesfailed

| Xanax, Ambien, GHB, etc.)?* ( ) Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: sedativesfriend |
| ID: 282 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) No ( ) Yes |
| Shortnamo / Alias: codativocatan |
| Shortname / Alias: sedativesstop |
| ID: 283 |
| · |
| ID: 283 In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* |
| In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* |
| In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) No ( ) Yes Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used |
| In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) No ( ) Yes Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? |
| In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) No ( ) Yes Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used |
| In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* ( ) No ( ) Yes Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? Please check all that apply." is one of the following answers ("Hallucinogens (LSD, acid, mushrooms, |
| In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* () No () Yes Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? Please check all that apply." is one of the following answers ("Hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)") |

In the past 3 months, how often have you used hallucinogens (LSD, acid, mushrooms, PCP,

Ketamine, etc.)?\*

() Once or twice

() Never

During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol,

| ( ) Daily or almost daily |
|---|
| Personatura India, This make will show whom #127 Occasion "In the most 2 months, how often have you |
| <b>Page entry logic:</b> This page will show when: #137 Question "In the past 3 months, how often have you used hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?" is one of the following answers |
| ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Hollyginggong (gont) |
| Hallucinogens (cont.) |
| Shortname / Alias: hallucinogensdesire |
| ID: 286 |
| During the past 3 months, how often have you had a desire to use hallucinogens (LSD, acid, |
| mushrooms, PCP, Ketamine, etc.)?* |
| () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensproblems |
| ID: 287 |
| During the past 3 months, how often has your use of hallucinogens (LSD, acid, mushrooms, PCP, |
| Ketamine, etc.) led to health, social, legal or financial problems?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensfailed |
| ID: 288 |
| During the past 3 months, how often have you failed to do what was normally expected of you |
| because of your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* () Never |

( ) Monthly( ) Weekly

() Once or twice

| ( ) Monthly |
|---|
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensfriend |
| ID: 289 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) No |
| () Yes |
| Shortname / Alias: hallucinogensstop |
| ID: 290 |
| In the last 3 months, have you tried and failed to control, cut down or stop using hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) No |
| () Yes |
| <b>Page entry logic:</b> This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? |
| Please check all that apply." is one of the following answers ("Opioids (heroin, morphine, methadone, |
| codeine, Oxycotin, Percocet, Vicodin, etc.)") |
| Opioids |
| Opiolas |
| Shortname / Alias: opioids3months |
| ID: 291 |
| In the past 3 months, how often have you used opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

**Page entry logic:** This page will show when: #143 Question "In the past 3 months, how often have you used opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?" is one of the following answers ("Once or twice", "Monthly", "Weekly", "Daily or almost daily")

### **Opioids (cont.)**

() Never

() Once or twice

Logic: Show/hide trigger exists.

Shortname / Alias: opioidsheroin

| ID: 299 |
|---|
| In the past 3 months, has your opioid use included heroin?* ( ) Yes |
| ( ) No |
| Logic: Hidden unless: #144 Question "In the past 3 months, has your opioid use included heroin?" is one of the following answers ("Yes") |
| Shortname / Alias: heroinprimary |
| ID: 300 |
| In the past 3 months, was heroin the most common opioid that you used?* |
| ( ) No |
| Shortname / Alias: opioidssdesire |
| Shortname / Alias: opioidssdesire ID: 293 |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |

| Sexual Behaviors |
|---|
| In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) No ( ) Yes |
| ID: 297 |
| Shortname / Alias: opioidsstop |
| () Yes |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) No |
| ID: 296 |
| Shortname / Alias: opioidsfriend |
| ( ) Daily or almost daily |
| () Weekly |
| ( ) Monthly |
| ( ) Once or twice |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* () Never |
| ID: 295 |
| Shortname / Alias: opioidsfailed |
| ( ) Daily or almost daily |
| () Weekly |
| ( ) Monthly |

Page exit logic: Skip / Disqualify LogicIF: #151 Question "In the past 3 months, how many people have you had anal sex with?" is exactly equal to "0" THEN: Jump to page 120 - Perceived HIV Risk

The next section of questions will ask about your sexual behaviors. We know that this can be a sensitive topic, so we would like to remind you that your answers will be kept completely confidential. Please be as honest as possible in order to ensure the success of the current study.

The following questions refer to your sexual behavior during the past 3 months. Our focus will be only on anal sex. Therefore, do not include references to people with whom you did not engage in anal sex.

For these questions, anal sex refers to sex where the other person's penis was in your rectum (you were the bottom) and to sex where your penis was in the other person's rectum (you were the top).

These questions only ask about people assigned male at birth, which includes cisgender men (men assigned male at birth) and transgender women (women assigned male at birth). Therefore, do not include references to cisgender women (women assigned female at birth) or transgender men (men assigned female at birth).

Validation: Min = 0 Max = 999 Must be numeric Whole numbers only Positive numbers only

Shortname / Alias: numsexpartner

ID: 302

In the past 3 months, how many people have you had anal sex with?\*

\_\_\_\_\_

**Page entry logic:** This page will show when: #151 Question "In the past 3 months, how many people have you had anal sex with?" is greater than "0"

#### **HIV Status of Sexual Partners**

Logic: Hidden by default

ID: 677

The total number must equal the number of people you had anal sex with in the last 3 months ([question('value'), id='302']). Please correct this.

Validation: Must be numeric

Shortname / Alias: partnerhivstatus

Before you had sex, what did you know of the HIV status of your sexual partner(s)? Enter numerical values. Numbers must add up to [question('value'), id='302'], the number of people you reported having anal sex within the last three months.\* This person/these people told you they were HIV negative and you had no reason to doubt it You knew this person/these people were HIV positive You were not completely sure of this person/these people's HIV status Action: Custom Script: Script to check the continuous sum totals **Hidden Value: Num HIV Neg partners** Value: [question("option value"), id="676", option="12278"] **Hidden Value: Num HIV Pos partners** Value: [question("option value"), id="676", option="12279"] **Hidden Value: Num HIV Unk partners** Value: [question("option value"), id="676", option="12280"]

Page entry logic: This page will show when: Num HIV Neg partners is greater than "0"

### **HIV Negative Partners**

ID: 690

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Shortname / Alias: hivneg timesbot

| In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom?* |
|---|
| Shortname / Alias: hivneg_timestop ID: 702 |
| In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the top?* |
| Page entry logic: This page will show when: #153 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom?" is greater than "0" |
| HIV Negative Partners - Condomless Receptive Al |
| Logic: Hidden by default ID: 714 |
| This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='701']). Please correct this. |
| Shortname / Alias: hivneg_timesbotunp ID: 710 |
| In the past 3 months, how many of the [question('value'), id='701'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom were without a condom? * |
| Action: Custom Script: Check number condomless is not greater than total times |

**Page entry logic:** This page will show when: #155 Question "In the past 3 months, how many of the [question('value'), id='701'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom were without a condom? " is greater than "0"

### **HIV Negative Partners - Condomless Receptive Al**

ID: 721

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 999

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivneg\_botunp\_typ

ID: 711

Regarding the partners who told you they were HIV negative who you had <u>condomless receptive</u> anal sex with (where you were the bottom), how many were...

Enter numerical values.\*

| Romantic partner(s), someone you are in a relationship with |
|-------------------------------------------------------------|
| Casual hook-up(s) or one-night stand(s) |

\_\_\_\_A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc.

Logic: Hidden by default

ID: 1002

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivneg botunp gender

| ID: 964 |
|---|
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| <b>Page entry logic:</b> This page will show when: #154 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the top?" is greater than "0" |
| HIV Negative Partners - Condomless Insertive Al |
| ID: 722 |
| ID. 122 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative. |
| opasii 1227 o j coxuur pururer (e) iii tiid tuot o monure <u>who totu you tirey word fiir mogativor</u> |
| Logic: Hidden by default |
| ID: 719 |
| This number cannot be greater than the number of times you had anal sex where you were the top ([question('value'), id='702']). Please correct this. |
| top ([question( value ), Id= 702 ]). I lease correct this. |
| Shortname / Alias: hivneg_timestopunp |
| ID: 718 |
| In the past 3 months, how many of the [question('value'), id='702'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the top were without a condom? * |

| <b>Action: Custom Scrip</b> | ot: Script to check num | ber condomless is not | greater than the totals |
|---|---|---|---|
|---|---|---|---|

**Page entry logic:** This page will show when: #158 Question "In the past 3 months, how many of the [question('value'), id='702'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the top were without a condom?" is greater than "0"

### **HIV Negative Partners - Condomless Insertive Al**

ID: 723

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 1004

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivneg topunp typ

ID: 725

Regarding the partners who told you they were HIV negative who you had <u>condomless insertive</u> <u>anal sex with (where you were the top)</u>, how many were...

#### Enter numerical values.\*

\_\_\_\_\_Romantic partner(s), someone you are in a relationship with \_\_\_\_\_\_Casual hook-up(s) or one-night stand(s)

\_\_\_\_A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc.

Logic: Hidden by default

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivneg_topunp_gender |
| ID: 965 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: Num HIV Neg partners is greater than "0" |
| HIV Negative Partners - PrEP and Alcohol and Drug Use |
| ID: 992 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative. |
| Logic: Hidden by default |

This number cannot be greater than the number of partners who told you they were HIV negative

([question('option value'), id='676', option='12278']). Please correct this.

Shortname / Alias: hivneg\_toldyouprep

How many of your sexual partners who told you they were HIV negative told you they were taking PrEP?

Number must be less than or equal to [question('option value'), id='676', option='12278'].\*

\_\_\_\_\_

Logic: Show/hide trigger exists.

Shortname / Alias: hivneg youtoldprep

ID: 730

Regarding your sexual partners who told you they were HIV negative, did you tell any of them that you were taking PrEP?\*

() Yes

() No

() I was not taking PrEP at this time

Logic: Hidden by default

ID: 733

This number cannot be greater than the number of partners who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Logic: Hidden unless: #162 Question "Regarding your sexual partners who told you they were HIV negative, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivneg youtoldprepnum

ID: 731

How many of your sexual partner(s) who told you they were HIV negative did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12278'].\*

Shortname / Alias: hivneg timesdrunk

ID: 740

In the past 3 months, how many of the times you had anal sex with partners who told you they were HIV negative were you or this person under the influence of alcohol or drugs?\*

\_\_\_\_\_

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Page entry logic: This page will show when: Num HIV Pos partners is greater than "0"

#### **HIV Positive Partners**

ID: 770

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Shortname / Alias: hivpos timesbot

ID: 775

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom?\*

\_\_\_\_\_

Shortname / Alias: hivpos timestop

ID: 776

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the top?\*

\_\_\_\_\_\_

**Page entry logic:** This page will show when: #165 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom?" is greater than "0"

**HIV Positive Partners - Condomless Receptive AI** 

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 783

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='775']). Please correct this.

Shortname / Alias: hivpos timesbotunp

ID: 784

In the past 3 months, how many of the [question('value'), id='775'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom were without a condom? \*

Action: Custom Script: Check number condomless is not greater than total times

**Page entry logic:** This page will show when: #167 Question "In the past 3 months, how many of the [question('value'), id='775'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom were <u>without a condom?</u> " is greater than "0"

**HIV Positive Partners - Condomless Receptive AI** 

ID: 786

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 1008

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivpos_botunp_typ |
| ID: 788 |
| Regarding the partners who told you they were HIV positive who you had <u>condomless receptive</u> <u>anal sex with (where you were the bottom)</u> , how many were |
| Enter numerical values.* |
| Romantic partner(s), someone you are in a relationship with |
| Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |
| Logic: Hidden by default |
| ID: 1009 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivpos_botunp_gender |
| ID: 994 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, and gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |

**Page entry logic:** This page will show when: #166 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the top?" is greater than "0"

#### **HIV Pos Partners - Condomless Insertive AI**

ID: 792

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 793

This number cannot be greater than the number of times you had anal sex where you were the top ([question('value'), id='776']). Please correct this.

Shortname / Alias: hivpos timestopunp

ID: 794

In the past 3 months, how many of the [question('value'), id='776'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the top were without a condom? \*

\_\_\_\_\_

Action: Custom Script: Script to check number condomless is not greater than the totals

**Page entry logic:** This page will show when: #170 Question "In the past 3 months, how many of the [question('value'), id='776'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the top were without a condom? " is greater than "0"

**HIV Positive Partners - Condomless Insertive AI** 

ID: 796

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this. |
|---|
| Validation: Must be numeric |
| Shortname / Alias: hivpos_topunp_typ |
| ID: 798 |
| Regarding the partners who told you they were HIV positive who you had <u>condomless insertive</u> anal sex with (where you were the top), how many were |
| Enter numerical values.*Romantic partner(s), someone you are in a relationship with |
| Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |
| Logic: Hidden by default |
| ID: 1013 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivpos_topunp_gender |
| ID: 995 |
| How many were |
| Enter numerical values.* |

Action: Custom Script: Script to check continuous sum totals

Logic: Hidden by default

ID: 1012

274

Action: Custom Script: Script to check continuous sum totals

Page entry logic: This page will show when: Num HIV Pos partners is greater than "0"

#### **HIV Positive Partners - HIV Trt and PrEP**

Logic: Hidden by default

ID: 799

This number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Shortname / Alias: hivpos\_toldyouhivmeds

ID: 800

How many of your sexual partners who told you they were HIV positive told you they were taking medication to treat HIV?

Number must be less than or equal to [question('option value'), id='676', option='12279'].

\_\_\_\_\_

Logic: Hidden by default

ID: 920

The number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Shortname / Alias: hivpos toldyouundetect

ID: 918

How many of your sexual partners who told you they were HIV positive told you they were undetectable?

**Number must be less than or equal to** [question('option value'), id='676', option='12279'].

\_\_\_\_\_

Logic: Show/hide trigger exists.

Shortname / Alias: hivpos youtoldprep

| Regarding your s | exual partners w | ho told you the | y were HIV | positive, did | you tell any | of them that |
|---|---|---|---|---|---|---|
| you were taking F | PrEP?* | | | | | |

() Yes

() No

() I was not taking PrEP at this time

Logic: Hidden by default

ID: 802

This number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Logic: Hidden unless: #175 Question "Regarding your sexual partners who told you they were HIV positive, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivpos youtoldprepnum

ID: 803

How many of your sexual partner(s) who told you they were HIV positive did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12279'].

\_\_\_\_\_\_

Shortname / Alias: hivpos timesdrunk

ID: 807

In the past 3 months, how many of the times you had anal sex with partners who told you they were HIV positive were you or this person under the influence of alcohol or drugs?\*

Action: Custom Script: Script to check med number not greater than the total number of partners

Action: Custom Script: Script to check undetectable number not greater than the total number of partners

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Page entry logic: This page will show when: Num HIV Unk partners is greater than "0"

#### **HIV Status Unknown Partners**

ID: 810

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Shortname / Alias: hivunk\_timesbot

ID: 815

In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom?\*

Shortname / Alias: hivunk\_timestop

ID: 816

In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?\*

**Page entry logic:** This page will show when: #178 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of <a href="where you were the bottom?">where you were the bottom?</a>" is greater than "0"

## **HIV Status Unknown Partners - Condomless Receptive AI**

ID: 822

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='815']). Please correct this.

Shortname / Alias: hivunk\_timesbotunp

ID: 824

In the past 3 months, how many of the [question('value'), id='815'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom were without a condom? \*

Action: Custom Script: Check number condomless is not greater than total times

**Page entry logic:** This page will show when: #180 Question "In the past 3 months, how many of the [question('value'), id='815'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom were without a condom? " is greater than "0"

### **HIV Status Unknown Partners - Condomless Receptive AI**

ID: 826

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 1016

The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivunk\_botunp\_typ

| Regarding the partners whose HIV status you were not sure of who you had <u>condomless</u> <u>receptive anal sex with (where you were the bottom)</u> , how many were |
|---|
| Enter numerical values.* Romantic partner(s), someone you are in a relationship with Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |
| Logic: Hidden by default |
| ID: 1017 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. |
| Validation: Must be numeric |
| Validation: Must be numeric Shortname / Alias: hivunk_botunp_gender ID: 996 |
| Shortname / Alias: hivunk_botunp_gender |
| Shortname / Alias: hivunk_botunp_gender ID: 996 |
| Shortname / Alias: hivunk_botunp_gender ID: 996 How many were Enter numerical values.* |
| Shortname / Alias: hivunk_botunp_gender ID: 996 How many were Enter numerical values.*Men |

**Action: Custom Script: Script to check continuous sum totals** 

Action: Custom Script: Script to check continuous sum totals

**Page entry logic:** This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?" is greater than "0"

**HIV Status Unknown Partners - Condomless Insertive AI** 

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 833

This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this.

Shortname / Alias: hivunk timestopunp

ID: 834

In the past 3 months, how many of the [question('value'), id='816'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top were without a condom?\*

Action: Custom Script: Script to check number condomless is not greater than the totals

**Page entry logic:** This page will show when: #183 Question "In the past 3 months, how many of the [question('value'), id='816'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top were without a condom?" is greater than "0"

HIV Status Unknown Partners - Condomless Insertive Al

ID: 836

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivunk_topunp_typ |
| ID: 838 |
| Regarding the partners whose HIV status you were not sure of who you had <u>condomless</u> <u>insertive anal sex with (where you were the top)</u> , how many were |
| Enter numerical values.* Romantic partner(s), someone you are in a relationship with Casual hook-up(s) or one-night stand(s) A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |
| Logic: Hidden by default |
| ID: 1021 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivunk_topunp_gender |
| ID: 997 |
| How many were |
| Enter numerical values.*MenTranswomenNon-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals Action: Custom Script: Script to check continuous sum totals |

Page entry logic: This page will show when: Num HIV Unk partners is greater than "0"

#### **HIV Status Unknown Partners - PrEP**

Logic: Hidden by default

ID: 839

This number cannot be greater than the number of partners whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Shortname / Alias: hivunk\_toldyouprep

ID: 840

How many of your sexual partners whose HIV status you were not sure of told you they were taking PrEP?

Number must be less than or equal to [question('option value'), id='676', option='12280'].\*

\_\_\_\_\_\_

Logic: Show/hide trigger exists.

Shortname / Alias: hivunk youtoldprep

ID: 841

Regarding your sexual partners whose HIV status you were not sure of, did you tell any of them that you were taking PrEP?\*

- () Yes
- () No
- () I was not taking PrEP at this time

Logic: Hidden by default

ID: 842

This number cannot be greater than the number of partners whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Logic: Hidden unless: #187 Question "Regarding your sexual partners whose HIV status you were not sure of, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivunk youtoldprepnum

ID: 843

How many of your sexual partner(s) whose HIV status you were not sure of did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12280'].\*

\_\_\_\_\_

Shortname / Alias: hivunk timesdrunk

ID: 847

In the past 3 months, how many of the times you had anal sex with partners whose HIV status you were not sure of were you or this person under the influence of alcohol or drugs?\*

\_\_\_\_\_\_

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

#### **Perceived HIV Risk**

Shortname / Alias: perceivedrisk1

ID: 762

Based on your reported sexual activities over the last 3 months, how at risk do you think you were for contracting HIV in the last 3 months?\*

- () Not at all at risk for contracting HIV
- () Somewhat at risk for contracting HIV
- () High risk for contracting HIV

Shortname / Alias: perceivedrisk2

ID: 763

What is your gut feeling about how likely you are to get infected with HIV?\*

- () Extremely unlikely
- () Very unlikely
- () Somewhat likely
- () Very likely
- () Extremely likely

Shortname / Alias: perceivedrisk3 ID: 764 I worry about getting infected with HIV:\* () None of the time () Rarely () Some of the time () A moderate amount of time () A lot of the time () All of the time **Perceived HIV Risk** Shortname / Alias: perceivedrisk4 ID: 765 Getting HIV is something I am...\* () Not concerned about () A little concerned about () Moderately concerned about () Concerned about a lot () Extremely concerned about Shortname / Alias: perceivedrisk5 ID: 766 There is a chance, no matter how small, I could get HIV:\* () Strongly Disagree () Disagree () Agree () Strongly Agree

Shortname / Alias: perceivedrisk6

ID: 767

I think my chances of getting infected with HIV are:\*

() Zero

| () Almost zero |
|----------------|
| () Small |
| () Moderate |
| ( ) Large |

() Very large

### PHQ-2/GAD-2

ID: 768

Now we are going to ask you about your mental health and how you have been feeling recently.

Shortname / Alias: mentalhealthscreener

ID: 388

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Little interest or pleasure in doing things | () | () | () | () |
| Feeling<br>down,<br>depressed,<br>or<br>hopeless | () | () | () | () |
| Feeling<br>nervous,<br>anxious or<br>on edge | () | () | () | () |
| Not being<br>able to<br>stop or | () | () | () | () |

| control<br>worrying |
|---------------------|
|---------------------|

### **Hidden Mental Health Screener Script**

Hidden Value: psychdistress1

Value:

Hidden Value: psychdistress2

Value:

**Action: Custom Script: Mental Health Script** 

Page entry logic: This page will show when: psychdistress1 is greater than or equal to "3"

### PHQ-8

Shortname / Alias: phq8

ID: 397

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Trouble falling or staying asleep, or sleeping too much | () | () | () | () |
| Feeling tired<br>or having<br>little energy | () | () | () | () |

| | | | | _ |
|---|---|---|---|---|
| Poor appetite or overeating | () | () | () | () |
| Feeling bad<br>about<br>yourself - or<br>that you are<br>a failure or<br>have let<br>yourself or<br>your family<br>down | () | () | () | () |
| Trouble concentrating on things, such as reading the newspaper or watching television | () | () | () | () |
| Moving or<br>speaking so<br>slowly that<br>other people<br>could have<br>noticed, or<br>the opposite<br>- being so<br>fidgety or<br>restless that<br>you have<br>been moving<br>around a lot<br>more than<br>usual | () | () | () | () |

Page entry logic: This page will show when: psychdistress2 is greater than or equal to "3"

## GAD-7

Shortname / Alias: gad7

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Worrying<br>too much<br>about<br>different<br>things | () | () | () | () |
| Trouble relaxing | () | () | () | () |
| Being so<br>restless<br>that it is<br>hard to sit<br>still | () | () | () | () |
| Becoming<br>easily<br>annoyed<br>or irritable | () | () | () | () |
| Feeling<br>afraid as if<br>something<br>awful<br>might<br>happen | () | () | () | () |

### **Social Isolation**

Shortname / Alias: socialisolation

ID: 432

Please respond to each item by marking one circle per row.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---------------------|-------|--------|-----------|---------|--------|
| I feel<br>left out. | () | () | () | () | () |
| I feel<br>that<br>people<br>barely<br>know<br>me. | () | () | () | () | () |
|---------------------------------------------------|----|----|----|----|----|
| I feel isolated from others. | () | () | () | () | () |
| I feel that people are around me but not with me. | () | () | () | () | () |

# **Emotional Support**

Shortname / Alias: emotionalsupport

ID: 411

Please respond to each item by marking one circle per row.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| I have someone who will listen to me when I need to talk. | () | () | () | () | () |
| I have someone to confide in or talk to about myself or my problems. | () | () | () | () | () |
| I have someone | () | () | () | () | () |

| who makes<br>me feel<br>appreciated. | | | | | |
|---|---|---|---|---|---|
| I have<br>someone to<br>talk with<br>when I have<br>a bad day. | () | () | () | () | () |

# **Informational Support**

Shortname / Alias: informational support

ID: 417

Please respond to each item by marking one circle per row.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| I have someone to give me good advice about a crisis if I need it. | () | () | () | () | () |
| I have someone to turn to for suggestions about how to deal with a problem. | () | () | () | () | () |
| I have someone to give me information if I need it. | () | () | () | () | () |
| I get useful<br>advice<br>about<br>important | () | () | () | () | () |

# **Instrumental Support**

Shortname / Alias: instrumentalsupport

ID: 422

Please respond to each item by marking one circle per row.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| Do you have someone to help you if you are confined to bed? | () | () | () | () | () |
| Do you have someone to take you to the doctor if you need it? | () | () | () | () | () |
| Do you have someone to help with your daily chores if you are sick? | () | () | () | () | () |
| Do you<br>have<br>someone<br>to run<br>errands | () | () | () | () | () |

## Companionship

Shortname / Alias: companionship

ID: 427

Please respond to each item by marking one circle per row.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| Do you have someone with whom to have fun? | () | () | () | () | () |
| Do you have someone with whom to relax? | () | () | () | () | () |
| Do you have someone with whom you can do something enjoyable? | () | () | () | () | () |
| Do you find companionship when you want it? | () | () | () | () | () |

## Thank You!

ID: 1

Thank you for taking this survey and for participating! We greatly appreciate your involvement!

## P3-T RCT Month-6 Follow-up

ID: 93

Thank you for participating in the P3-T study! The purpose of the study is to test a PrEP adherence intervention for young men who have sex with men who are starting PrEP. As part of the P3-T study, there are three surveys: one when you enrolled, one at your follow up appointment today, and one at your follow up appointment in 3 months.

Try to answer every question as best you can. If you need help, please ask the study staff. Your answers will be used only for research purposes. Let's get started!

#### **Cell Phone**

ID: 120

Now, we'd like to ask you about your cell phone and internet use.

Logic: Show/hide trigger exists.

Shortname / Alias: paychange

ID: 1068

In the last 3 months, has who pays for your cellphone or smart phone changed?\*

- () Yes
- () No

Logic: Hidden unless: #2 Question "In the last 3 months, has who pays for your cellphone or smart phone changed?" is one of the following answers ("Yes")

Shortname / Alias: phonepay

ID: 127

Who usually pays for your cell phone or smartphone plan?\*

- ( ) I do
- () Someone else does

Logic: Show/hide trigger exists.

Shortname / Alias: disconnect

| () res |
|---|
| ( ) No |
| Logic: Hidden unless: #4 Question "In the last 3 months, did you ever not have access to your |
| phone or phone service?" is one of the following answers ("Yes") |
| Shortname / Alias: disconnecttimes |
| ID: 129 |
| How many times in the last 3 months did you not have access to your phone or phone service?* |
| () Once |
| () Twice |
| ( ) 3 to 5 times |
| () More than 5 times |
| Logic: Hidden unless: #4 Question "In the last 3 months, did you ever not have access to your |
| phone or phone service?" is one of the following answers ("Yes") |
| Shortname / Alias: disconnectlength |
| ID: 130 |
| The <i>last</i> time you did not have access to your phone or phone service, for how long did you not |
| have access?* |
| () 1 day or less |
| ( ) 2 to 6 days |
| () 1 to 4 weeks |
| ( ) More than 4 weeks |
| Employment, Income |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: employed |
| ID: 109 |
| Are you currently employed?* ( ) Yes |
| ( ) No |

Logic: Hidden unless: #7 Question "Are you currently employed?" is one of the following

answers ("Yes")

Shortname / Alias: employedhours

In the last 3 months, did you ever not have access to your phone or phone service?\*

294

| ID: 110 |
|---|
| Are you employed full-time or part-time? Part-time means that you work less than 35 hours per week during most weeks.* ( ) Full time |
| ( ) Part time |
| Shortname / Alias: income_30d |
| ID: 564 |
| How much money did you make altogether during the past 30 days?* |
| ( ) Don't know |
| Shortname / Alias: incomelevel |
| ID: 111 |
| How would you describe your income level?* ( ) Low income |
| ( ) Middle income |
| () High income |
| ( ) Decline to answer |
| Food, Shelter |
| 1 Ood, Olleitei |
| Shortname / Alias: cutmeal |
| ID: 112 |
| In the past 3 months, how often did you or your family have to cut meal size or skip a meal because there was not enough money for food?* ( ) Almost every week |
| ( ) Several weeks but not every week |
| ( ) Only a few weeks |
| ( ) Did not have to skip or cut the size of meals |
| ( ) Dia not have to only of out the olde of modic |
| Shortname / Alias: shelter |

In the past 3 months, have you spent at least one night (check all that apply):\*

[] In a public place not intended for sleeping (e.g., bus station, car, abandoned building)?

ID: 113

[] In a shelter?

| [] On the street or anywhere outside (e.g., park, sidewalk)? |
|---|
| [] Temporarily doubled up with a friend or family member? |
| [] In a temporary housing program? |
| [] In a welfare or voucher hotel/motel? |
| [] In jail, prison, or a halfway house? |
| [] In drug treatment, a detox unit, or drug program housing? |
| [] In a hospital, nursing home, or hospice? |
| [] I have not spent a night in any of the above places. |
| Insurance |
| Shortname / Alias: insurance |
| ID: 206 |
| Do you currently have health insurance or health care coverage? ( ) Yes |
| ( ) No |
| ( ) I don't know |
| Sexual Identity, Relationships |
| ID: 565 |
| The following questions ask about your sexual identity and relationship status. |
| Please answer to the best of your ability. |
| Shortname / Alias: sexualid |
| ID: 102 |
| What is your current sexual identity?* ( ) Gay, homosexual, same gender loving |
| () Bisexual |
| () Queer |
| ( ) Straight or heterosexual |
| ( ) Other, specify::* |
| Shortname / Alias: relationship |

### How do you define your primary relationship status?\*

- () Single, not currently dating
- () Single, casually dating
- () In a relationship
- () Married or other legal commitment

**Page entry logic:** This page will show when: #20 Question "How do you define your primary relationship status?" is one of the following answers ("In a relationship","Married or other legal commitment")

#### **Sexual Health Priorities with Partner**

ID: 566

People have different sexual health priorities. For example, some people prioritize staying HIV-negative; others want to have as much fun as possible with their partners; others want to feel as close and connected to their partners as possible.

For these next questions, we are interested in you and your primary romantic partner's sexual health priorities.

Shortname / Alias: shpriorities\_scale

ID: 569

Thinking about you and your partner's sexual health priorities, please indicate the extent to which you agree or disagree with the following statements.\*

| | Strongly<br>Agree | Agree | Disagree | Strongly<br>Disagree |
|---|---|---|---|---|
| I feel like my partner and I are "on the same page" in terms of the decisions we make about sexual health and risk | () | () | () | () |
| When it comes to sexual decision-making, I feel like my partner and | () | () | () | () |

| I are "of the same mind" | | | | |
|---|---|---|---|---|
| Sometimes I feel like my priorities for my sexual health are incompatible with my partner's goals | () | () | () | () |
| I'm confident that my partner and I generally share the same priorities when it comes to sexual health | () | () | () | () |
| Making sexual health decisions with my partner can be difficult because we have different priorities | () | () | () | () |

## **Health Providers**

ID: 157

Now, we are going to ask you about your health care and health care decision making.

Logic: Show/hide trigger exists.

| Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?* ( ) Yes |
|---|
| ( ) No |
| Logic: Hidden unless: #22 Question "Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?" is one of the following answers ("Yes") |
| Shortname / Alias: pcpawareness |
| ID: 105 |
| How open are you about your sexual identity to your primary medical care provider?* ( ) Primary medical provider definitely does NOT know your sexual identity |
| ( ) Primary medical provider MIGHT know about your sexual identity |
| ( ) Primary medical provider PROBABLY knows about your sexual identity |
| ( ) Primary medical provider DEFINITELY knows about your sexual identity |
| Logic: Hidden unless: #22 Question "Do you have a primary health care provider (for example, a pediatrician, a doctor, or other health care provider that you see regularly)?" is one of the following answers ("Yes") |
| Shortname / Alias: pcptalksex |
| ID: 160 |
| How comfortable are you discussing your sexual behavior with your primary health care provider?* ( ) Very comfortable ( ) Somewhat comfortable |
| ( ) Somewhat uncomfortable |
| `` |
| ( ) Very uncomfortable |
| STI Testing |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: stitest3m |
| ID: 170 |

Shortname / Alias: pcp

| A sexually transmitted infection (STI) is an infection transmitted through sexual activity, such as syphilis, gonorrhea, chlamydia, herpes, or genital warts. In the past 3 months, have you been tested for an STI that was not HIV?* () Yes |
|---|
| ( ) No |
| Logic: Hidden unless: #25 Question "A sexually transmitted infection (STI) is an infection transmitted through sexual activity, such as syphilis, gonorrhea, chlamydia, herpes, or genital warts. In the past 3 months, have you been tested for an STI that was not HIV?" is one of the following answers ("Yes") |
| Shortname / Alias: sti3mo |
| ID: 171 |
| Please indicate whether you have been diagnosed with any of the following sexually transmitted infections in the past 3 months. Please select all that apply.* [] Chlamydia |
| [] Genital warts, anal warts, HPV |
| [] Gonorrhea |
| [] Hepatitis B |
| [] Hepatitis C |
| [] Herpes, HSV1/HSV2 |
| [] Syphilis |
| [] Urethritis |
| [] Other, please specify:: |
| [] None of these |
| HIV Testing |
| Shortname / Alias: recenthivtest_mon |
| ID: 165 |
| When did you have your most recent HIV test? |
| Please enter the month and year. |
| Month:* ( ) January |
| () February |

| () March |
|---|
| ( ) April |
| ( ) May |
| () June |
| ( ) July |
| ( ) August |
| () September |
| () October |
| ( ) November |
| () December |
| Validation: Min = 1980 Must be numeric Whole numbers only Positive numbers only Max character count |
| = 4 |
| Shortname / Alias: recenthivtest_yr |
| ID: 166 |
| Year:* |
| Page entry logic: This page will show when: (#27 Question "When did you have your most recent HIV test? |
| test? |
| Please enter the month and year. |
| Please enter the month and year. |
| test? Please enter the month and year. Month:" AND #28 Question "Year:" ) |
| test? Please enter the month and year. Month:" AND #28 Question "Year:" ) PrEP Use |
| test? Please enter the month and year. Month:" AND #28 Question "Year:" ) PrEP Use Shortname / Alias: prepstartafterP3-T |
| test? Please enter the month and year. Month: AND #28 Question "Year:") PrEP Use Shortname / Alias: prepstartafterP3-T ID: 1201 Did you start taking PrEP after you started the P3-T study?* |
| test? Please enter the month and year. Month:" AND #28 Question "Year:" ) PrEP Use Shortname / Alias: prepstartafterP3-T ID: 1201 Did you start taking PrEP after you started the P3-T study?* ( ) Yes |

Logic: Show/hide trigger exists.

| Are you taking PrEP right now?* ( ) Yes |
|---|
| ( ) No |
| Logic: Hidden unless: Fix logic- If no to Did you start taking PrEP after you enrolled in P3-T |
| Shortname / Alias: noprep_why |
| ID: 1203 |
| Why did you decide not to start PrEP? Select all of the factors below that were related to why you didn't start PrEP.* [] I couldn't afford it |
| [] I was not having sex |
| [] I was no longer having sex with a person living with HIV |
| [] I was only having sex with one person and they were undetectable or HIV negative |
| [] I didn't want to take a pill every day |
| [] My parent(s) or guardian(s) found out and wouldn't let me start |
| [] I kept forgetting to take my pill |
| [] I could no longer see my PrEP provider and haven't found another PrEP provider |
| [] I was worried about experiencing side effects |
| [] I was worried about the long term effects of PrEP on my health |
| [] It was medically unsafe for me to take PrEP (due to kidney/renal function, bone density, or another medical issue) |
| [] I was worried that if I were to become HIV-positive certain medications may no longer work or I might be resistant to them |
| [] I was worried that PrEP might not provide complete protection against HIV |
| [] I started using condoms all of the time |
| [] I was worried that the medication would taste bad and/or the pill would be too big |
| [] Other, please specify:: |

**Page entry logic:** This page will show when: #32 Question "Why did you decide not to take PrEP? Select all of the factors below that were related to why you didn't take PrEP."

## PrEP Use, why didn't start

Shortname / Alias: nowprep

ID: 1202

Action: Custom Script: Script to count checkboxes and skip if q <2

ID: 1204

Piping: Piped Values From Question 32. (Why did you decide not to take PrEP? Select all of the factors below that were related to why you didn't take PrEP.)

Please rank the reasons you did not start taking PrEP in order of importance.\*

Page entry logic: Fix logic- If yes to Did you start taking PrEP after you enrolled in P3-T

### **PrEP Start**

Shortname / Alias: startprep why

| ID: 943 |
|---|
| Why did you choose to start taking PrEP? Select all that apply.* [] I'm having sex with or thinking about having sex with someone who is HIV+ |
| [] I'm having sex with or thinking about having sex with someone whose HIV status I don't know |
| [] I want to be in control of my sexual health |
| [] I want to reduce my anxiety around sex |
| [] I want to increase my sexual satisfaction and intimacy |
| [] I want to be safe and healthy |
| [] I want to have a better future |
| [] I am having sex with multiple partners |
| [] I don't like to use condoms |
| [] My partner won't use condoms |
| [] I had a previous HIV scare |
| [] My health care provider recommended it |
| [] I was recently diagnosed with an STI |
| [] Many people in my community take PrEP |
| [] Other, please specify:: |

#### **PrEP Start**

Action: Custom Script: Script to count checkboxes and skip q if < 2

Shortname / Alias: startprep primwhy

ID: 945

Piping: Piped Values From Question 34. (Why did you choose to start taking PrEP? Select all that apply.)

What was the main reason you started PrEP?\*

**Page entry logic:** This page will show when: (#30 Question "Did you start taking PrEP after you started the P3-T study?" is one of the following answers ("Yes") OR #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes"))

### **PrEP Start and Stop**

Validation: %s format expected

Logic: Hidden unless: #30 Question "Did you start taking PrEP after you started the P3-T study?"

is one of the following answers ("Yes")

Shortname / Alias: prep\_firststart

ID: 947

When did you start taking PrEP after enrolling in P3-T?

If you do not know the exact day of the month, please give your best estimate. \*

\_\_\_\_\_

Logic: Hidden unless: #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes")

Shortname / Alias: prepstoP3-Tmo

ID: 576

Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?\*

() Yes

() No

**Action: Custom Script: Check date not in future** 

Action: Custom Script: Script to populate - 3 months date

Hidden Value: Date for prompt - today minus 3 months

Value:

**Page entry logic:** This page will show when: #37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes")

### PrEP Stop, last 3 months



The date re-started is before the date stopped. Please correct this.

Logic: Hidden unless: #38 Question "How many times did you <u>stop taking PrEP for 7 days in a row or more</u> in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("1")

Shortname / Alias: time1 dates

ID: 1027

ID: 1159

Please enter the dates you were off PrEP (from [question('value'), id='1026'] to today):

Validation: %s format expected

| Validation: %s format expected |
|---|
| ID: 1029 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1160 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("2","3","4","5","6","7","8","9","10","11","12 or more") |
| Shortname / Alias: timefirst_dates |
| ID: 1030 |
| Please enter the dates you were off PrEP for the first time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1031 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1032 |
| Date re-started:*: |
| Date re-started:*: |
| Date re-started:*: |
| Date re-started:*: Logic: Hidden by default |
| Logic: Hidden by default ID: 1161 |
| Logic: Hidden by default |

Date stopped:\*:

Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("2","3","4","5","6","7","8","9","10","11","12 or more")

Shortname / Alias: timesecond\_dates

| Please enter the dates you were <u>off</u> PrEP for the <u>second</u> time (from [question('value'), id='1026'] to today): |
|---|
| Validation: %s format expected |
| ID: 1034 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1035 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1162 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("3","4","5","6","7","8","9","10","11","12 or more") |
| Shortname / Alias: timethird_dates |
| ID: 1036 |
| Please enter the dates you were off PrEP for the third time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1037 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1038 |
| Date re-started:*: |
| Logic: Hidden by default |

The date re-started is before the date stopped. Please correct this.

| Logic: Hidden unless: #38 Question "How many times did you <u>stop taking PrEP for 7 days in a row or more</u> in the last three months ( <i>from [question('value'), id='1026'] to today)</i> ?" is one of the following answers ("4","5","6","7","8","9","10","11","12 or more") |
|---|
| Shortname / Alias: timefourth_dates ID: 1039 |
| Please enter the dates you were <u>off</u> PrEP for the <u>fourth</u> time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected ID: 1040 |
| Date stopped:*: |
| Validation: %s format expected ID: 1041 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1164 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefifth_dates |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefifth_dates ID: 1042 Please enter the dates you were off PrEP for the fifth time (from [question('value'), |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefifth_dates ID: 1042 Please enter the dates you were off PrEP for the fifth time (from [question('value'), id='1026'] to today): |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefifth_dates ID: 1042 Please enter the dates you were off PrEP for the fifth time (from [question('value'), id='1026'] to today): Validation: %s format expected |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefifth_dates ID: 1042 Please enter the dates you were off PrEP for the fifth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1043 Date stopped:*: Validation: %s format expected |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefifth_dates ID: 1042 Please enter the dates you were off PrEP for the fifth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1043 Date stopped:*: |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefifth_dates ID: 1042 Please enter the dates you were off PrEP for the fifth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1043 Date stopped:*: Validation: %s format expected |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("5","6","7","8","9","10","11","12 or more") Shortname / Alias: timefifth_dates ID: 1042 Please enter the dates you were off PrEP for the fifth time (from [question('value'), id='1026'] to today): Validation: %s format expected ID: 1043 Date stopped:*: |

| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("6","7","8","9","10","11","12 or more") |
|---|
| Shortname / Alias: timesixth_dates |
| ID: 1045 |
| Please enter the dates you were <u>off</u> PrEP the <u>sixth</u> time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1046 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1047 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1166 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("7","8","9","10","11","12 or more") |
| Shortname / Alias: timeseventh_dates |
| ID: 1048 |
| Please enter the dates you were off PrEP for the seventh time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1049 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1050 |
| Date re-started:*: |

| ID: 1167 |
|---|
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("8","9","10","11","12 or more") |
| Shortname / Alias: timeeighth_dates |
| ID: 1051 |
| Please enter the dates you were off PrEP for the eighth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1052 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1053 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1168 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("9","10","11","12 or more") |
| Shortname / Alias: timeninth_dates |
| ID: 1054 |
| Please enter the dates you were off PrEP for the ninth time (from [question('value'), id='1026'] to today): |
| Validation: %s format expected |
| ID: 1055 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1056 |
| 310 |

Logic: Hidden by default

| Logic: Hidden by default |
|---|
| ID: 1169 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("10","11","12 or more") |
| Shortname / Alias: timetenth_dates |
| ID: 1057 |
| Please enter the dates you were off PrEP for the tenth time (from [question('value'), id='1026'] to today):* |
| Validation: %s format expected |
| ID: 1058 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1059 |
| Date re-started:*: |
| Logic: Hidden by default |
| ID: 1170 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a |

Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("11","12 or more")

Shortname / Alias: timeeleventh\_dates

Date re-started:\*:

ID: 1060

Please enter the dates you were off PrEP for the eleventh time (from [question('value'), id='1026'] to today):\*

Validation: %s format expected

| Date re-started:*: |
|---|
| Logic: Hidden by default |
| ID: 1171 |
| The date re-started is before the date stopped. Please correct this. |
| Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a |
| row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("12 or more") |
| Shortname / Alias: timetwelfth_dates |
| ID: 1063 |
| Please enter the dates you were off PrEP for the twelfth time (from [question('value'), id='1026'] to today):* |
| Validation: %s format expected |
| ID: 1064 |
| Date stopped:*: |
| Validation: %s format expected |
| ID: 1065 |
| Date re-started:*: |

**Page entry logic:** This page will show when: ((#37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes") OR (#29 Question "When you started the P3-T study, were you taking PrEP?" is one of the following answers ("Yes") AND #31 Question "Are you taking PrEP right now?" is one of the following answers ("No"))) OR (#30 Question "Did you start taking PrEP after you started the P3-T study?" is one of the following answers ("Yes") AND #31 Question "Are you taking PrEP right now?" is one of the following answers ("No")))

## **PrEP Stop**

Date stopped:\*:

ID: 1062

Validation: %s format expected

Logic: Hidden by default

This number cannot be greater than the number of times you stopped taking PrEP for 7 days in a row or more in the last 3 months ([question('value'), id='950']). Please correct this.

Validation: Must be numeric Whole numbers only Positive numbers only Logic: Hidden unless: #38 Question "How many times did you stop taking PrEP for 7 days in a row or more in the last three months (from [question('value'), id='1026'] to today)?" is one of the following answers ("1","2","3","4","5","6","7","8","9","10","11","12 or more") Shortname / Alias: prepstop\_drconsult ID: 578 Of the [question("value"), id="950"] times you stopped taking PrEP, how many did you talk with your medical provider about before you stopped taking PrEP?\* Shortname / Alias: stopprep why ID: 581 Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP.\* [] I couldn't afford it anymore [] I was not having sex [] I was no longer having sex with a person living with HIV [] I was only having sex with one person and they were undetectable or HIV negative [] I didn't want to keep taking a pill every day [] My parent(s) or guardian(s) found out and made me stop [] I kept forgetting to take my pill [ ] I haven't been able to make it to my follow-up appointments [] I could no longer see my PrEP provider and haven't found another PrEP provider [] I experienced side effects [] I was worried about the long term effects of PrEP on my health [] It was medically unsafe for me to continue taking PrEP (due to kidney/renal function, bone density, or another medical issue) [] I was worried that if I were to become HIV-positive certain medications may no longer work or I might be resistant to them [] I was worried that PrEP might not provide complete protection against HIV [] I started using condoms all of the time

[] The medication tastes bad and/or the pill is too big

[] Other, please specify:: \_\_\_\_\_

**Page entry logic:** This page will show when: #38 Question "How many times did you <u>stop taking PrEP for 7 days in a row or more</u> in the last three months (*from [question('value'), id='1026'] to today)?*" is one of the following answers ("1","2","3","4","5","6","7","8","9","10","11")

Action: Custom Script: Script to check number of times off PrEP

**Page entry logic:** This page will show when: #53 Question "Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP."

### **PrEP Stop Continued**

Action: Custom Script: Script to count checkboxes and skip if q <2

Shortname / Alias: stopprep primwhy

ID: 582

Piping: Piped Values From Question 53. (Think about the most recent time you stopped taking PrEP. Select all of the factors below that were related to why you stopped PrEP.)

Please rank the reasons you stopped taking PrEP in order of importance.\*

**Page entry logic:** This page will show when: #37 Question "Have you stopped taking PrEP for 7 days in a row or more in the last 3 months?" is one of the following answers ("Yes")

#### PrEP Restart, current users

Shortname / Alias: restart why

| Why did you choose to restart taking PrEP the last time? Select all that ap |
|-----------------------------------------------------------------------------|
|-----------------------------------------------------------------------------|

- [] I was able to start seeing my PrEP provider again
- [] I found a new PrEP provider
- [] I was having issues with side effects, but I found a way to deal with them
- [] I was having issues taking my pill every day, but I found a way to deal with it
- [] I'm having sex with or thinking about having sex with someone who is HIV+
- [] I'm having sex with or thinking having sex with someone whose status HIV I don't know
- [] I want to be in control of my sexual health
- [] I want to reduce my anxiety around sex

| [] I want to increase my sexual satisfaction and intimacy |
|---|
| [] I want to be safe and healthy |
| [] I want to have a better future |
| [] I am having sex with multiple partners |
| [] I don't like to use condoms |
| [] My partner won't use condoms |
| [] I had a previous HIV scare |
| [] My health care provider recommended it |
| [] I was recently diagnosed with an STI |
| [] Many people in my community take PrEP |
| [] Other, please specify:: |
| <b>Page entry logic:</b> This page will show when: #55 Question "Why did you choose to restart taking PrEP the last time? Select all that apply." |
| Restart reason, current users |
| Action: Custom Script: Script to count checkboxes and skip if q <2 |
| Shortname / Alias: restart_primwhy |

ID: 957

Piping: Piped Values From Question 55. (Why did you choose to restart taking PrEP the last time?

Select all that apply.)

What was the main reason you decided to restart PrEP?\*

## **Healthcare Visits**

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Show/hide trigger exists.

Shortname / Alias: numdrvisits3m

ID: 584

In the last 3 months, how many times did you go to the doctor for any reason?\*

\_\_\_\_\_\_

Logic: Hidden by default

ID: 940

This number cannot be greater than the total number of doctor's visits entered above.

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Show/hide trigger exists. Hidden unless: #57 Question "In the last 3 months, how many times did you go to the doctor for any reason?" is greater than "0"

Shortname / Alias: numprepvisits3m

ID: 586

Out of all these visits, how many were routine/scheduled PrEP appointments?\*

Logic: Hidden by default

ID: 988

This number cannot be greater than the total number of routine PrEP appointments.

Validation: Must be numeric Whole numbers only Positive numbers only

Logic: Hidden unless: #58 Question "Out of all these visits, how many were routine/scheduled PrEP appointments?" is greater than "0"

Shortname / Alias: missedprepvisits3m

ID: 587

In the last 3 months, how many of your scheduled PrEP appointments did you miss because you didn't show or forgot?

By scheduled appointments, we mean routine PrEP appointments, not walk-in or urgent care appointments for acute/urgent issues. \*

Action: Custom Script: Script to check number of visits

Action: Custom Script: Script to check number of days

| Logic: Hidden unless: #31 Question "Are you taking PrEP right now?" is one of the following answers ("Yes") |
|---|
| Shortname / Alias: preplastweek |
| ID: 177 |
| How many of the last 7 days did you take your PrEP medication?* () 0 days |
| ( ) 1 day |
| ( ) 2 days |
| ( ) 3 days |
| ( ) 4 days |
| ( ) 5 days |
| () 6 days |
| ( ) 7 days |
| Validation: Min = 0 Max = 100 |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: prepmonth |
| ID: 178 |
| In the last month, what percent of the time did you take your PrEP as prescribed (once a day)? Use the scale below. 0% would mean 'NONE' of the time and 100% would mean 'ALL' of the time. If you are unsure, make a guess. |
| % medication taken:* |
| 0 100 |
| PrEP Dose Barriers |
| Shortname / Alias: dose_ |
| ID: 959 |
| What has gotten in the way of you taking your PrEP on a daily basis? Please select all that apply.* [] I have not had any trouble taking PrEP on a daily basis |
| [] I get tired of taking a pill every day |
| [] I forget to take it |
| [] I don't always have my pills with me |
| [] My work/school schedule |

| [] My social life [] I'm around people I don't want to take it in front of [] I experience side effects [] I was drinking or using drugs and I didn't take it |
|---|
| Action: Custom Script: Script to count checkboxes and skip if q <2 |
| Shortname / Alias: does_rank |
| ID: 960 |
| Piping: Piped Values From Question 62. (What has gotten in the way of you taking your PrEP on a daily basis? Please select all that apply.) |
| Please rank the things that have gotten in the way of you taking your PrEP on a daily basis.* |
| PrEP Adherence Continued |
| Logic: Hidden unless: #61 Question "In the last month, what percent of the time did you take your PrEP as prescribed (once a day)? Use the scale below. 0% would mean 'NONE' of the time and 100% would mean 'ALL' of the time. If you are unsure, make a guess. |
| % medication taken:" |
| Shortname / Alias: prepadher_protection |
| ID: 588 |
| You said you took your PrEP [question("value"), id="178"] percent of the time in the last month. Based on this adherence level, how protected do you think you were from HIV in the last month?* () Not protected at all |
| ( ) Somewhat protected |

- () Mostly protected
- () Fully protected

Shortname / Alias: prepadher\_decisionbot

ID: 589

In the last month, how much did your adherence to PrEP (if you took it every day or not) affect how often you used a condom during anal sex when you bottom?\*

( ) My decision about condom use when I bottom was not influenced by whether or not I took my pill every day

| ( ) My decision about condom use when I bottom <u>was somewh</u> pill every day | at influenced by whether or not I took my |
|---|---|
| ( ) My decision about condom use when I bottom <u>was</u> influence day | ed by whether or not I took my pill every |
| ( ) I did not bottom in the last month | |
| () | |
| Shortname / Alias: prepadher_decisiontop | |
| ID: 590 | |
| In the last month, how much did your adherence to PrEP (in how often you used a condom during anal sex when you to ( ) My decision about condom use when I top was not influence day | op?* |
| ( ) My decision about condom use when I top <u>was somewhat</u> in every day | nfluenced by whether or not I took my pill |
| ( ) My decision about condom use when I top <u>was</u> influenced b | y whether or not I took my pill every day |
| ( ) I did not top in the last month | |
| PrEP Confidence | |
| ID: 907 | |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). | |
| We are interested in how you feel about the following indicating your confidence about each statement on a | |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). | |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). Validation: Min = 1 Max = 10 | |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: keepappts | |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: keepappts ID: 903 How confident are you that you can Keep your PrEP medical appointments:* | a scale from 1 (not confident) to 10 |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: keepappts ID: 903 How confident are you that you can | a scale from 1 (not confident) to 10 |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: keepappts ID: 903 How confident are you that you can Keep your PrEP medical appointments:* | a scale from 1 (not confident) to 10 |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: keepappts ID: 903 How confident are you that you can Keep your PrEP medical appointments:* 1 | a scale from 1 (not confident) to 10 |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: keepappts ID: 903 How confident are you that you can Keep your PrEP medical appointments:* 1 [ ] Validation: Min = 1 Max = 10 Shortname / Alias: followplan | a scale from 1 (not confident) to 10 |
| We are interested in how you feel about the following indicating your confidence about each statement on a (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: keepappts ID: 903 How confident are you that you can Keep your PrEP medical appointments:* 1 | a scale from 1 (not confident) to 10 |

| Validation: Min = 1 Max = 10 | |
|---|---|
| Shortname / Alias: atworkschool | |
| ID: 905 | |
| Take PrEP at work/school:* | |
| 1 10 | |
| Validation: Min = 1 Max = 10 | |
| Shortname / Alias: onweekday | |
| ID: 906 | |
| Take PrEP on a weekday:* | |
| 110 | |
| PrEP Confidence 2 | _ |
| ID: 908 | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: onweekend | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: onweekend ID: 909 How confident are you that you can | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: onweekend ID: 909 | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: onweekend ID: 909 How confident are you that you can Take PrEP on a weekend:* | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: onweekend ID: 909 How confident are you that you can Take PrEP on a weekend:* | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: onweekend ID: 909 How confident are you that you can Take PrEP on a weekend:* | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: onweekend ID: 909 How confident are you that you can Take PrEP on a weekend:* 1 | |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: onweekend ID: 909 How confident are you that you can Take PrEP on a weekend:* 1 | |

| Validation: Min = 1 Max = 10 Shortname / Alias: prepdrinking ID: 911 |
|---|
| Take PrEP when I'm drinking or using drugs:* 1 10 |
| Validation: Min = 1 Max = 10 |
| Shortname / Alias: schedulechange ID: 912 |
| Take PrEP when my schedule changes:* 1 10 |
| PrEP Confidence 3 |
| ID: 913 |
| We are interested in how you feel about the following statements. Please answer by indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). |
| indicating your confidence about each statement on a scale from 1 (not confident) to 10 |
| indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). |
| indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: whiletraveling |
| indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: whiletraveling ID: 914 |
| indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: whiletraveling ID: 914 How confident are you that you can Take PrEP while traveling:* |
| indicating your confidence about each statement on a scale from 1 (not confident) to 10 (totally confident). Validation: Min = 1 Max = 10 Shortname / Alias: whiletraveling ID: 914 How confident are you that you can Take PrEP while traveling:* 1 |

| Validation: Min = 1 Max = 10 |
|---------------------------------|
| Shortname / Alias: havingcrisis |

ID: 916

| Take PrEP when you are having a crisis:* |
|------------------------------------------|
|------------------------------------------|

| 1 | 1 | 1 | 10 | ) |
|---|---|---|----|---|

## **PrEP Delivery**

Shortname / Alias: prep\_prefmode

ID: 597

Right now there are no other approved options for taking PrEP. However, if there were more than one option and each method was equally good at protecting you from getting HIV, which method would you most prefer?\*

- () Taking one pill, every day
- () Taking two pills before you had sex and a pill a day for the next two days
- ( ) Taking one pill a day just on Tuesday, Thursday, Saturday, and Sunday
- () Getting an injection about every 2 to 3 months
- ( ) Putting medicated lubrication (lube) in your anus (and/or your partner's anus) before having anal sex
- ( ) Douching with a medicated solution (microbicide) before having anal sex

#### **PrEP Beliefs**

Shortname / Alias: prepbeliefs

ID: 598

Please rate your agreement with the following statements:\*

| Tiouso rate ye | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| People are<br>less likely<br>to use<br>condoms<br>for anal sex<br>if they are<br>using PrEP | () | () | () | () |
| I feel as if<br>starting to<br>take PrEP | () | () | () | () |

| would allow<br>me to have<br>more sex<br>partners | | | | |
|---|---|---|---|---|
| I feel as if<br>starting to<br>take PrEP<br>would allow<br>me to have<br>more<br>condomless<br>anal sex | () | () | () | () |

## **PrEP and People**

Shortname / Alias: prepppl

ID: 193

We are interested in how you feel about the following statements. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I worry people will assume I sleep around if they know I take PrEP | () | () | () | () |
| I worry people will assume that I am HIV- positive if they know I take PrEP | () | () | () | () |
| I worry people will think my partner(s) are HIV- positive if | () | () | () | () |

| they know I | | | | |
|---|---|---|---|---|
| take PrEP | | | | |
| I worry about listing PrEP as one of my current medications during appointments such as at a dentist's or specialist's office | () | () | () | () |
| I feel<br>ashamed to<br>tell other<br>people that I<br>am taking<br>PrEP | () | () | () | () |
| I worry people will think I am a bad person if they know I take PrEP | () | () | () | () |
| I worry people will think I am gay if they know I take PrEP | () | () | () | () |
| I worry my<br>friends will<br>find out that I<br>take PrEP | () | () | () | () |
| I worry my<br>family will<br>find out that I<br>take PrEP | () | () | () | () |
| I worry my<br>sexual<br>partners will<br>find out that I<br>take PrEP | () | () | () | () |
| I think people<br>will give me a<br>hard time if I<br>tell them I<br>take PrEP | () | () | () | () |
|---|---|---|---|---|
| I think people<br>will judge me<br>if they know I<br>am taking<br>PrEP | () | () | () | () |

### **PrEP Concerns**

Shortname / Alias: prepconc

ID: 210

We are interested in how you feel about the following statements. Read each statement carefully and indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| My family<br>does not<br>support me<br>taking PrEP | () | () | () | () |
| My friends<br>do not<br>support me<br>taking PrEP | () | () | () | () |
| People<br>taking PrEP<br>are<br>portrayed<br>poorly in the<br>media and<br>online | () | () | () | () |
| People in my<br>community<br>talk poorly<br>about people<br>taking PrEP | () | () | () | () |

| I feel<br>embarrassed<br>about taking<br>PrEP | () | () | () | () |
|---|---|---|---|---|
| I think I am<br>not following<br>the 'rules' of<br>my<br>community if<br>I take PrEP | () | () | () | () |
| I have been blamed by people in my community for spreading HIV through PrEP use | () | () | () | () |
| I have been blamed by people in my community for spreading sexually transmitted infections through not using condoms | () | () | () | () |
| I have been rejected romantically because I take PrEP | () | () | () | () |
| I have been slut-shamed because I take PrEP (or told that I am a "Truvada-slut/whore") | () | () | () | () |
| I have been judged by a health care provider for taking PrEP | () | () | () | () |

| | | | | <u>.</u> |
|---|---|---|---|---|
| I don't think<br>that I need to<br>take PrEP<br>anymore | () | () | () | () |
| I have been told by a health care provider that I don't need PrEP or I shouldn't take PrEP | () | () | () | () |
| I have been<br>yelled at or<br>scolded<br>because I<br>take PrEP | () | () | () | () |
| I have been unfairly discriminated against because I take PrEP | () | () | () | () |
| I have<br>experienced<br>physical<br>violence<br>because I<br>am taking<br>PrEP | () | () | () | () |

Logic: Hidden unless: Question "I don't think that I need to take PrEP anymore" is one of the following answers ("Agree","Strongly Agree")

Shortname / Alias: whydontneed

ID: 1067

| Why do you think that you do not need to take PrEP anymore? Select all that apply.* [] My relationship status changed I became single |
|---|
| [] My relationship status changed I became monogamous (only having sex with one person) |
| [] I stopped having sex with an HIV-positive person |
| [] I am having less sex |
| [] I am sexually inactive (I haven't been having sex for a period of time) |
| [] I have started using condoms every time I have sex |
| [] Other, please specify:: |

### **PrEP Difficulties**

Shortname / Alias: prepdifficulties

ID: 602

In making your decision to continue taking PrEP, please rate how much the following items

concern you.\*

| | Not at all concerned | A little concerned | Concerned | Very<br>concerned |
|---|---|---|---|---|
| Getting the costs of PrEP covered (including office visits or office visit copays, lab costs, transportation costs) | () | () | () | () |
| Using insurance to get coverage for PrEP costs (including office visits, lab costs) | () | () | () | () |
| Getting<br>transportation<br>to PrEP<br>appointments<br>and labs | () | () | () | () |
| Returning for PrEP follow-<br>up appointments and labs | () | () | () | () |
| Getting PrEP prescription refilled | () | () | () | () |

### **PrEP Difficulties Continued**

Shortname / Alias: prepdifficulties2

ID: 649

In making your decision to continue taking PrEP, please rate how much the following items

concern you.\*

| | Not at all concerned | A little concerned | Concerned | Very<br>concerned |
|---|---|---|---|---|
| The possibility that if I were to become HIV+, certain medications might no longer work or I might be resistant to them | () | () | () | () |
| The possibility that PrEP might not provide complete protection against HIV | () | () | () | () |
| Having to talk to a health care provider about PrEP | () | () | () | () |
| Having to talk to a health care provider about my sex life | () | () | () | () |
| Experiencing side effects from PrEP | () | () | () | () |
| The long-<br>term effects | () | () | () | () |

| of PrEP on<br>my health | | | | |
|----------------------------------------------------------|----|----|----|----|
| Having to<br>remember to<br>take PrEP<br>every day | () | () | () | () |
| Friends<br>finding out<br>that I am on<br>PrEP | () | () | () | () |
| Family<br>members<br>finding out<br>that I am on<br>PrEP | () | () | () | () |
| Sexual partners finding out that I am on PrEP | () | () | () | () |

Logic: Hidden unless: Question "The possibility that PrEP might not provide complete protection against HIV" is one of the following answers ("Concerned", "Very concerned")

Shortname / Alias: prepworry

ID: 665

# Why do you worry about the possibility that PrEP might not provide complete protection against HIV? (Check all that apply)\*

- [] I worry that the drug is not effective at preventing HIV
- [] Because I don't take PrEP every day consistently
- [] Because I feel I am at very high risk for becoming infected with HIV
- [] Other, please specify::

### **HIV** perceptions

Shortname / Alias: hivthoughts

ID: 667

Imagine how you would feel if you became infected with HIV. Read each statement carefully and

indicate how strongly you agree or disagree with the following statements.\*

| | Strongly<br>Disagree | Disagree | Agree | Strongly<br>Agree |
|---|---|---|---|---|
| I would<br>be afraid<br>people<br>would<br>judge me<br>when<br>they<br>learn I<br>have HIV | () | () | () | () |
| If I got infected, people would not want to have sex with me | () | () | () | () |
| I would<br>feel<br>guilty if I<br>got HIV | () | () | () | () |
| I would<br>feel<br>ashamed<br>if I got<br>HIV | () | () | () | () |

### PEP and PrEP On-Demand

Shortname / Alias: pep3m

ID: 230

In the past 3 months, have you taken post-exposure prophylaxis (PEP) <u>AFTER</u> a sexual or drug use exposure to reduce the risk of getting HIV?\*

() Yes

() No

| Shortname / Alias: prepondemand3m<br>ID: 674 |
|---|
| In the past 3 months, have you taken PrEP on-demand (taking two pills before you had sex and a pill a day for the next two days)? It is not an approved method and has not been shown to be an effective method for preventing HIV.* () Yes () No |
| Substances |
| ID: 232 |
| Now we'd like to ask you a little bit about your experiences using alcohol, tobacco products, and other drugs. Please be assured that this information will be treated as <i>strictly confidential</i> . The questions will concern your experiences with using these substances in the past three months. These substances can be smoked, swallowed, snorted, inhaled, injected, or taken in the form of pills. Some of the substances may be prescribed by a doctor (like amphetamines, sedatives, or pain medications). For this survey, do not report on medications that are used as prescribed by your doctor. However, if you have taken such medications for reasons other than prescription, or taken them more frequently or at higher doses than prescribed, please report on this use. Once again, please remember that all information provided will be treated as <i>strictly confidential</i> . |
| Shortname / Alias: substanceuse3m |
| ID: 233 |
| Which of the following drugs have you used in the last 3 months? Please check all that apply.* [] Tobacco (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) [] Alcohol (beer, wine, spirits, etc.) |
| [] Cannabis (marijuana, pot, weed, grass, hash, synthetic cannabis, etc.) |
| [] Cocaine (coke, crack, etc.) |

Which of the following drugs have you used in the last 3 months?

Please check all that apply.\*

[] Tobacco (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)

[] Alcohol (beer, wine, spirits, etc.)

[] Cannabis (marijuana, pot, weed, grass, hash, synthetic cannabis, etc.)

[] Cocaine (coke, crack, etc.)

[] Amphetamines (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)

[] Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)

[] Sedatives, tranquilizers, or sleeping pills (valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)

[] Hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)

[] Opioids (heroin, morphine, methadone, codeine, Oxycotin, Percocet, Vicodin, etc.)

[] None of these

**Page entry logic:** This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

Please check all that apply." is one of the following answers ("Tobacco (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)")

### **Tobacco**

| Shortname / Alias: tobacco3months |
|---|
| ID: 234 |
| In the past 3 months, how often have you used tobacco products (cigarettes, chewing tobacco cigars, e-cigarettes, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccodesire |
| ID: 235 |
| During the past 3 months, how often have you had a desire to use tobacco products (cigarettes chewing tobacco, cigars, e-cigarettes, etc.)?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccoproblems |
| ID: 236 |
| During the past 3 months, how often has your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.) led to health, social, legal or financial problems?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: tobaccofriend |
| ID: 238 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () No |
| () Yes |
| Shortname / Alias: tobaccostop |
| ID: 239 |
| In the last 3 months, have you tried and failed to control, cut down or stop using tobacco products (cigarettes, chewing tobacco, cigars, e-cigarettes, etc.)?* () No |
| () Yes |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? |
| Please check all that apply." is one of the following answers ("Alcohol (beer, wine, spirits, etc.)") |
| Alcohol |

In the past 3 months, how often have you used alcoholic beverages (beer, wine, spirits, etc.)?\*

Shortname / Alias: tobaccofailed

Logic: Show/hide trigger exists.

Shortname / Alias: alcohol3months

ID: 240

() Never

ID: 237

334

| ( ) Once or twice |
|---|
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Logic: Hidden unless: #97 Question "In the past 3 months, how often have you used alcoholic beverages (beer, wine, spirits, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily","Decline to answer") |
| Shortname / Alias: alcoholdaily |
| ID: 241 |
| How many drinks containing alcohol do you have on a typical day?* |
| () 1 or 2 |
| () 3 or 4 |
| () 5 or 6 |
| () 7 to 9 |
| ( ) 10 or more |
| Shortname / Alias: alcoholbinge |
| Shortname / Alias: alcoholbinge ID: 242 |
| ID: 242 How often do you have 5 or more drinks on one occasion?* |
| How often do you have 5 or more drinks on one occasion?* ( ) Never |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: alcoholdesire |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: alcoholdesire ID: 243 During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: alcoholdesire ID: 243 During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: alcoholdesire ID: 243 During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice |
| How often do you have 5 or more drinks on one occasion?* ( ) Never ( ) Less than monthly ( ) Monthly ( ) Weekly ( ) Daily or almost daily Shortname / Alias: alcoholdesire ID: 243 During the past 3 months, how often have you had a desire to use alcoholic beverages (beer, wine, spirits, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly |

| Shortname / Alias: alcoholproblems ID: 244 |
|---|
| During the past 3 months, how often has your use of alcoholic beverages (beer, wine, spirits, etc.) led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholfailed |
| ID: 245 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of alcoholic beverages (beer, wine, spirits, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: alcoholfriend |
| ID: 246 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of alcoholic beverages (beer, wine, spirits, etc.)?* |
| () Yes |
| Shortname / Alias: alcoholstop |
| ID: 247 |
| In the last 3 months, have you tried and failed to control, cut down or stop using alcoholic beverages (beer, wine, spirits, etc.)?* ( ) No |
| () Yes |
| Action: JavaScript: Hide General Error Message |

**Page entry logic:** This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months?

*Please check all that apply.*" is one of the following answers ("Cannabis (marijuana, pot, weed, grass, hash, synthetic cannabis, etc.)")

### **Cannabis**

Shortname / Alias: cannabisproblems

ID: 253

| Shortname / Alias: cannabis3months |
|---|
| ID: 251 |
| In the past 3 months, how often have you used cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Page entry logic: This page will show when: #107 Question "In the past 3 months, how often have you used cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?" is one of the following answer ("Once or twice", "Monthly", "Weekly", "Daily or almost daily") |
| Cannabis (cont.) |
| Shortname / Alias: cannabisdesire |
| ID: 252 |
| During the past 3 months, how often have you had a desire to use cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |

| During the past 3 months, how often has your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis led to health, social, legal or financial problems?* ( ) Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisfailed |
| ID: 254 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cannabisfriend |
| ID: 255 |
| In the past 3 months, has a friend or relative or anyone else expressed concern about your use of cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* |
| ()Yes |
| Shortname / Alias: cannabisstop |
| ID: 256 |
| In the last 3 months, have you tried and failed to control, cut down or stop using cannabis (marijuana, pot, grass, hash, etc.) or synthetic cannabis?* |
| ()Yes |
| <b>Page entry logic:</b> This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? Please check all that apply." is one of the following answers ("Cocaine (coke, crack, etc.)") |

# Cocaine

| Shortname / Alias: cocaine3months |
|---|
| ID: 257 |
| In the past 3 months, how often have you used cocaine (coke, crack, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |
| Page entry logic: This page will show when: #113 Question "In the past 3 months, how often have you used cocaine (coke, crack, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Cocaine (cont.) |
| Shortname / Alias: cocainedesire |
| ID: 258 |
| During the past 3 months, how often have you had a desire to use cocaine (coke, crack, etc.)?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: cocaineproblems |
| ID: 259 |
| During the past 3 months, how often has your use of cocaine (coke, crack, etc.) led to health, social, legal or financial problems?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |

| () Weekly |
|---|
| ( ) Daily or almost daily |
| Shortname / Alias: cocainefriend |
| ID: 261 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of cocaine (coke, crack, etc.)?* ( ) No |
| () Yes |
| Shortname / Alias: cocainestop |
| ID: 262 |
| In the last 3 months, have you tried and failed to control, cut down or stop using cocaine (coke, crack, etc.)?* ( ) No |
| () Yes |
| De constant la colon This was a still all a constant #00 Occasion WA/Isiah af the fall a citizen decomposition |
| <b>Page entry logic:</b> This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? |
| Please check all that apply." is one of the following answers ("Amphetamines (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)") |
| Amphotomino |
| Amphetamine |

In the past 3 months, how often have you used amphetamine type stimulants (speed, meth, diet

During the past 3 months, how often have you failed to do what was normally expected of you

Shortname / Alias: cocainefailed

because of your use of cocaine (coke, crack, etc.)?\*

Shortname / Alias: amphetamine3months

pills, ecstasy, Ritalin, Adderall, etc.)?\*

ID: 263

() Never

ID: 260

() Never

() Monthly

() Once or twice

| ( ) Once or twice |
|---|
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |
| December 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| <b>Page entry logic:</b> This page will show when: #119 Question "In the past 3 months, how often have you used amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Amphetamine (cont.) |
| Shortname / Alias: amphetaminedesire |
| ID: 265 |
| During the past 3 months, how often have you had a desire to use amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetamineproblems |
| ID: 266 |
| During the past 3 months, how often has your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.) led to health, social, legal or financial problems?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetaminefailed |
| ID: 267 |

| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* () Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: amphetaminefriend |
| ID: 268 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* () No |
| () Yes |
| Shortname / Alias: amphetaminestop |
| ID: 269 |
| In the last 3 months, have you tried and failed to control, cut down or stop using amphetamine type stimulants (speed, meth, diet pills, ecstasy, Ritalin, Adderall, etc.)?* |
| () Yes |
| Action: JavaScript: Hide General Error Message |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used in the last 2 months? |
| in the last 3 months? Please check all that apply." is one of the following answers ("Inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)") |
| Inhalants |

Shortname / Alias: inhalants3months

In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?\*

() Never

| ( ) Once or twice |
|---|
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |
| <b>Page entry logic:</b> This page will show when: #125 Question "In the past 3 months, how often have you used inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Inhalants (cont.) |
| Shortname / Alias: inhalantsdesire |
| ID: 272 |
| During the past 3 months, how often have you had a desire to use inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsproblems |
| ID: 273 |
| During the past 3 months, how often has your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.) led to health, social, legal or financial problems?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: inhalantsfailed |
| ID: 274 |

| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) Never ( ) Once or twice ( ) Monthly ( ) Weekly ( ) Daily or almost daily |
|---|
| Shortname / Alias: inhalantsfriend ID: 275 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) No ( ) Yes |
| Shortname / Alias: inhalantsstop<br>ID: 276 |
| In the last 3 months, have you tried and failed to control, cut down or stop using inhalants (poppers, nitrous, glue, petrol, paint thinner, etc.)?* ( ) No ( ) Yes Action: JavaScript: Hide General Error Message |
| <b>Page entry logic:</b> This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? Please check all that apply." is one of the following answers ("Sedatives, tranquilizers, or sleeping pills (valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)") |

### **Sedatives**

Shortname / Alias: sedatives3months

ID: 277

In the past 3 months, how often have you used sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?\*

() Never

| ( ) Once or twice |
|---|
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |
| Alone Cavaceriph rings Conoral Error mossage |
| <b>Page entry logic:</b> This page will show when: #131 Question "In the past 3 months, how often have you used sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)? is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Sedatives (cont.) |
| Shortname / Alias: sedativesdesire |
| ID: 279 |
| During the past 3 months, how often have you had a desire to use sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: sedativesproblems |
| ID: 280 |
| During the past 3 months, how often has your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.) led to health, social, legal or financial problems?* () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: sedativesfailed |
| ID: 281 |

| () Never |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: sedativesfriend |
| ID: 282 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* () No |
| () Yes |
| Shortname / Alias: sedativesstop |
| ID: 283 |
| In the last 3 months, have you tried and failed to control, cut down or stop using sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol, Xanax, Ambien, GHB, etc.)?* |
| () Yes |
| Page entry logic: This page will show when: #90 Question "Which of the following drugs have you used |
| in the last 3 months? |
| Please check all that apply." is one of the following answers ("Hallucinogens (LSD, acid, mushrooms, |
| PCP, Ketamine, etc.)") |
| Hallucinogens |
| Shortname / Alias: hallucinogens3months |
| ID: 285 |
| In the past 3 months, how often have you used hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| 246 |

During the past 3 months, how often have you failed to do what was normally expected of you because of your use of sedatives, tranquilizers, or sleeping pills (Valium, Serepax, Rohypnol,

Xanax, Ambien, GHB, etc.)?\*

| () Weekly |
|---|
| ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |
| Action duragon par mad Condital Error modelage |
| <b>Page entry logic:</b> This page will show when: #137 Question "In the past 3 months, how often have you used hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Hallucinogens (cont.) |
| Trandemogens (cont.) |
| Shortname / Alias: hallucinogensdesire |
| ID: 286 |
| During the past 3 months, how often have you had a desire to use hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensproblems |
| ID: 287 |
| During the past 3 months, how often has your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.) led to health, social, legal or financial problems?* ( ) Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensfailed |
| ID: 288 |

| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* |
|---|
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: hallucinogensfriend |
| ID: 289 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* ( ) No |
| () Yes |
| Shortname / Alias: hallucinogensstop |
| ID: 290 |
| In the last 3 months, have you tried and failed to control, cut down or stop using hallucinogens (LSD, acid, mushrooms, PCP, Ketamine, etc.)?* |
| () Yes |
| Action: JavaScript: Hide General Error Message |
| <b>Page entry logic:</b> This page will show when: #90 Question "Which of the following drugs have you used in the last 3 months? Please check all that apply." is one of the following answers ("Opioids (heroin, morphine, methadone, codeine, Oxycotin, Percocet, Vicodin, etc.)") |

## **Opioids**

Shortname / Alias: opioids3months

ID: 291

In the past 3 months, how often have you used opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?\*

- () Never
- () Once or twice

| ( ) Monthly |
|---|
| () Weekly |
| ( ) Daily or almost daily |
| Action: JavaScript: Hide General Error Message |
| Page entry logic: This page will show when: #143 Question "In the past 3 months, how often have you |
| used opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?" is one of the following answers ("Once or twice","Monthly","Weekly","Daily or almost daily") |
| Tollowing answers ( Office of twice , Worlding , Weekly , Daily of annost daily ) |
| Opioids (cont.) |
| Logic: Show/hide trigger exists. |
| Shortname / Alias: opioidsheroin |
| ID: 299 |
| In the past 2 months, has your enjoid use included havein?* |
| In the past 3 months, has your opioid use included heroin?* ( ) Yes |
| ( ) No |
| Logic: Hidden unless: #144 Question "In the past 3 months, has your opioid use included |
| heroin?" is one of the following answers ("Yes") |
| Shortname / Alias: heroinprimary |
| ID: 300 |
| In the past 3 months, was heroin the most common opioid that you used?* ( ) Yes |
| ( ) No |
| ()110 |
| Shortname / Alias: opioidssdesire |
| ID: 293 |
| During the past 3 months, how often have you had a desire to use opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* |
| () Never |
| () Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| 27 |

| ID: 294 |
|---|
| During the past 3 months, how often has your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.) led to health, social, legal or financial problems?* () Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: opioidsfailed |
| ID: 295 |
| During the past 3 months, how often have you failed to do what was normally expected of you because of your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) Never |
| ( ) Once or twice |
| ( ) Monthly |
| () Weekly |
| ( ) Daily or almost daily |
| Shortname / Alias: opioidsfriend |
| ID: 296 |
| In the last 3 months, has a friend or relative or anyone else expressed concern about your use of opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* () No |
| () Yes |
| Shortname / Alias: opioidsstop ID: 297 |
| In the last 3 months, have you tried and failed to control, cut down or stop using opioids (heroin, morphine, methadone, codeine, Oxycontin, Percocet, Vicodin, etc.)?* ( ) No ( ) Yes |

Shortname / Alias: opioidsproblems

### **Sexual Behaviors**

Action: JavaScript: Hide General Error Message

**Page exit logic:** Skip / Disqualify Logic**IF:** #151 Question "In the past 3 months, how many people have you had anal sex with?" is exactly equal to "0" **THEN:** Jump to page 120 - Perceived HIV Risk

ID: 368

The next section of questions will ask about your sexual behaviors. We know that this can be a sensitive topic, so we would like to remind you that your answers will be kept completely confidential. Please be as honest as possible in order to ensure the success of the current study.

The following questions refer to your sexual behavior during the past 3 months. Our focus will be only on anal sex. Therefore, do not include references to people with whom you did not engage in anal sex.

For these questions, anal sex refers to sex where the other person's penis was in your rectum (you were the bottom) and to sex where your penis was in the other person's rectum (you were the top).

These questions only ask about people assigned male at birth, which includes cisgender men (men assigned male at birth) and transgender women (women assigned male at birth). Therefore, do not include references to cisgender women (women assigned female at birth) or transgender men (men assigned female at birth).

Validation: Min = 0 Max = 999 Must be numeric Whole numbers only Positive numbers only

Shortname / Alias: numsexpartner

ID: 302

In the past 3 months, how many people have you had anal sex with?\*

\_\_\_\_\_\_

Action: JavaScript: Hide General Error Message

**Page entry logic:** This page will show when: #151 Question "In the past 3 months, how many people have you had anal sex with?" is greater than "0"

### **HIV Status of Sexual Partners**

| Logic: Hidden by default |
|---|
| ID: 677 |
| The total number must equal the number of people you had anal sex with in the last 3 months ([question('value'), id='302']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: partnerhivstatus |
| ID: 676 |
| Before you had sex, what did you know of the HIV status of your sexual partner(s)? |
| Enter numerical values. Numbers must add up to [question('value'), id='302'], the number of people you reported having anal sex within the last three months.* This person/these people told you they were HIV negative and you had no reason to doubt it |
| You knew this person/these people were HIV positive |
| You were not completely sure of this person/these people's HIV status |
| Action: Custom Script: Script to check the continuous sum totals |
| Hidden Value: Num HIV Neg partners |
| Value: [question("option value"), id="676", option="12278"] |
| Hidden Value: Num HIV Pos partners |
| Value: [question("option value"), id="676", option="12279"] |
| Hidden Value: Num HIV Unk partners |

Value: [question("option value"), id="676", option="12280"]

Page entry logic: This page will show when: Num HIV Neg partners is greater than "0"

### **HIV Negative Partners**

ID: 690

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Shortname / Alias: hivneg\_timesbot

ID: 701

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom?\*

\_\_\_\_\_

Shortname / Alias: hivneg\_timestop

ID: 702

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the top?\*

**Page entry logic:** This page will show when: #153 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative <a href="where you were the bottom">where you were the bottom</a>?" is greater than "0"

### **HIV Negative Partners - Condomless Receptive AI**

Logic: Hidden by default

ID: 714

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='701']). Please correct this.

Shortname / Alias: hivneg timesbotunp

| In the past 3 months, how many of the [question('value'), id='701'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom were without a condom? * ——————————————————————————————————— |
|---|
| Action: Custom Script: Check number condomless is not greater than total times |
| <b>Page entry logic:</b> This page will show when: #155 Question "In the past 3 months, how many of the [question('value'), id='701'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the bottom were without a condom? " is greater than "0" |
| HIV Negative Partners - Condomless Receptive Al |
| ID: 721 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative |
| Logic: Hidden by default |
| ID: 999 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivneg_botunp_typ |
| ID: 711 |
| Regarding the partners who told you they were HIV negative who you had <u>condomless receptive</u> <u>anal sex with (where you were the bottom)</u> , how many were |
| Enter numerical values.* Romantic partner(s), someone you are in a relationship with |

\_Casual hook-up(s) or one-night stand(s)

ID: 710

| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |
|---|
| Logic: Hidden by default |
| ID: 1002 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivneg_botunp_gender |
| ID: 964 |
| How many were |
| Enter numerical values.* Men Transwomen Non-binary, genderqueer, or gender non-conforming Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| <b>Page entry logic:</b> This page will show when: #154 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV negative where you were the top?" is greater than "0" |
| HIV Negative Partners - Condomless Insertive Al |
| ID: 722 |

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 719

This number cannot be greater than the number of times you had anal sex where you were the top ([question('value'), id='702']). Please correct this.

Shortname / Alias: hivneg timestopunp

ID: 718

In the past 3 months, how many of the [question('value'), id='702'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the top were without a condom? \*

Action: Custom Script: Script to check number condomless is not greater than the totals

**Page entry logic:** This page will show when: #158 Question "In the past 3 months, how many of the [question('value'), id='702'] times you had anal sex with sexual partner(s) who told you they were HIV negative where you were the top were without a condom?" is greater than "0"

**HIV Negative Partners - Condomless Insertive AI** 

ID: 723

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 1004

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivneg topunp typ |
| ID: 725 |
| Regarding the partners who told you they were HIV negative who you had <u>condomless insertive</u> anal sex with (where you were the top), how many were |
| Enter numerical values.*Romantic partner(s), someone you are in a relationship with |
| Casual hook-up(s) or one-night stand(s) |
| A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |
| Logic: Hidden by default |
| ID: 1005 |
| option='12278']). Please correct this. Validation: Must be numeric |
| Shortname / Alias: hivneg_topunp_gender |
| ID: 965 |
| How many were |
| Enter numerical values.*MenTranswomenNon-binary, genderqueer, or gender non-conforming |
| Men<br>Transwomen |

Page entry logic: This page will show when: Num HIV Neg partners is greater than "0"

### **HIV Negative Partners - PrEP and Alcohol and Drug Use**

ID: 992

The next set of questions will ask only about your [question('option value'), id='676', option='12278'] sexual partner(s) in the last 3 months who told you they were HIV negative.

Logic: Hidden by default

ID: 732

This number cannot be greater than the number of partners who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Shortname / Alias: hivneg toldyouprep

ID: 729

How many of your sexual partners who told you they were HIV negative told you they were taking PrEP?

Number must be less than or equal to [question('option value'), id='676', option='12278'].\*

Logic: Show/hide trigger exists.

Shortname / Alias: hivneg youtoldprep

ID: 730

Regarding your sexual partners who told you they were HIV negative, did you tell any of them that you were taking PrEP?\*

- () Yes
- () No
- () I was not taking PrEP at this time

Logic: Hidden by default

ID: 733

This number cannot be greater than the number of partners who told you they were HIV negative ([question('option value'), id='676', option='12278']). Please correct this.

Logic: Hidden unless: #162 Question "Regarding your sexual partners who told you they were HIV negative, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivneg\_youtoldprepnum
ID: 731

How many of your sexual partner(s) who told you they were HIV negative did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12278'].\*

Shortname / Alias: hivneg timesdrunk

ID: 740

In the past 3 months, how many of the times you had anal sex with partners who told you they were HIV negative were you or this person under the influence of alcohol or drugs?\*

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Action: Custom Script: Script to check PrEP number not greater than the total number of partners

Page entry logic: This page will show when: Num HIV Pos partners is greater than "0"

**HIV Positive Partners** 

ID: 770

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Shortname / Alias: hivpos timesbot

ID: 775

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom?\*

\_\_\_\_\_

Shortname / Alias: hivpos\_timestop

ID: 776

In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the top?\*

\_\_\_\_\_\_

**Page entry logic:** This page will show when: #165 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom?" is greater than "0"

**HIV Positive Partners - Condomless Receptive AI** 

ID: 782

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 783

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='775']). Please correct this.

Shortname / Alias: hivpos timesbotunp

ID: 784

In the past 3 months, how many of the [question('value'), id='775'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom were without a condom? \*
Action: Custom Script: Check number condomless is not greater than total times

**Page entry logic:** This page will show when: #167 Question "In the past 3 months, how many of the [question('value'), id='775'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the bottom were without a condom? " is greater than "0"

## **HIV Positive Partners - Condomless Receptive AI**

ID: 786

The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive.

Logic: Hidden by default

ID: 1008

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivpos botunp typ

ID: 788

Regarding the partners who told you they were HIV positive who you had <u>condomless receptive</u> anal sex with (where you were the bottom), how many were...

| ニハナヘア | numerical | 1/2/1 | 100 ^ |
|-------|--------------------|-------|-------|
| _,,, | IIIIIIII EI II. AI | vali | 162 |

| | _remarks partier(s), someone you are in a relationship with |
|---|---|
| | _Casual hook-up(s) or one-night stand(s) |
| | _A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, |
| etc. | |

Romantic partner(s) someone you are in a relationship with

Logic: Hidden by default

ID: 1009

The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

| Validation: Must be numeric |
|---|
| Shortname / Alias: hivpos_botunp_gender |
| ID: 994 |
| How many were |
| Enter numerical values.*Men |
| Transwomen |
| Non-binary, genderqueer, and gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: #166 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) who told you they were HIV positive where you were the top?" is greater than "0" |
| HIV Pos Partners - Condomless Insertive Al |
| ID: 792 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive. |
| Logic: Hidden by default |

This number cannot be greater than the number of times you had anal sex where you were the top ([question('value'), id='776']). Please correct this.

ID: 793

| Shortname / Alias: hivpos_timestopunp |
|---|
| ID: 794 |
| In the past 3 months, how many of the [question('value'), id='776'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the top were without a condom? * |
| Action: Custom Script: Script to check number condomless is not greater than the totals |
| Page entry logic: This page will show when: #170 Question "In the past 3 months, how many of the [question('value'), id='776'] times you had anal sex with sexual partner(s) who told you they were HIV positive where you were the top were without a condom? " is greater than "0" |
| HIV Positive Partners - Condomless Insertive Al |
| ID: 796 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12279'] sexual partner(s) in the last 3 months who told you they were HIV positive. |
| Logic: Hidden by default |
| ID: 1012 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivpos_topunp_typ |
| ID: 798 |
| Regarding the partners who told you they were HIV positive who you had <u>condomless insertive</u> <u>anal sex with (where you were the top)</u> , how many were |
| Enter numerical values.* Romantic partner(s), someone you are in a relationship with |
| Enter numerical values.* Romantic partner(s), someone you are in a relationship with Romantic partner(s) or one-night stand(s) |

| etc. |
|---|
| Logic: Hidden by default |
| ID: 1013 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivpos_topunp_gender |
| ID: 995 |
| How many were |
| Enter numerical values.* Men Transwomen Non-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: Num HIV Pos partners is greater than "0" |
| HIV Positive Partners - HIV Trt and PrEP |
| Logic: Hidden by default |
| ID: 799 |
| This number cannot be greater than the number of partners who told you they were HIV positive ([question('option value') id='676', option='12279']). Please correct this |

\_A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs,

| Shortname / Alias: hivpos_toldyouhivmeds |
|------------------------------------------|
| ID: 800 |

How many of your sexual partners who told you they were HIV positive told you they were taking medication to treat HIV?

Number must be less than or equal to [question('option value'), id='676', option='12279'].

\_\_\_\_\_\_

## Logic: Hidden by default

ID: 920

The number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Shortname / Alias: hivpos toldyouundetect

ID: 918

How many of your sexual partners who told you they were HIV positive told you they were undetectable?

Number must be less than or equal to [question('option value'), id='676', option='12279'].

## Logic: Show/hide trigger exists.

Shortname / Alias: hivpos youtoldprep

ID: 801

Regarding your sexual partners who told you they were HIV positive, did you tell any of them that you were taking PrEP?\*

- () Yes
- () No
- () I was not taking PrEP at this time

## Logic: Hidden by default

ID: 802

This number cannot be greater than the number of partners who told you they were HIV positive ([question('option value'), id='676', option='12279']). Please correct this.

Logic: Hidden unless: #175 Question "Regarding your sexual partners who told you they were HIV positive, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivpos\_youtoldprepnum

ID: 803

How many of your sexual partner(s) who told you they were HIV positive did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12279'].

| Shortname / Alias: hivpos_timesdrunk |
|---|
| ID: 807 |
| In the past 3 months, how many of the times you had anal sex with partners who told you they were HIV positive were you or this person under the influence of alcohol or drugs?* |
| Action: JavaScript: Hide General Error Message |
| Action: Custom Script: Script to check med number not greater than the total number of partners |
| Action: Custom Script: Script to check undetectable number not greater than the total number of partners |
| Action: Custom Script: Script to check PrEP number not greater than the total number of partners |

Page entry logic: This page will show when: Num HIV Unk partners is greater than "0"

**HIV Status Unknown Partners** 

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Shortname / Alias: hivunk timesbot

ID: 815

In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom?\*

\_\_\_\_\_\_\_

Shortname / Alias: hivunk\_timestop

ID: 816

In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top?\*

\_\_\_\_\_

**Page entry logic:** This page will show when: #178 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of <a href="where you were the bottom?" where you were the bottom?" is greater than "0"</a>

**HIV Status Unknown Partners - Condomless Receptive Al** 

ID: 822

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 823

This number cannot be greater than the number of times you had anal sex where you were the bottom ([question('value'), id='815']). Please correct this.

| ID: 824 |
|---|
| In the past 3 months, how many of the [question('value'), id='815'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom were without a condom? * |
| Action: Custom Script: Check number condomless is not greater than total times |
| Page entry logic: This page will show when: #180 Question "In the past 3 months, how many of the [question('value'), id='815'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the bottom were without a condom? " is greater than "0" |
| HIV Status Unknown Partners - Condomless Receptive Al |
| ID: 826 |
| The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of. |
| Logic: Hidden by default |
| ID: 1016 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivunk_botunp_typ |
| ID: 828 |
| Regarding the partners whose HIV status you were not sure of who you had <u>condomless</u> <u>receptive anal sex with (where you were the bottom)</u> , how many were |
| receptive anal sex with (where you were the bottom), how many were Enter numerical values.* |
| Enter numerical values.* Romantic partner(s), someone you are in a relationship with |

Logic: Hidden by default ID: 1017 The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. Validation: Must be numeric Shortname / Alias: hivunk botunp gender ID: 996 How many were... Enter numerical values.\* Men Transwomen Non-binary, genderqueer, or gender non-conforming **Action: Custom Script: Script to check continuous sum totals Action: Custom Script: Script to check continuous sum totals** 

**Page entry logic:** This page will show when: #179 Question "In the past 3 months, how many times did you have anal sex with sexual partner(s) whose HIV status you were not sure of <a href="where you were the top?" where you were the top?" is greater than "0" where you were the top?" where you were the top?" is greater than "0" where you were the you wer

## **HIV Status Unknown Partners - Condomless Insertive AI**

ID: 832

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 833

This number cannot be greater than the number of times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top ([question('value'), id='816']). Please correct this.

Shortname / Alias: hivunk\_timestopunp

ID: 834

In the past 3 months, how many of the [question('value'), id='816'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top were without a condom?\*

Action: Custom Script: Script to check number condomless is not greater than the totals

**Page entry logic:** This page will show when: #183 Question "In the past 3 months, how many of the [question('value'), id='816'] times you had anal sex with sexual partner(s) whose HIV status you were not sure of where you were the top were without a condom?" is greater than "0"

**HIV Status Unknown Partners - Condomless Insertive AI** 

ID: 836

The next set of questions will ask only about your [question('option value'), id='676', option='12280'] sexual partner(s) in the last 3 months whose HIV status you were not sure of.

Logic: Hidden by default

ID: 1020

The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Validation: Must be numeric

Shortname / Alias: hivunk topunp typ

Logic: Hidden by default

| Regarding the partners whose HIV status you were not sure of who you had <u>condomless</u> <u>insertive anal sex with (where you were the top)</u> , how many were |
|---|
| Enter numerical values.* Romantic partner(s), someone you are in a relationship with Romantic partner(s) or one-night stand(s) A transactional partner(s), who you had sex with in exchange for money, housing, food, drugs, etc. |
| Logic: Hidden by default ID: 1021 |
| The total number cannot be greater than the number of sexual partner(s) in the last 3 months whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this. |
| Validation: Must be numeric |
| Shortname / Alias: hivunk_topunp_gender ID: 997 |
| How many were |
| Enter numerical values.*MenTranswomenNon-binary, genderqueer, or gender non-conforming |
| Action: Custom Script: Script to check continuous sum totals |
| Action: Custom Script: Script to check continuous sum totals |
| Page entry logic: This page will show when: Num HIV Unk partners is greater than "0" |
| HIV Status Unknown Partners - PrEP |

This number cannot be greater than the number of partners whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Shortname / Alias: hivunk\_toldyouprep

ID: 840

How many of your sexual partners whose HIV status you were not sure of told you they were taking PrEP?

Number must be less than or equal to [question('option value'), id='676', option='12280'].\*

\_\_\_\_\_

Logic: Show/hide trigger exists.

Shortname / Alias: hivunk youtoldprep

ID: 841

Regarding your sexual partners whose HIV status you were not sure of, did you tell any of them that you were taking PrEP?\*

- ()Yes
- () No
- () I was not taking PrEP at this time

Logic: Hidden by default

ID: 842

This number cannot be greater than the number of partners whose HIV status you were not sure of ([question('option value'), id='676', option='12280']). Please correct this.

Logic: Hidden unless: #187 Question "Regarding your sexual partners whose HIV status you were not sure of, did you tell any of them that you were taking PrEP?" is one of the following answers ("Yes")

Shortname / Alias: hivunk youtoldprepnum

ID: 843

How many of your sexual partner(s) whose HIV status you were not sure of did you tell you were taking PrEP?

Numbers must be less than or equal to [question('option value'), id='676', option='12280'].\*

| ID: 847 |
|---|
| In the past 3 months, how many of the times you had anal sex with partners whose HIV status you were not sure of were you or this person under the influence of alcohol or drugs?* |
| Action: Custom Script: Script to check PrEP number not greater than the total number of partners |
| Action: Custom Script: Script to check PrEP number not greater than the total number of partners |
| Perceived HIV Risk |
| Shortname / Alias: perceivedrisk1 |
| ID: 762 |
| Based on your reported sexual activities over the last 3 months, how at risk do you think you were for contracting HIV in the last 3 months?* ( ) Not at all at risk for contracting HIV |
| ( ) Somewhat at risk for contracting HIV |
| ( ) High risk for contracting HIV |
| Shortname / Alias: perceivedrisk2 |
| ID: 763 |
| What is your gut feeling about how likely you are to get infected with HIV?* ( ) Extremely unlikely |
| ( ) Very unlikely |
| ( ) Somewhat likely |
| ( ) Very likely |
| ( ) Extremely likely |
| Shortname / Alias: perceivedrisk3 |

| () None of the time |
|----------------------------------------------------------------|
| () Rarely |
| () Some of the time |
| ( ) A lot of the time |
| ( ) All of the time |
| ( ) All of the time |
| Perceived HIV Risk |
| Shortname / Alias: perceivedrisk4 |
| ID: 765 |
| Getting HIV is something I am* ( ) Not concerned about |
| ( ) A little concerned about |
| ( ) Moderately concerned about |
| ( ) Concerned about a lot |
| ( ) Extremely concerned about |
| ( ) Extremely concerned about |
| Shortname / Alias: perceivedrisk5 |
| ID: 766 |
| There is a chance, no matter how small, I could get HIV:* |
| ( ) Strongly Disagree |
| () Disagree |
| () Agree |
| ( ) Strongly Agree |
| Shortname / Alias: perceivedrisk6 |
| ID: 767 |
| I think my chances of getting infected with HIV are:* ( ) Zero |
| ( ) Almost zero |
| () Small |
| ( ) Moderate |

I worry about getting infected with HIV:\*

() Large

| ( | ) | Very | large |
|----|---|------|-------|
| ١. | , | , | |

## PHQ-2/GAD-2

ID: 768

Now we are going to ask you about your mental health and how you have been feeling recently.

Shortname / Alias: mentalhealthscreener

ID: 388

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Little interest or pleasure in doing things | () | () | () | () |
| Feeling<br>down,<br>depressed,<br>or<br>hopeless | () | () | () | () |
| Feeling<br>nervous,<br>anxious or<br>on edge | () | () | () | () |
| Not being<br>able to<br>stop or<br>control<br>worrying | () | () | () | () |

Page entry logic: This page will show when: psychdistress1 is greater than or equal to "3"

# PHQ-8

Shortname / Alias: phq8

ID: 397

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| Over the past 2 | weeks, | now often | nave you | been both |
|---|---|---|---|---|
| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
| Trouble falling or staying asleep, or sleeping too much | () | () | () | () |
| Feeling tired<br>or having<br>little energy | () | () | () | () |
| Poor appetite or overeating | () | () | () | () |
| Feeling bad<br>about<br>yourself - or<br>that you are<br>a failure or<br>have let<br>yourself or<br>your family<br>down | () | () | () | () |
| Trouble concentrating on things, such as reading the newspaper or watching television | () | () | () | () |
| Moving or speaking so | () | () | () | () |

| slowly that other people could have noticed, or the opposite - being so fidgety or restless that you have been moving around a lot more than usual |
|---|
|---|

Page entry logic: This page will show when: psychdistress2 is greater than or equal to "3"

## GAD-7

Shortname / Alias: gad7

ID: 404

Over the past 2 weeks, how often have you been bothered by any of the following problems?\*

| | Not<br>at<br>all | Several<br>days | More<br>than<br>half<br>the<br>days | Nearly<br>every<br>day |
|---|---|---|---|---|
| Worrying<br>too much<br>about<br>different<br>things | () | () | () | () |
| Trouble relaxing | () | () | () | () |
| Being so<br>restless<br>that it is<br>hard to sit<br>still | () | () | () | () |
| Becoming easily | () | () | () | () |

| annoyed<br>or irritable | | | | |
|---|---|---|---|---|
| Feeling<br>afraid as if<br>something<br>awful<br>might<br>happen | () | () | () | () |

## **Social Isolation**

Shortname / Alias: socialisolation

ID: 432

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| I feel<br>left out. | () | () | () | () | () |
| I feel<br>that<br>people<br>barely<br>know<br>me. | () | () | () | () | () |
| I feel<br>isolated<br>from<br>others. | () | () | () | () | () |
| I feel that people are around me but not with me. | () | () | () | () | () |

# **Emotional Support**

Shortname / Alias: emotionalsupport

ID: 411

Please respond to each item by marking one circle per row.\*

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| I have someone who will listen to me when I need to talk. | () | () | () | () | () |
| I have someone to confide in or talk to about myself or my problems. | () | () | () | () | () |
| I have someone who makes me feel appreciated. | () | () | () | () | () |
| I have someone to talk with when I have a bad day. | () | () | () | () | () |

# **Informational Support**

Shortname / Alias: informational support

ID: 417

| • | Never | Rarely | Sometimes | Usually | Always |
|---|-------|--------|-----------|---------|--------|
|---|-------|--------|-----------|---------|--------|

| I have someone to give me good advice about a crisis if I need it. | () | () | () | () | () |
|---|---|---|---|---|---|
| I have someone to turn to for suggestions about how to deal with a problem. | () | () | () | () | () |
| I have someone to give me information if I need it. | () | () | () | () | () |
| I get useful<br>advice<br>about<br>important<br>things in<br>life. | () | () | () | () | () |

# **Instrumental Support**

Shortname / Alias: instrumentalsupport

ID: 422

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| Do you have someone to help you if you are | () | () | () | () | () |

| confined to bed? | | | | | |
|---|---|---|---|---|---|
| Do you have someone to take you to the doctor if you need it? | () | () | () | () | () |
| Do you have someone to help with your daily chores if you are sick? | () | () | () | () | () |
| Do you have someone to run errands if you need it? | () | () | () | () | () |

# Companionship

Shortname / Alias: companionship

ID: 427

| | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|
| Do you have someone with whom to have fun? | () | () | () | () | () |
| Do you have someone with | () | () | () | () | () |

| whom to relax? | | | | | |
|---|---|---|---|---|---|
| Do you have someone with whom you can do something enjoyable? | () | () | () | () | () |
| Do you find companionship when you want it? | () | () | () | () | () |

## Thank You!

ID: 1

Thank you for taking this survey and for participating! We greatly appreciate your involvement!

## In-depth Interview Guide

Participant study ld:

#### PRE-INTERVIEW PARTICIPANT DATA CHECK

Check participants use to determine whether they are low or high use. Note we want to know the average number of days per week participants used a key component of the app (medication tracker, daily quest, social wall).

| | Average<br># days<br>per week |
|------------------------------|-------------------------------|
| Moderate to high use (n ~ 5) | <u>&gt;</u> 4 |
| Low to no use (n ~ 5) | <4 |

Circle participants defined use: MODERATE TO HIGH USE LOW TO NO USE

#### **INTERVIEW GUIDE**

#### Introduction

Hello, my name is \_\_\_\_\_. I am a P3-T study staff member and I want to thank you for taking time out of your day to talk to me today.

We are talking to you today about the P3-T app study that you have been participating in. I am going to ask you questions about your experience and impressions of the app, how you used it, and how it may have impacted your behaviors over the past 3 months. I will also ask for your suggestions on how we might improve the app to make it more useful to others like yourself.

There are no right or wrong answers and you are really the expert here today. I am most interested in your honest thoughts and opinions. If there are any questions I ask that you don't wish to answer, you can just say "skip" and we will just move on to the next question. Our talk today will last about 30-45 minutes and we will be audio recording your responses so that we can better remember everything you say. We will not be using your name or any other personal identifying information and we will destroy the recording within 6 months of the end of the study. Anything we talk about today is confidential and we will not be sharing your responses with any of your medical providers or anyone else outside of the study team. Ok, do you have any questions before we get started?

Note for interviewers: the interview questions will split for moderate to high users and low to no users, and are noted as such.

#### **PrEP** experience

It's helpful if you tell me a little bit about your experiences taking PrEP, so to start...

What prompted you to start taking PrEP?

Had you taken PrEP at any time before the P3-T study?

## If YES:

Tell me about your experience taking PrEP before you joined P3-T What systems or routines did you have – if any - for taking PrEP every day?

## If NO:

How was the experience of starting P3-T when you started taking PrEP?

Did you ever stop taking PrEP for a week or more during the trial?

If YES:

What led to that break in taking PrEP?
Did you start taking PrEP again after that?

If YES:

What made you decide to restart taking PrEP?

Are you taking PrEP now?

If NO:

What led you to stop?

If YES:

How long do you think you will stay on PrEP for?

Do you have people in your life that you can talk to about being on PrEP?

#### **Overall experience**

When you first joined the study, what did you hope to get out of using the P3-T app?

How well did your experience using the P3-T app meet these expectations?

What were your favorite app features? (and why)

How did P3-T impact your experience with PrEP?

How useful were the daily P3-T reminders for taking PrEP?

Did you start remembering to take PrEP without them?

How long did it take for your P3-T PrEP-taking strategy to become routine? After it became routine, what kept you coming back to the app?

Did you tell anyone or show anyone the app while you were using it?

If YES:

Why?

#### FOR LOW TO NO USERS ONLY

It looks like you didn't use the app very much, can you tell me about that?

What did you want from the app that you weren't getting?

What would have made you use the app more?

## **Technical issues**

Did you receive notifications from the app?

Could you describe any technical problems you had?

#### **Features**

#### Medication tracker

How was your experience setting up the medication tracker?

Tell me about setting it up for the first time, what strategy did you pick? How did that strategy work out for you?

Did you ever change your strategy during the trial?

If yes, can you tell me about what prompted you to change it? How did changing your strategy work for you?

How easy was it to use the app to track whether or not you took PrEP each day?

Can you tell me about days you didn't log your meds?

What was going on for you?

Did you ever notice a pattern to days you didn't log meds (weekends?)

How often did you review your medication calendar? Did you ever show it to anybody?

#### **Daily Quests**

Tell me about your experience with the daily quests...

What suggestions do you have for new Daily Quests? (or other ways to improve this feature?)

## Knowledge Center

Tell me about your experience with the knowledge center...

Where else do you go to get health, and sexual health, information?

What kind of sexual health questions do you google?

What kind of information would you like to see more of in this app?

## Social Wall

Tell me about your experience with the social wall...

How often did you read the discussions on the social wall? How often did you comment or interact with other users?

What were topics that you liked reading about on the social wall?

How connected did you feel to the other users on the app?

Could something be added that would make you feel more connected?

What made you want to contribute/not contribute to the social wall?

What would you change about this feature of the app to make it better?

#### Rewards

What did you think about the rewards that were offered within the app?

How did the rewards motivate you to continue to use the app?

## Bank account

What did you think about the bank account feature?

Did you notice when your amount went up or down?

How did the bank account impact your app use?

#### Adherence Counseling

Tell me about your experiences talking to the P3-T adherence counselor...

What did you like about it?

What did you not like about it?

What was useful to you?

What did you discuss with the adherence counselor?

How did you feel about having those kinds of conversations over text?

How would you feel about having on a phone call? By video chat?

How easy was it for you to get in touch with your counselor?

How convenient were the times that the counselor was available?

## Wrap up

Before we wrap up, I'd like to give you a chance to share any other thoughts you have about the P3-T app that I didn't ask you about yet. What else would you like us to know about your experience with the app or with being in the study?

Thank you for your time today and for your experiences and willingness to test the P3-T app!



BA-CF-G-006 Version 6

Effective Date: 06Mar2019

#### **AMS-BAT**

## Materials needed for methods of DBS and Plasma collection for TFV-DP testing

Reference: BA-SOP-G-011

- 1. Materials needed for methods of DBS and Plasma collection for one PK single time point
  - 1.1 Equipment needed
    - 1.1.1 Centrifuge (can centrifuge with 800xg for 10 minutes, non-temperature setting),
    - 1.1.2 Freezer (-20°C or -70°C or-80°C).
  - 1.2 Materials needed for DBS and plasma preparation
    - 1.2.1 K2-EDTA Spray Dried Tube (1 tube),
      - Product code; BD Vacutainer spray-coated K2 EDTA Tubes.
    - 1.2.2 Whatman Protein Saver Card (#903) (1 card),
      - Product code; Whatman™ 10534612 | 903 Protein Saver Card
    - 1.2.3 Cryovial Tube (2 tubes per sample),
      - Product code; SARSTEDT cryotubes (2 mL, product code: 72.694.006
    - 1.2.4 Gas-impermeable (zip-lock) bag (1 bag)
      - Prodect code: Whatman 10534321 Foil-Barrier Ziploc Bags for Card, Pack of 100
    - 1.2.5 Desiccant (1 pack),
      - **Product code:** Whatman™ 10548234 Desiccant Packs for 903 Protein Saver Cards (Pack of 100)
    - 1.2.6 Pipette for DBS preparation: Auto Pipette (Max Vol. 100 uL),
    - 1.2.7 Pipette for transfer plasma: Auto Pipette (Max Vol. 1000 uL) or Transfer Pipette,
    - 1.2.8 Whatman card drying rack,
    - 1.2.9 Sample Sticker labels (waterproof sticker label),
    - 1.2.10 Gloves (preferably powder-free),
    - 1.2.11 Permanent marker and Pen.

## 2. DBS and Plasma Collection Procedure for TFV-DP testing

#### 2.1 EDTA Blood collection

- 2.1.1 Collect the blood into K2-EDTA containing Tube (at least 2 mL size of K2-EDTA containing tube),
- 2.1.2 Gently invert the tube (10 times) to mix the blood thoroughly,
- 2.1.3 Label the tubes with the patient ID number, initial, visit, date and time of blood draw using label,
- 2.1.4 Blood sample should be processed as soon as possible (within 1-2 hours), but need to be initiated within 24 hours of draw time. No more than 24 hours should elapse.
- 2.1.5 If the site staff cannot process the DBS and plasma preparation within 1-2 hours, the EDTA whole blood sample should be kept at 4°C and ship with Ice or Gel Cold Shipping Pack (to remain temperature at 4-10°C).

#### 2.2 Dried Blood Spots (DBS) Collection

- 2.2.1 Label the Whatman Protein Saver 903 Card with the patient ID number, initial, visit, date and time of blood draw using provided sticker label (waterproof sticker label).
- 2.2.2 If the whole blood has been kept or shipped under the cold temperature (4-10°C). The samples should sit at room temperature for about 15 mins in order to reach room temp before spotting.
- 2.2.3 Gently invert the tube (8 to 10 times) to mix the blood thoroughly. After the blood is completely mixed, remove the cap, and apply 25 µL of the whole blood to a single spot on the Whatman Protein Saver 903 Card (Slowly expel blood from the tip and touch the drop to the paper, allowing the blood to absorb. Do not touch the card with the pipette tip). Repeat four times to fill all five spots on the card. Do not touch the DBS circle once blood is applied.
- 2.2.4 Written down; initials of staff who spotted blood on card, date and time of spotting on the right bottom of filter paper.
- 2.2.5 Allow the Dried Blood Spots Cards to air dry without the card flap covering the spots in a drying rack that is clean and dry and protected from rodents, insects and direct sunlight for <u>at least 3</u> hours or overnight is acceptable. (check that it completely dried before storage)
  - **Note**; Do not use electric dryer or heat, stack or allow DBS to touch other surfaces during the drying process.
- 2.2.6 Put the card in a gas-impermeable (zip-lock bag) containing 1 pack of desiccant. Store no more than one card per bag.

#### **DBS Preparation Flowchart:**



## **2.3 Plasma Collection Procedure** (should be performed after DBS sample is collected)

- 2.3.1 Separate plasma from blood by centrifuging at least 800xg for 10 minutes at room temperature,
- 2.3.2 Label the cryovials with the patient ID number, initial, visit, date and time of blood draw using provided sticker label,
- 2.3.3 Transfer plasma (at least 0.25 mL/tube is required) into two storage cryovials with a screw cap.

## 2.4 Freezer log Recording

2.4.1 Record all sample information (site, patient identification number, patient initials, visit, date/time of blood draw and date/time etc) on the freezer record log form (BA-FM-G-046 Freezer Log for Plasma-Sample and BA-FM-G-047 Freezer Log for DBS).

### 2.5 Sample Storage

2.5.1 Store Dried Blood Spots Card (DBS) and Plasma in the freezer (-20°C or -70°C or -80°C) within 1 hour after preparation.

#### Note:

- DBS should be stored at -20°C or lower (-70°C or -80°C are preferable) and it can be stored at 4°C for about one month.
- DBS sample should not be stored at room temp more than one week because the sample is degraded in the first week of storage at room temperature. Note in the freezer log for if the DBS has been store at room temperature.

## 2.6 Sample Shipment

2.6.1 Ship Dried Blood Spots Card (DBS) and Plasma on dry ice.

## **RCT Eligibility Screening Form**

Informed Consent Script for Eligibility Screening Study Staff Instructions: Please read the script below before conducting eligibility screening.

Thank you for your interest in the P3-T research study. The purpose of our research study is to test a PrEP adherence app for young gay and bisexual men who are starting PrEP. We are currently looking for young gay or bisexual men who can take part in our study. Participation in the P3-T study is six months long and involves 3 study visits: 1) an enrollment visit, 2) a follow-up visit at 3 months, and 3) a follow-up visit at 6 months. Participants complete a survey at every study visit and give a blood sample at 3- and 6-months visits. Since this is a randomized control study, some participants will get the app and some participants will not. For those who get the app, participation will involve using the app daily during the first three months of the study. Daily app use takes about 5-10 minutes.

Before we can move forward, we need to ensure that you meet a few eligibility requirements. The screening process is optional, and you may choose at any time not to participate. If you choose to proceed, you will be asked a few questions, and your answers will determine whether or not you are eligible to participate in the research study. This will take approximately 5 minutes. The screener asks questions about sensitive topics, such as age, gender identity and sexual partner preference(s). Some of these questions are of personal nature and you may feel uncomfortable or embarrassed answering them -you can decide to stop answering questions at any time. If you don't answer all the questions, we may not be able to find out if you meet the eligibility criteria for the study - therefore, we might not be able to schedule a study visit. If you meet the eligibility criteria for this study and are interested in participating, we will begin the study visit. Any information shared in this survey is strictly confidential and will only be used for research study purposes. All the information that is gathered from you is safely stored.

Data collected in this screening survey will not be connected to the main study should you screen eligible and choose to participate in the main study. The information I am entering into this eligibility screening form on my laptop will be stored on a secure server.

You may not benefit personally from screening for study eligibility. If you have questions, or concerns about the study eligibility screener you may call INSERT NUMBER.

| Study Staff Instructions: Please ask the following questi | on and reply based on the response. |
|---|---|
| Do you consent to be screened for the P3T study? Yes No | |
| Great. Let's get started with the screener! | |
| Sorry, if you do not consent to be screened, you cannot o | continue the screener. Thank you for your time. |
| Section 1: Inclusion Criteria | |
| Study Staff Instructions: Please ask the following questi | on and reply based on the response. |
| Do you understand, and are you comfortable speaking and reading Thai? | ○Yes<br>○No<br>(must be yes to be eligible) |
| Are you between the ages of 16 to 24? | ○Yes<br>○ No<br>(must be yes to be eligible) |
| Do you currently own an Android or iOS smartphone? | Yes No (must own a phone (iOS or Android) to be eligible) |

| **** | 0.771 |
|---|---|
| What sex were you assigned at birth? | Male |
| | Female |
| | (must be male to be eligible) |
| What is your current gender identity? | ○ Male |
| | ○ Female |
| | O Trans-female, trans-woman, or trans-feminine |
| | Trans-male, trans-man, or trans-masculine |
| | Genderqueer, gender non-conforming or non- |
| | binary |
| | Another Gender |
| | (must be male to be eligible) |
| If identified as 'another gender,' what is | |
| it? (please state) | <del></del> |
| Who do you have sex with or intend to have sex | Men |
| with? (check all that apply) | Women |
| | Transmen |
| | Transwomen |
| | (must be men and/or transwomen to be eligible) |
| | (and the first that the first to the first to the first to |
| Do you plan to start taking PrEP in the next 14 days? | O Yes |
| | O No |
| | (must be yes to be eligible) |
| Section 2: Exclusion Criteria | |
| Are you participating in another experimental PrEP | ○Yes |
| adherence intervention? | $\bigcirc$ No |
| | (must be no to be eligible) |
| Do you plan move out of Bangkok in the next 6 | ○ Yes |
| months? | O No |
| | (must be no to be eligible) |
| Section 3: Staff Verification of Eligibility Criteria | |
| Does the participant have an Android or iPhone | ○ Yes |
| smartphone with them? | O No |
| | (must be yes to be eligible) |
| If yes, which type of operating system? | <ul><li>○ Android</li><li>○ iOS (iPhone)</li></ul> |

| If And | roid which version: | | |
|---|---|---|---|
| Go to | eck the operating system version: settings > About phone vice > tap Android | | |
| If iOS<br>To che | (iPhone) which version: eck the operating system version: Go to seneral > About > Version | ettings | |
| Does 1 | he smartphone meet the phone operating | | |
| systen | 1 | $\circ$ | Yes version requirements for |
| the ap | o? | Ŏ | No (must be yes to be eligible) |
| | rements: | | (must be yes to be engione) |
| | id: must have | | |
| | 1 4.4 or newer<br>e: must have iOS | | |
| 10 or 1 | | | |
| | individual unable to be consented due to a | | Yes |
| active | substance use or psychological condition? | O | No |
| | yould only be yes if one of these condition to be eligible) evident at the time of scre | | (must<br>might |
| | dividual from providing informed consen | ıt. | |
| | | | Yes |
| Is the study? | participant eligible to participate in the | $\mathcal{O}$ | No |

# Appendix A

All documents will be translated into Thai and back-translated into English by the Thai study team.

Contents include:

1. RCT Consent Form

- 2. RCT 3-month Blood Draw
- 3. RCT 6-month Blood Draw

## Consent Form- Full Study

## P3-T Randomized Controlled Trial Consent

Chulalongkorn University & Thai Red Cross AIDS Research Centre (TRC-ARC) Consent to Participate in a Research Study Participants ages 16-24 years old

Duke IRB Study # xxxxxxx

Consent Form Version Date: Version 1.0 dated DD-MM-YEAR

Title of Study: P3-T: Novel mHealth Technologies to Enhance PrEP Adherence among Thai YMSM, Collaborative Adaptation and Evaluation

## **Principal Investigators:**

Sara LeGrand, PhD +1 (919) 438-0448 sara.legrand@duke.edu

Wipaporn Natalie Songtaweesin, MBBS +66 (662) 256-4930 wipaporn@doctors.org.uk

**Sponsor:** Duke University

**Funding Source:** National Institutes of Health (NIH)

#### **Study Contact:**

Wipaporn Natalie Songtaweesin, MBBS +66 (662) 256-4930 wipaporn@doctors.org.uk

## **Key Study Information**

- The purpose of this study is to gain your perspective as a young man who has sex with men on a mobile phone app called P3-T. The purpose of P3-T is to help young men who have sex with men take PrEP, a medicine that helps prevent HIV.
- You are being asked to take part in a research study. You do not have to join. You can quit the study at any time, for any reason, and nothing bad will happen as a result.
- This form contains details about the study that will help you make a choice about participating.
- We are asking about 60 people to take part in the study.
- Participants in the study will be randomly sorted into two groups. One group will get the P3-T app and one group will not get the P3-T app. Research staff have no control over what group you are sorted into and no one can change what group you are in.
- All participants will be in the study for 6 months.

- The study involves three clinic visits:
  - At the enrollment visit you will meet with research study staff who will guide you through the visit.
    - You will complete a survey to collect information about your demographics, factors related to PrEP adherence, sexual risk, among other items, and review the intervention materials.
  - At the 3- and 6-month visits, a research study staff will guide you through the visit.
    - You will complete a survey similar to the enrollment survey.
    - A trained phlebotomist will draw a small amount of blood (2mL) from a vein in your arm or your hand.
    - At the 3-month visit, some participants will have an opportunity to complete an interview with a study staff member about their experience using the app.
- The study will include daily use of the intervention materials (about 5-10 minutes) for the first three months of the study period.
- While you may not personally benefit from participating in the study, your feedback about
  the intervention and your experience in the study may help other young men who have sex
  with men by adding to the resources available to help them protect their health.
- There are potential risks or discomforts involved with being in this study including:
  - While completing the survey, you may find some of the questions a little embarrassing or difficult to answer.
  - Study staff will make every effort to keep your information confidential, but there is a small possibility that your name and information that you share during this research study could become known to others. The efforts we will take to prevent this from happening are described in detail below.
  - o For the blood draws, you may experience discomfort or bruising at site where the blood is drawn. There is a small risk of fainting and a rare risk of infection.
- Study staff will make every effort to keep your information confidential. The efforts we will take to protect your confidentiality are described in detail below.
- For participating in this study, you will receive \$20 at each of the three visits (total \$60). Depending on what group you are randomly sorted into, you may have the opportunity to earn additional money, up to \$15 for app use and \$20 for the qualitative interview (total \$95).
- There are no costs to you for participating in this study.

#### What are some general things you should know about research studies?

You are being asked to take part in a research study. You do not have to join. You can quit the study at any time, for any reason, and nothing bad will happen as a result.

We are doing this research to learn information that could help young people like you, in the future. All research has risks and benefits. We will talk about these risks and benefits with you before you decide if you want to join the study.

This form contains details about the study that will help you make a choice about participating. You will be given a copy of this form to keep. You can ask any questions you want of the study staff, or the researchers listed at the top of this form.

#### What is the purpose of this study?

The purpose of this study is to gain your perspective as a young man who has sex with men on a mobile phone app called P3-T. The purpose of P3-T is to help young men who have sex with men take PrEP, a medicine that helps prevent HIV. This study will help us see if the app helps

young men who have sex with men who are starting PrEP take it regularly. HIV rates are high among young men who have sex with men. If people at risk of HIV take an HIV treatment medicine on a regular basis, they are much less likely to get infected with HIV.

The idea of taking a medicine to prevent HIV is called pre-exposure prophylaxis, or "PrEP" for short. Some people have trouble taking PrEP, so we developed P3-T to help them be active in their own health care and remember to take their PrEP. The P3-T app includes features such as a medication tracker and reminders, daily activities including a social wall where you can anonymously connect with other PrEP users, access to an adherence counselor, and resources about PrEP and sexual health. We don't know if the app will work, and that is why we are testing it out.

## How many people will take part in this study?

We are asking about 60 people to take part in the study.

#### How long will your part in this study last?

Your participation in the study will last 6 months.

#### What will happen if you take part in the study?

Participants in the study will be randomly sorted into two groups. One group will get the P3-T app and one group will not get the P3-T app. Research staff have no control over what group you are sorted into and no one can change what group you are in.

All participants will be in the study for 6 months. This study involves three clinic visits as well as daily use of the intervention materials (about 5-10 minutes) for the first three months of the study period.

At the enrollment visit you will meet with research study staff who will guide you through the visit. You will complete a survey to collect information about your demographics, factors related to PrEP adherence, sexual risk, among other items, and review the intervention materials.

You will then have the intervention materials for 3 three months to use. During those months, we ask that you use them a little bit every day (about 5-10 minutes of use).

After 3 months, you will come back in for a follow up visit. At the 3-month follow up visit you will meet again with a research study staff member. You will complete a survey similar to the one completed at enrollment and a trained phlebotomist will draw a small amount of blood (2mL) from a vein in your arm or your hand and several drops of the collected blood will be used to fill in a dried blood spot (DBS) card.

Some participants will have an opportunity to complete an interview with a study staff member about your experience using the app. If you are chosen and are available to participate, audio from the interview will be recorded to make sure we have an accurate record of the information you give us.

After this period, if you were in the group that got the P3-T app, you will still have access, but you will not be required to use it daily. You will not have access to some features, including the adherence counselor and the virtual bank account.

After 6 months, you will come back in for the final follow-up visit. At the follow up visit you will meet again with a research study staff member to guide you through your visit. You will

complete a survey similar to those completed at prior visits and a trained phlebotomist will draw a small amount of blood (2mL) from a vein in your arm or your hand and several drops of the collected blood will be used to fill in a dried blood spot (DBS) card.

At the end of the study, the DBS cards collected at 3- and 6-months will be sent to the Program for HIV Prevention and Treatment (PHPT) Research Unit at Chiang Mai University to be analyzed by Dr. Tim Cressey for the levels of PrEP in your blood. To protect your privacy, your name will not be recorded on any of the samples shipped to PHPT.

We will not be able to provide you with the results of your blood test because samples will not be analyzed until all participants have completed the study.

## What are the possible benefits from being in this study?

You may not benefit personally from being in this research study. However, your feedback about the intervention and your experience in the study may help other young men who have sex with men by adding to the resources available to help them protect their health.

## What are the possible risks or discomforts involved with being in this study?

While completing the survey, you may find some of the questions a little embarrassing or difficult to answer. Your participation is entirely voluntary. You may choose to not answer any question or leave the study at any time. If you are upset by anything we discuss, please let a research staff member know.

You will have 2mL of blood drawn from a vein in your arm or hand at the follow up visits at 3 and 6 months. The total amount of blood taken for the whole study will be 4mL. You may experience discomfort or bruising at site where the blood is drawn. There is a small risk of fainting and a rare risk of infection. Even though we are confident these risks are unlikely if you have any questions or concerns please let the research team know. If you have experienced discomfort, bruising, fainting, or infections from previous blood draws, please let us know.

You will be informed if the study staff learns of any new risks associated with PrEP use or any study activities.

#### What if you want to stop before your part in the study is complete?

You can leave the study at any time you want. The investigators also have the right to stop your participation at any time. This could be because you have failed to follow instructions, have undermined the right or privacy of another participant, or because the entire study has been stopped.

## How will your confidentiality be protected?

To protect you, all of the information collected about you during the study will be identified by a study ID number, not your name. A file that links your name to your study ID number will be kept in a secure folder on a secure server at Duke University separate from the secure folders where your study records are stored. This file will only be accessible to key study staff using a strong password only known to them.

If you participate in an interview with a study staff member at your 3-month visit, your name will not be audio recorded during the interview and the recording will only be used by research team members. The audio recording will be kept confidential, meaning it will only be identified by your study ID number. It will be stored in a secure folder on a secure server at Duke University only

accessible to select study staff. All audio recordings will be permanently destroyed within six months of study completion.

DBS cards sent to PHPT and sample results will only be identified by their study ID number, therefore, the lab at PHPT will not be able to link DBS cards or sample results to participant names. DBS cards will be stored in locked storage at PHPT. The results of the PrEP drug level testing will be sent in a password protected spreadsheet via secure email to the P3-T Principal Investigator in Thailand. The Principal Investigator will store the sample results in a secure folder on a secure server at Duke University only accessible to select study staff.

Your original blood samples, identified only by your study ID number, will be stored securely at Chulalongkorn University. Your DBS card, identified only by your study ID number, will be stored securely at PHPT Research Unit at Chiang Mai University. These samples will be destroyed 3 years after the completion of the study.

All data collected from you after you enroll in the study, including survey, interview, app use, and blood sample data will be linked by your study ID number only.

The project's industry partner, Ayogo, may use de-identified app data from the study for quality improvement of their digital healthcare platform in commercial products such as health apps.

A description of this study will be available on <a href="http://clinicaltrials.gov">http://clinicaltrials.gov</a>, as required by United States Law. This website will not include information that can identify you. At most, the website will include a summary of the study results. You can access this website at any time.

To help further protect your privacy, we have obtained a Certificate of Confidentiality for the study from the United States Department of Health and Human Services (DHHS). It adds special protection for research information that identifies you. It says that we do not have to identify you, even under a court order or subpoena. With this Certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any United States federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of Federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). In addition, your records may be reviewed by certain agencies or people who make sure that the study staff are doing what they are supposed to and everyone in the study is being protected. Under the guidelines of the Federal Privacy Act, the sponsoring agency at the National Institutes of Health (NIH) and the Duke University and Chulalongkorn University IRBs may look at your records. If your study records are reviewed, your identity could become known to them. However, these persons are expected to maintain your individual confidentiality. This means that they will not tell others information about you or that you are in the study. By signing this form, you are allowing such access.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

While every effort will be made to keep your participation in the study and any personal information about you private and confidential, absolute confidentiality cannot be guaranteed. For example, if a study staff member learns something that would immediately put you or others in danger, the study staff member may be required by law to take steps to keep you and others safe. This means that study staff members have to report to the authorities (hospital, police, or social services) any information you say that suggests that you might be in danger, such as telling study staff that you plan to hurt or kill yourself, hurt or kill someone else, or if someone is abusing or neglecting you.

#### Will you receive anything for being in this study?

You will receive \$20 at each of the three visits (total \$60). Depending on what group you are randomly sorted into, you may have the opportunity to earn additional money, up to \$15 for appuse and \$20 for the qualitative interview (total \$95).

## Are there any costs to you for taking part in this study?

You will not be charged for anything that is done for this study.

#### Who is sponsoring this study?

This research is being sponsored by Duke University and is funded by the National Institutes of Health (NIH). This means that the sponsor, Duke University, is providing money from the NIH to Chulalongkorn University and TRC-ARC to help conduct this study. The researchers do not, however, have a direct financial interest with the sponsor or funding source or in the final results of the study.

#### What if you have questions about this study?

You have the right to ask, and have answered, any questions you may have about this research at any time before, during, or after your participation. The Chulalongkorn University investigator in charge of this study is Dr. Wipaporn Natalie Songtaweesin. If you ever have questions, or concerns about this study, you may call or email Dr. Songtaweesin: +66 (662) 256-4930 or <a href="wipaporn@doctors.org.uk">wipaporn@doctors.org.uk</a>

## What if you have questions about your rights as a research participant?

All research on human volunteers is reviewed by a committee that works to protect your rights and welfare. If you have questions or concerns about your rights as a research subject you may contact, anonymously if you wish, the Duke University IRB at +1 (919) 684-3030 or campusirb@duke.edu

| Participant's Agreement: I have read the information provided above. | • |
|---|---|
| Signature of Research Participant | Date |
| Printed Name of Research Participant | |

| Signature of Person Obtaining Consent | Date |
|------------------------------------------|------|
| Printed Name of Person Obtaining Consent | |